# STATISTICAL ANALYSIS PLAN

PROTOCOL NO: NCIG-006

# Randomized, Double Blind, Placebo-Controlled Trial of the Safety and Efficacy of HORIZANT® (Gabapentin Enacarbil) Extended-Release Tablets for the Treatment of Alcohol Use Disorder

**Protocol Version No.:** 5.0 Version Date: 18Aug2016

### **Study Sponsor:**

National Institute on Alcohol Abuse and Alcoholism

#### **Plan Authors:**

Charles B. Scott, Ph.D. Senior Biostatistician

Janet H. Ransom, Ph.D.
President
Fast-Track Drugs & Biologics, LLC
5 Paramus Ct.
North Potomac, Maryland 20878

Daniel E. Falk, Ph.D.
Director of Biostatistics
Division of Medications Development
National Institute on Alcohol Abuse and Alcoholism
National Institutes of Health
5635 Fishers Lane
Bethesda MD 20892

**Version Number 2.0** 

**Date: 22 August 2016** 

#### STATISTICAL ANALYSIS PLAN

#### PROTOCOL NO: NCIG-006

# Randomized, Double Blind, Placebo-Controlled Trial of the Safety and Efficacy of HORIZANT® (Gabapentin Enacarbil) Extended-Release Tablets for the Treatment of Alcohol Use Disorder

| Prepared by: | • | Date: | |
|---|---|---|---|
| p | Charles Scott, Ph.D. | | - |
| | Senior Biostatistician | | |
| | Fast-Track Drugs & Biologics, I | LLC | |
| | Janet Ranson | Digitally signed by Janet Ransom DN: cn=Janet Ransom, o=Fast-Track Drugs & Biologic LLC, ou, email=jransom@fasttrackresearch.com, c=U Date: 2016.08.22 14:42:58 -04'00' | is,<br>S |
| Prepared by: | : | Date: | |
| | Janet H. Ransom, Ph.D. | | |
| | President | | |
| | Fast-Track Drugs & Biologics, I | LLC | |
| | Daniel E. Falk - | Digitally signed by Daniel E. Falk -S<br>DN: c=US, o=U.S. Government, ou=HHS,<br>ou=NIH, ou=People, cn=Daniel E. Falk-S,<br>0.9.2342.19200300.100.1.1=0013044014<br>Date: 2016.08.22 16:06:56 -04'00' | |
| Prepared by: | | Date: | |
| | Daniel Falk, Ph.D. | | |
| | Director of Biostatistics | | |
| | Division of Medications Develop | • | |
| | National Institute on Alcohol Ab | ouse and Alcoholism | |

# **Table of Contents**

| 1. | ABBREVIATIONS 26 |
|---|---|
| 2. | INTRODUCTION 28 |
| 3. | PROTOCOL SUMMARY 29 3.1. Study Objectives 29 3.1.1 Primary 29 3.1.2 Secondary 29 3.2. Study Design 29 3.3. Study Endpoints 32 3.3.1 Primary Efficacy Endpoint 34 3.3.2 Secondary Efficacy Endpoints 34 3.3.3 Safety Endpoints 34 3.3.4 Compliance 35 |
| | 3.3.5. Pharmacokinetics |
| 4. | DEFINITION OF ANALYSIS SETS |
| 5. | ASSSESSMENT AND JUSTIFICATION OF STUDY ENDPOINTS 5.1. Alcohol Consumption Endpoints |
| 6. | HYPOTHESES TO BE TESTED426.1. Primary Efficacy Endpoint426.2. Secondary Efficacy Endpoints426.3 Exploratory Efficacy Endpoints42 |
| 7. | SAMPLE SIZE CONSIDERATIONS |
| 8. | DATA QUALITY ASSURANCE45 |
| 9. | STATISTICAL CONSIDERATIONS 46 9.1. General Considerations 46 9.2. Participant Accountability and Protocol Deviations 46 9.3. Demographics and Other Baseline Characteristics 46 9.4. Efficacy Analysis 47 9.4.1. Primary Analysis of the Primary Efficacy Endpoint 47 |

| | | 9.4.2. | | Adjustment for the Primary Analysis of the Primary Efficac | |
|---|---|---|---|---|---|
| | | 9.4.3. | | f the Secondary Efficacy Endpoints | |
| | | | 9.4.3.1. | Key Secondary Endpoint: Percentage of Subjects Abstiner | |
| | | | 9.4.3.2. | Secondary Drinking Endpoints | |
| | | | 9.4.3.3. | Alcohol Consequences and Craving Scales | |
| | | | 9.4.3.4. | Smoking Quantity | |
| | | | 9.4.3.5. | Depression, Anxiety, and Sleep Scales | |
| | | 9.4.4. | | Adjustment for the Analysis of Secondary Efficacy Endpoin | |
| | 9.5. | Handlii | ng of Missin | g Data | 50 |
| | | 9.5.1. | Primary Ar | nalysis of the Primary Efficacy Endpoint | 50 |
| | | 9.5.2. | Analysis of | f the Secondary Efficacy Endpoints | 50 |
| | 9.6. | Safety | Analysis | | 50 |
| | | 9.6.1. | Adverse Ev | vents | 50 |
| | | 9.6.2. | Clinical La | boratory and Point of Care Tests | 51 |
| | | 9.6.3. | Vital Signs | s, ECG, and Body Weight | 51 |
| | | 9.6.4. | CIWA-AR | Scores | 51 |
| | | 9.6.5. | Profile of N | Mood States | 51 |
| | 9.7. | Drug E | exposure and | Retention Analyses | 52 |
| | 9.8. | | | d Analysis | |
| | 9.9. | | | ntent | |
| | 9.10. | | | | |
| | 9.11. | | | ses | |
| | | | • | y Endpoint: Percentage of Subjects Abstinent from Smoking | |
| | | | | y Endpoint: MINI AUD Number of Symptoms | |
| | | | | y Endpoint: Blood PEth Levels | |
| | | | | d Secondary Endpoints With or Without Imputation over | 00 |
| | | J.11. I. | | tudy Periods | 53 |
| | | 9 11 5 | | s of Drinking Outcomes | |
| 1.0 | ***** | | | | |
| 10. | VALI | DATION | OF PROGE | RAMMING CODE | 55 |
| 11. | REFE | RENCES | S | | 56 |
| 12. | TARI | F LISTI | NG AND E | TIGURE SHELLS | 58 |
| 12. | 12.1. | | | TOOKE STILLES | |
| | 12.1. | | | sposition, Participation, Compliance | |
| | | | | hic and Baseline Characteristics | |
| | | | | ficacy Endpoint | |
| | | | | Efficacy Endpoints. | |
| | | | • | lyses | |
| | | | | y Analyses | |
| | | 12.1.0. | 12.1.6.1. | No Heavy Drinking Days by Week, Month and Grace Peri | |
| | | | 12.1.6.1. | Abstinent from Alcohol by Week, Month, and Grace Period | |
| | | | | taran da antara da a | )U141 |
| | | | 12.1.6.3. | WHO Drinking Grade Shifts by Week, Month, and Grace | 1.47 |
| | | | 10 1 6 4 | Period Abstinant from Cicaratta Smaking | |
| | | | 12.1.6.4. | Abstinent from Cigarette Smoking | |
| | | | 12.1.6.5. | Blood PEth Levels | |
| | | | 12.1.6.6. | MINI AUD Symptoms | . 103 |
| | | | 12.1.6.7 | Continuous Secondary Endpoints With and Without | 11.65 |
| | | | 10 1 6 0 | Imputation for Last 4 Weeks and Entire Maintenance Period | |
| | | | 12.1.6.8 | Subjects with No Heavy Drinking Days by Moderators | . 172 |

| | 12.2. Listings | |
|---|---|---|
| Appendix A. | Scale and Scoring Instructions for Pittsburg Sleep Quality Index | |
| | List of Tables | |
| Table 1: | Subject Disposition - All Randomized Subjects | 59 |
| Table 2: | Exposure to Investigational Products – mITT Subjects | 60 |
| Table 3: | Exposure to Investigational Products – Evaluable Subjects | 61 |
| Table 4: | Drug Compliance – mITT Subjects | 61 |
| Table 5: | Drug Compliance – Evaluable Subjects | 62 |
| Table 6: | Summary of HORIZANT Blood Levels – HORIZANT Group (mITT Subjects) | 62 |
| Table 7: | Summary of HORIZANT Blood Levels – HORIZANT Group (Evaluable Subjects) | 62 |
| Table 8: | Self Report of HORIZANT Use (within 24 hours prior to PK sample) Versus Positive Gabapentin Blood Level – mITT Subjects | 63 |
| Table 9: | Self Report of HORIZANT Use (within 24 hours prior to PK sample) Versus Positive<br>Gabapentin Blood Level – Evaluable Subjects | 63 |
| Table 10: | Exit Interview – mITT Subjects | 64 |
| Table 11: | Exit Interview – Evaluable Subjects | 65 |
| Table 12: | Dropouts by Treatment Group and Week – mITT Subjects | 66 |
| Table 13: | Dropouts by Treatment Group and Week – Evaluable Subjects | 66 |
| Table 14: | Number and Percent of Subjects Using Summary Drinking Questions after Discontinuing TLFB – mITT Subjects | _ |
| Table 15: | Number and Percent of Subjects Using Summary Drinking Questions after Discontinuing TLFB – Evaluable Subjects | |
| Table 16: | Demographic Characteristics - mITT Subjects | 69 |
| Table 17: | Demographic Characteristics - Evaluable Subjects | 71 |
| Table 18: | Psychiatric Baseline Characteristics – mITT Subjects | 72 |
| Table 19: | Psychiatric Baseline Characteristics – Evaluable Subjects. | 75 |
| Table 20: | Baseline POMS – mITT Subjects | 76 |
| Table 21: | Baseline POMS – Evaluable Subjects | 77 |
| Table 22: | Baseline PSQI – mITT Subjects | 78 |
| Table 23: | Baseline PSQI – Evaluable Subjects | 79 |
| Table 24: | Drinking-related Behavior and Characteristics – mITT Subjects | 80 |
| Table 25: | Drinking-related Behavior and Characteristics – Evaluable Subjects | 82 |

| Table 26: | Baseline Drinking by TLFB – mITT Subjects | 83 |
|---|---|---|
| Table 27: | Baseline Drinking by TLFB – Evaluable Subjects | 84 |
| Table 28: | Baseline Alcohol-Related Craving, Consequences, and Withdrawal - mITT Subjects | 85 |
| Table 29: | Baseline Alcohol-Related Craving, Consequences, and Withdrawal – Evaluable Subject | s86 |
| Table 30: | Baseline Other Substance Use – mITT Subjects | 87 |
| Table 31: | Baseline Other Substance Use – Evaluable Subjects | 88 |
| Table 32: | Subjects with No Heavy Drinking Days (mITT) – Full Model, Logistic Regression, Wed 22-25, with Imputation <sup>a</sup> | |
| Table 33: | Subjects with No Heavy Drinking Days (Evaluable) – Full Model, Logistic Regression, Weeks 22-25, with Imputation | |
| Table 34: | Percent Subjects Abstinent from Alcohol (mITT) - Weeks 22-25, With Imputation <sup>a</sup> | 92 |
| Table 35: | Subjects Abstinent from Alcohol (mITT) – Full Model, Logistic Regression, Weeks 22-With Imputation <sup>a</sup> | |
| Table 36: | Percent Subjects Abstinent from Alcohol (Evaluable) - Weeks 22-25, With Imputation <sup>a</sup> | . 92 |
| Table 37: | Subjects Abstinent from Alcohol (Evaluable) – Full Model, Logistic Regression, Weeks 22-25, with Imputation <sup>a</sup> | |
| Table 38: | WHO Shift Baseline to Weeks 22-25, No Imputation | 93 |
| Table 39: | WHO 1-Level Decrease in Alcohol Consumption (mITT) - Weeks 22-25, No Imputation | n93 |
| Table 40: | WHO 1-Level Decrease in Alcohol Consumption (mITT) – Full Model, Logistic Regression, Weeks 22-25, No Imputation | 93 |
| Table 41: | WHO 1-Level Decrease in Alcohol Consumption (Evaluable) – Weeks 22-25, No Imputation. | 94 |
| Table 42: | WHO 1-Level Decrease in Alcohol Consumption (Evaluable) – Full Model, Logistic Regression, Weeks 22-25, No Imputation | 94 |
| Table 43: | WHO 2-Level Decrease in Alcohol Consumption (mITT) – Weeks 22-25, No Imputation | n95 |
| Table 44: | WHO 2-Level Decrease in Alcohol Consumption (mITT) – Full Model, Logistic Regression, Weeks 22-25, No Imputation | 95 |
| Table 45: | WHO 2-Level Decrease in Alcohol Consumption (Evaluable) – Weeks 22-25, No Imputation | 95 |
| Table 46: | WHO 2-Level Decrease in Alcohol Consumption (Evaluable) – Full Model, Logistic Regression, Weeks 22-25, No Imputation | 95 |
| Table 47: | Percentage of Days Abstinent per Week (mITT) Full Model, Mixed Effects, Transformed, Weeks 22-25, No Imputation | 96 |
| Table 48: | Percentage of Days Abstinent per Week (Evaluable) Full Model, Mixed Effects, Transformed, Weeks 22-25, No Imputation | 96 |
| Table 49: | Percentage of Days Abstinent per Week (mITT) – Untransformed, Weeks 2-25, No | |

| | Imputation |
|---|---|
| Table 50: | Percentage of Days Abstinent per Week (Evaluable) – Untransformed, Weeks 2-25, No<br>Imputation |
| Table 51: | Percentage of Heavy Drinking Days per Week (mITT) – Full Model, Mixed Effects, Transformed, Weeks 22-25, No Imputation |
| Table 52: | Percentage of Heavy Drinking Days per Week (Evaluable) – Full Model, Mixed Effects, Transformed, Weeks 22-25, No Imputation |
| Table 53: | Percentage of Heavy Drinking Days per Week (mITT) – Untransformed, Weeks 2-25, No<br>Imputation |
| Table 54: | Percentage of Heavy Drinking Days per Week (Evaluable) – Untransformed, Weeks 2-25, No Imputation |
| Table 55: | Drinks per Week (mITT) – Full Model, Mixed Effects, Transformed, Weeks 22-25, No<br>Imputation |
| Table 56: | Drinks per Week (Evaluable) – Full Model, Mixed Effects, Transformed, Weeks 22-25, No<br>Imputation |
| Table 57: | Drinks per Week (mITT) – Untransformed, Weeks 2-25, No Imputation |
| Table 58: | Drinks per Week (Evaluable) – Untransformed, Weeks 2-25, No Imputation |
| Table 59: | Drinks per Drinking Day (mITT) – Full Model, Mixed Effects, Transformed, Weeks 22-25, No Imputation |
| Table 60: | Drinks per Drinking Day (Evaluable) – Full Model, Mixed Effects, Transformed, Weeks 22-25, No Imputation |
| Table 61: | Drinks per Drinking Day (mITT) – Untransformed, Weeks 2-25, No Imputation |
| Table 62: | Drinks per Drinking Day (Evaluable) – Untransformed, Weeks 2-25, No Imputation 103 |
| Table 63: | ACQ-SR-R Score (mITT) – Full Model, Mixed Effects, Transformed, Weeks 24 + 26 (covering last 4 weeks of maintenance phase), No Imputation |
| Table 64: | ACQ-SR-R Score (Evaluable) – Full Model, Mixed Effects, Transformed, Weeks 24 + 26 (covering last 4 weeks of maintenance phase), No Imputation |
| Table 65: | ACQ-SR-R Score (mITT) – Untransformed, Each Evaluation During Maintenance Period,<br>No Imputation |
| Table 66: | ACQ-SR-R Score (Evaluable) – Untransfomed, Each Evaluation During Maintenance<br>Period, No Imputation |
| Table 67: | ImBIBe Score (mITT) – Full Model, Mixed Effects, Transformed, Weeks 24 + 26 (covering last 4 weeks of maintenance phase), No Imputation |
| Table 68: | ImBIBe Score (Evaluable) – Full Model, Mixed Effects, Transformed, Weeks 24 + 26 (covering last 4 weeks of maintenance phase), No Imputation |
| Table 69: | ImBIBe Score (mITT) – Untransformed, Each Evaluation During Maintenance Period, No<br>Imputation |

| Table 70: | ImBIBe Score (Evaluable) – Untransformed, Each Evaluation During Maintenance Period,<br>No Imputation |
|---|---|
| Table 71: | Mean Cigarettes Smoked (mITT) – Full Model, Mixed Effects, Transformed, Weeks 24 + 26 (covering last 4 weeks of maintenance phase), No Imputation |
| Table 72: | Mean Cigarettes Smoked (Evaluable) – Full Model, Mixed Effects, Transformed, Weeks 24 + 26 (covering last 4 weeks of maintenance phase), No Imputation |
| Table 73: | Mean Cigarettes Smoked (mITT) – Untransformed, Each Evaluation During Maintenance<br>Period, No Imputation |
| Table 74: | Mean Cigarettes Smoked (Evaluable) – Untransformed, Each Evaluation During Maintenance Period, No Imputation |
| Table 75: | PSQI Score (mITT) – Full Model, Mixed Effects, Transformed, Weeks 24 + 26 (covering last 4 weeks of maintenance phase), No Imputation |
| Table 76: | PSQI Score (Evaluable) – Full Model, Mixed Effects, Transformed, Weeks 24 + 26 (covering last 4 weeks of maintenance phase), No Imputation |
| Table 77: | PSQI Score (mITT) – Untransformed, Each Evaluation During Maintenance Period, No<br>Imputation |
| Table 78: | PSQI Score (Evaluable) – Untransformed, Each Evaluation During Maintenance Period, No Imputation |
| Table 79: | PSQI Sleep Quality Score (mITT) – Full Model, Mixed Effects, Transformed, Weeks 24 + 26 (covering last 4 weeks of maintenance phase), No Imputation |
| Table 80: | PSQI Sleep Quality Score (Evaluable) – Full Model, Mixed Effects, Transformed, Weeks 24 + 26 (covering last 4 weeks of maintenance phase), No Imputation |
| Table 81: | PSQI Sleep Quality Score (mITT) – Untransformed, Each Evaluation During Maintenance<br>Period, No Imputation |
| Table 82: | PSQI Sleep Quality Score (Evaluable) – Untransformed, Each Evaluation During Maintenance Period, No Imputation |
| Table 83: | PSQI Sleep Latency Score (mITT) – Full Model, Mixed Effects, Transformed, Weeks 24 + 26 (covering last 4 weeks of maintenance phase), No Imputation |
| Table 84: | PSQI Sleep Latency Score (Evaluable) – Full Model, Mixed Effects, Transformed, Weeks 24 + 26 (covering last 4 weeks of maintenance phase), No Imputation |
| Table 85: | PSQI Sleep Latency Score (mITT) – Untransformed, Each Evaluation During Maintenance<br>Period, No Imputation |
| Table 86: | PSQI Sleep Latency Score (Evaluable) – Untransformed, Each Evaluation During Maintenance Period, No Imputation |
| Table 87: | PSQI Sleep Duration Score (mITT) – Full Model, Mixed Effects, Transformed, Weeks 24 + 26 (covering last 4 weeks of maintenance phase), No Imputation |
| Table 88: | PSQI Sleep Duration Score (Evaluable) – Full Model, Mixed Effects, Transformed, Weeks 24 + 26 (covering last 4 weeks of maintenance phase), No Imputation |

| Table 89: | PSQI Sleep Duration Score (mITT) – Untransformed, Each Evaluation During Maintenance Period, No Imputation |
|---|---|
| Table 90: | PSQI Sleep Duration Score (Evaluable) – Untransformed, Each Evaluation During<br>Maintenance Period, No Imputation |
| Table 91: | PSQI Sleep Disturbance Score (mITT) – Full Model, Mixed Effects, Transformed, Weeks 24 + 26 (covering last 4 weeks of maintenance phase), No Imputation |
| Table 92: | PSQI Sleep Disturbance Score (Evaluable) – Full Model, Mixed Effects, Transformed, Weeks 24 + 26 (covering last 4 weeks of maintenance phase), No Imputation |
| Table 93: | PSQI Sleep Disturbance Score (mITT) – Untransformed, Each Evaluation During Maintenance Period, No Imputation |
| Table 94: | PSQI Sleep Disturbance Score (Evaluable) – Untransformed, Each Evaluation During Maintenance Period, No Imputation |
| Table 95: | PSQI Use of Sleep Medication Score (mITT) – Full Model, Mixed Effects, Transformed, Weeks 24 + 26 (covering last 4 weeks of maintenance phase), No Imputation |
| Table 96: | PSQI Use of Sleep Medication Score (Evaluable) – Full Model, Mixed Effects,<br>Transformed, Weeks 24 + 26 (covering last 4 weeks of maintenance phase), No Imputation 11 |
| Table 97: | PSQI Use of Sleep Medication Score (mITT) – Untransformed, Each Evaluation During Maintenance Period, No Imputation |
| Table 98: | PSQI Use of Sleep Medication Score (Evaluable) – Untransformed, Each Evaluation During Maintenance Period, No Imputation |
| Table 99: | PSQI Daytime Dysfunction Score (mITT) – Full Model, Mixed Effects, Transformed, Weeks 24 + 26 (covering last 4 weeks of maintenance phase), No Imputation |
| Table 100: | PSQI Daytime Dysfunction Score (Evaluable) – Full Model, Mixed Effects, Transformed, Weeks 24 + 26 (covering last 4 weeks of maintenance phase), No Imputation |
| Table 101: | PSQI Daytime Dysfunction Score (mITT) – Untransformed, Each Evaluation During Maintenance Period, No Imputation |
| Table 102: | PSQI Daytime Dysfunction Score (Evaluable) – Untransformed, Each Evaluation During Maintenance Period, No Imputation |
| Table 103: | BAI Score (mITT) – Full Model, Mixed Effects, Transformed, Weeks 24 + 26 (covering last 4 weeks of maintenance phase), No Imputation |
| Table 104: | BAI Score (Evaluable) – Full Model, Mixed Effects, Transformed, Weeks 24 + 26 (covering last 4 weeks of maintenance phase), No Imputation |
| Table 105: | BAI Score (mITT) – Untransformed, Each Evaluation During Maintenance Period, No<br>Imputation |
| Table 106: | BAI Score (Evaluable) – Untransformed, Each Evaluation During Maintenance Period, No<br>Imputation |
| Table 107: | BDI-II Score (mITT) – Full Model, Mixed Effects, Transformed, Weeks 24 + 26 (covering last 4 weeks of maintenance phase), No Imputation |

| Table 108: | BDI-II Score (Evaluable) – Full Model, Mixed Effects, Transformed, Weeks 24 + 2 (covering last 4 weeks of maintenance phase), No Imputation | |
|---|---|---|
| Table 109: | BDI-II Score (mITT) – Untransformed, Each Evaluation During Maintenance Perio Imputation | |
| Table 110: | BDI-II Score (Evaluable) – Untransformed, Each Evaluation During Maintenance P<br>No Imputation | |
| Table 111: | Overall Summary of Adverse Events – mITT Subjects | 117 |
| Table 112: | Number and Percentage of Subjects with Adverse Events - mITT Subjects | 117 |
| Table 113: | Summary of Subjects with Adverse Events by Severity and Relationship – HORIZA | ANT118 |
| Table 114: | Summary of Subjects with Adverse Events by Severity and Relationship – Placebo . | 118 |
| Table 115: | Number and Percentage of Subjects with Adverse Events by Maximum Severity - n<br>Subjects | |
| Table 116: | Number and Percentage of Subjects Adverse Events by Relatedness - mITT Subject | s 119 |
| Table 117: | Number and Percentage of Subjects with Treatment-Related Adverse Events by Ma<br>Severity- mITT Subjects | |
| Table 118: | Number and Percentage of Subjects with Adverse Events Occurring in >= 5% - mIT Subjects | |
| Table 119: | Number and Percentage of Subjects with Adverse Events Leading to Discontinuation Study - mITT Subjects | |
| Table 120: | Number and Percentage of Subjects with Adverse Events Leading to Discontinuation Study Medication – mITT Subjects | |
| Table 121: | Number and Percentage of Subjects with Somnolence or Dizziness AEs that Started Drinking Day – mITT Subjects | |
| Table 122: | CIWA-AR Score > 10 at Least Once During Treatment – mITT Subjects | 122 |
| Table 123: | Summary of Vital Signs and Body Weights – mITT Subjects | 122 |
| Table 124: | Summary of Other Services Used During Treatment Period – mITT Subjects | 123 |
| Table 125: | Summary of ECG Results - mITT Subjects | 123 |
| Table 126: | Summary of Blood Chemistries – mITT Subjects | 124 |
| Table 127: | Summary of Positive Urine Drug Tests, Preganancy Test or BAC > 0.000 Any Time During the Study–mITT Subjects | |
| Table 128: | POMS Total Mood Disturbance Score (mITT) Full Model, Mixed Effects, Trans<br>Entire Maintenance Period, No Imputation | |
| Table 129: | POMS Total Mood Disturbance Score (mITT)Untransformed, Each Evaluation D Maintenance Period, No Imputation | • |
| Table 130: | POMS Tension-Anxiety Score (mITT) Full Model, Mixed Effects, Transformed, Maintenance Period, No Imputation | |

| Table 131: | POMS Tension-Anxiety Score (mITT) Untransformed, Each Evaluation During Maintenance Period, No Imputation |
|---|---|
| Table 132: | POMS Anger-Hostility Score (mITT) Full Model, Mixed Effects, Transformed, Entire Maintenance Period, No Imputation |
| Table 133: | POMS Anger-Hostility Score (mITT) Untransformed, Each Evaluation During Maintenance Period, No Imputation |
| Table 134: | POMS Vigor-Activity Score (mITT) Full Model, Mixed Effects, Transformed, Entire Maintenance Period, No Imputation |
| Table 135: | POMS Vigor-Activity Score (mITT) Untransformed, Each Evaluation During Maintenance Period, No Imputation |
| Table 136: | POMS Fatigue-Inertia Score (mITT) Full Model, Mixed Effects, Transformed, Entire Maintenance Period, No Imputation |
| Table 137: | POMS Fatigue-Inertia Score (mITT) Untransformed, Each Evaluation During Maintenance Period, No Imputation |
| Table 138: | POMS Confusion-Bewilderment Score (mITT) Full Model, Mixed Effects, Transformed, Entire Maintenance Period, No Imputation |
| Table 139: | POMS Confusion-Bewilderment Score (mITT) Untransformed, Each Evaluation During Maintenance Period, No Imputation |
| Table 140: | POMS Depression-Dejection Score (mITT) Full Model, Mixed Effects, Transformed,<br>Entire Maintenance Period, No Imputation |
| Table 141: | POMS Depression-Dejection Score (mITT) Untransformed, Each Evaluation During Maintenance Period, No Imputation |
| Table 142: | Frequency of Subjects with Suicidal Ideation Any Time During the Study – mITT Subjects128 |
| Table 143: | Summary of Concomitant Medication Use – mITT Subjects |
| Table 144: | Percentage of Subjects No Heavy Drinking Days (mITT) – Weeks 22-25, with Imputation <sup>a</sup> 130 |
| Table 145: | Percentage of Subjects No Heavy Drinking Days Weeks 22-25 – No Imputation (mITT)130 |
| Table 146: | Percentage of Subjects with No Heavy Drinking Days Weeks 22-25 – Full Model No Imputation Logistic Regression (mITT) |
| Table 147: | Percentage of Subjects No Heavy Drinking Days Weekly with Imputation <sup>a</sup> (mITT) 132 |
| Table 148: | Summary of Percentage of Subjects No Heavy Drinking Days (mITT) – Full Model, Weekly, with Imputation <sup>a</sup> |
| Table 149: | Percentage of Subjects No Heavy Drinking Days Weekly No Imputation (mITT) 135 |
| Table 150: | Summary of Percentage of Subjects No Heavy Drinking Days (mITT) – Full Model, Weekly, No Imputation |
| Table 151: | Percentage of Subjects No Heavy Drinking Days Monthly with Imputation <sup>a</sup> (mITT) 136 |
| Table 152: | Summary of Percentage of Subjects No Heavy Drinking Days (mITT) – Full Model, Monthly, with Imputation <sup>a</sup> |

| Table 153: | Percentage of Subjects No Heavy Drinking Days Monthly No Imputation (mITT) 138 |
|---|---|
| Table 154: | Summary of Percentage of Subjects No Heavy Drinking Days (mITT) – Full Model, Monthly, No Imputation |
| Table 155: | Percentage of Subjects No Heavy Drinking Days - Weeks 18-25 with Imputation <sup>a</sup> (last 8 weeks) (mITT) |
| Table 156: | Subjects with No Heavy Drinking Days (mITT) – Logistic Regression, Weeks 18-25 (last 8 weeks), with Imputation <sup>a</sup> |
| Table 157: | Percentage of Subjects No Heavy Drinking Days - Weeks 18-25 No Imputation (last 8 weeks) (mITT) |
| Table 158: | Subjects with No Heavy Drinking Days (mITT) – Logistic Regression, Weeks 18-25 (last 8 weeks), No Imputation |
| Table 159: | Percentage of Subjects No Heavy Drinking Days - Weeks 14-25 with Imputation <sup>a</sup> (last 12 weeks) (mITT) |
| Table 160: | Subjects with No Heavy Drinking Days (mITT) – Logistic Regression, Weeks 14-25 (last 12 weeks), with Imputation <sup>a</sup> |
| Table 161: | Percentage of Subjects No Heavy Drinking Days - Weeks 14-25 No Imputation (last 12 weeks) (mITT) |
| Table 162: | Subjects with No Heavy Drinking Days (mITT) – Logistic Regression, Weeks 14-25 (last 12 weeks), No Imputation |
| Table 163: | Percentage of Subjects No Heavy Drinking Days - Weeks 10-25 (last 16 weeks) with Imputation <sup>a</sup> (mITT) |
| Table 164: | Subjects with No Heavy Drinking Days (mITT) – Logistic Regression, Weeks 10-25 (last 16 weeks), with Imputation <sup>a</sup> |
| Table 165: | Percentage of Subjects No Heavy Drinking Days - Weeks 10-25 (last 16 weeks) No Imputation (mITT) |
| Table 166: | Subjects with No Heavy Drinking Days (mITT) – Logistic Regression, Weeks 10-25 (last 16 weeks), No Imputation |
| Table 167: | Percentage of Subjects No Heavy Drinking Days - Weeks 6-25 (last 20 weeks) with Imputation <sup>a</sup> (mITT) |
| Table 168: | Subjects with No Heavy Drinking Days (mITT) – Logistic Regression, Weeks 6-25 (last 20 weeks) , with Imputation <sup>a</sup> |
| Table 169: | Percentage of Subjects No Heavy Drinking Days - Weeks 6-25 (last 20 weeks) No Imputation (mITT) |
| Table 170: | Subjects with No Heavy Drinking Days (mITT) – Logistic Regression, Weeks 6-25 (last 20 weeks) , No Imputation |
| Table 171: | Percentage of Subjects No Heavy Drinking Days - Weeks 2-25 (complete maintenance period) with Imputation <sup>a</sup> (mITT) |
| Table 172: | Subjects with No Heavy Drinking Days (mITT) – Logistic Regression, Weeks 2-25 |
| Statistical A | Analysis Plan: Protocol NCIG-006, Version 2.0 Dated: 22Aug2016 12 |

| | (complete maintenance period), with Imputation <sup>a</sup> | 140 |
|---|---|---|
| Table 173: | Percentage of Subjects No Heavy Drinking Days - Weeks 2-25 (complete maintenance period) No Imputation (mITT) | |
| Table 174: | Subjects with No Heavy Drinking Days (mITT) – Logistic Regression, Weeks 2-25 (complete maintenance period), No Imputation | 140 |
| Table 175: | Percentage of Subjects Abstinent from Alcohol Weeks 22-25 with Imputation <sup>a</sup> (mITT). | 141 |
| Table 176: | Subjects Abstinent from Alcohol (mITT) – Logistic Regression, Weeks 22-25, with Imputation <sup>a</sup> | 141 |
| Table 177: | Percentage of Subjects Abstinent from Alcohol Weekly with Imputation <sup>a</sup> (mITT) | 141 |
| Table 178: | Summary of Subjects Abstinent from Alcohol (mITT) – Logistic Regression, Weekly, v<br>Imputation <sup>a</sup> | |
| Table 179: | Percentage of Subjects Abstinent from Alcohol Weekly No Imputation (mITT) | 144 |
| Table 180: | Summary of Subjects Abstinent from Alcohol (mITT) – Logistic Regression, Weekly, Imputation | |
| Table 181: | Percentage of Subjects Abstinent Monthly with Imputation <sup>a</sup> (mITT) | 144 |
| Table 182: | Summary of Subjects Abstinent from Alcohol (mITT) – Logistic Regression, Monthly, With Imputation <sup>a</sup> | 145 |
| Table 183: | Percentage of Subjects Abstinent from Alcohol Monthly No Imputation (mITT) | 145 |
| Table 184: | Summary of Subjects Abstinent from Alcohol (mITT) – Logistic Regression, Weekly, Imputation | |
| Table 185: | Percentage of Subjects Abstinent from Alcohol - Weeks 18-25 with Imputation <sup>a</sup> (last 8 weeks) (mITT) | 145 |
| Table 186: | Subjects Abstinent from Alcohol (mITT) – Logistic Regression, Weeks 18-25 (last 8 weeks), with Imputation <sup>a</sup> | 145 |
| Table 187: | Percentage of Subjects Abstinent from Alcohol - Weeks 18-25 No Imputation (last 8 weeks) (mITT) | 146 |
| Table 188: | Subjects Abstinent from Alcohol (mITT) – Logistic Regression, Weeks 18-25 (last 8 weeks), No Imputation | 146 |
| Table 189: | Percentage of Subjects Abstinent from Alcohol - Weeks 14-25 with Imputation <sup>a</sup> (last 12 weeks) (mITT) | |
| Table 190: | Subjects Abstinent from Alcohol (mITT) – Logistic Regression, Weeks 14-25 (last 12 weeks), with Imputation <sup>a</sup> | 146 |
| Table 191: | Percentage of Subjects Abstinent from Alcohol - Weeks 14-25 No Imputation (last 12 weeks) (mITT) | 146 |
| Table 192: | Subjects Abstinent from Alcohol (mITT) – Logistic Regression, Weeks 14-25 (last 12 weeks), No Imputation | 146 |
| Table 193: | Percentage of Subjects Abstinent from Alcohol - Weeks 10-25 (last 16 weeks) with | |

| | Imputation <sup>a</sup> (mITT) | 146 |
|---|---|---|
| Table 194: | Subjects Abstinent from Alcohol (mITT) – Logistic Regression, Weeks 10-25 (last 16 weeks), with Imputation <sup>a</sup> | 146 |
| Table 195: | Percentage of Subjects Abstinent from Alcohol- Weeks 10-25 (last 16 weeks) No Imputation (mITT) | 146 |
| Table 196: | Subjects Abstinent from Alcohol (mITT) – Logistic Regression, Weeks 10-25 (last 16 weeks), No Imputation <sup>a</sup> | 146 |
| Table 197: | Percentage of Subjects Abstinent from Alcohol - Weeks 6-25 (last 20 weeks) with Imputation <sup>a</sup> (mITT) | 146 |
| Table 198: | Subjects Abstinent from Alcohol (mITT) – Logistic Regression, Weeks 6-25 (last 20 weeks), with Imputation <sup>a</sup> | 146 |
| Table 199: | Percentage of Subjects Abstinent from Alcohol - Weeks 6-25 (last 20 weeks) No Imputation (mITT) | 146 |
| Table 200: | Subjects Abstinent from Alcohol (mITT) – Logistic Regression, Weeks 6-25 (last 20 weeks), No Imputation | 146 |
| Table 201: | Percentage of Subjects Abstinent from Alcohol - Weeks 2-25 (complete maintenance period) with Imputation <sup>a</sup> (mITT) | 146 |
| Table 202: | Subjects Abstinent from Alcohol (mITT) – Logistic Regression, Weeks 2-25 (complete maintenance period), with Imputation <sup>a</sup> | 146 |
| Table 203: | Percentage of Subjects Abstinent from Alcohol - Weeks 2-25 (complete maintenance period) No Imputation (mITT) | 146 |
| Table 204: | Subjects Abstinent from Alcohol (mITT) – Logistic Regression, Weeks 2-25 (complete maintenance period), No Imputation | 146 |
| Table 205: | WHO Shift Baseline to Weeks 22-25, No Imputation (mITT) | 147 |
| Table 206: | WHO 1-Level Decrease in Alcohol Consumption Weeks 22-25 No Imputation (mITT). 1 | 47 |
| Table 207: | WHO 1-Level Decrease in Alcohol Consumption (mITT) – Logistic Regression, Weeks 22-25, No Imputation | 147 |
| Table 208: | WHO 2-Level Decrease in Alcohol Consumption Weeks 22-25 No Imputation (mITT). 1 | 48 |
| Table 209: | WHO 2-Level Decrease in Alcohol Consumption (mITT) – Logistic Regression, Weeks 22-25, No Imputation | 148 |
| Table 210: | WHO Shift Baseline to Weekly Time Period, with Imputation <sup>a</sup> (mITT) | 149 |
| Table 211: | Percentage of Subjects WHO 1-Level Decrease in Alcohol Consumption Weekly with Imputation <sup>a</sup> (mITT) | 149 |
| Table 212: | Summary of WHO 1-Level Decrease in Alcohol Consumption (mITT) – Logistic Regression, Weekly, with Imputation <sup>a</sup> | 150 |
| Table 213: | Percentage of Subjects WHO 2-Level Decrease in Alcohol Consumption Weekly with Imputation <sup>a</sup> (mITT) | 153 |

| Table 214: | Summary of WHO 2-Level Decrease in Alcohol Consumption (mITT) – Logistic Regression, Weekly, with Imputation <sup>a</sup> | 53 |
|---|---|---|
| Table 215: | WHO Shift Baseline to Weekly Time Period, No Imputation <sup>a</sup> (mITT) | 56 |
| Table 216: | Percentage of Subjects WHO 1-Level Decrease in Alcohol Consumption Weekly No Imputation (mITT) | 56 |
| Table 217: | Summary of WHO 1-Level Decrease in Alcohol Consumption (mITT) – Logistic Regression, Weekly, No Imputation | 56 |
| Table 218: | Percentage of Subjects WHO 2-Level Decrease in Alcohol Consumption Weekly No Imputation (mITT) | 56 |
| Table 219: | Summary of WHO 2-Level Decrease in Alcohol Consumption (mITT) – Logistic Regression, Weekly, No Imputation | 56 |
| Table 220: | WHO Shift Baseline to Monthly Time Period, with Imputation <sup>a</sup> (mITT) | 56 |
| Table 221: | Percentage of Subjects WHO 1-Level Decrease in Alcohol Consumption Monthly with Imputation (mITT) | 56 |
| Table 222: | Summary of WHO 1-Level Decrease in Alcohol Consumption (mITT) – Logistic Regression, Monthly, with Imputation <sup>a</sup> | 56 |
| Table 223: | Percentage of Subjects WHO 2-Level Decrease in Alcohol Consumption Monthly with Imputation <sup>a</sup> (mITT) | 56 |
| Table 224: | Summary of WHO 2-Level Decrease in Alcohol Consumption (mITT) – Logistic Regression, Monthly, with Imputation <sup>a</sup> | 56 |
| Table 225: | WHO Shift Baseline to Monthly Time Period, No Imputation <sup>a</sup> (mITT) | 56 |
| Table 226: | Percentage of Subjects WHO 1-Level Decrease in Alcohol Consumption Monthly No Imputation (mITT) | 56 |
| Table 227: | Summary of WHO 1-Level Decrease in Alcohol Consumption (mITT) – Logistic Regression, Monthly, No Imputation | 56 |
| Table 228: | Percentage of Subjects WHO 2-Level Decrease in Alcohol Consumption Monthly No Imputation (mITT) | 56 |
| Table 229: | Summary of WHO 2-Level Decrease in Alcohol Consumption (mITT) – Logistic Regression, Monthly, No Imputation | 56 |
| Table 230: | WHO Shift Baseline to Weeks 18-25 (last 8 weeks), with Imputation <sup>a</sup> (mITT) | 56 |
| Table 231: | Percentage of Subjects WHO 1-Level Decrease in Alcohol Consumption Weeks 18-25 with Imputation <sup>a</sup> (last 8 weeks) (mITT) | 56 |
| Table 232: | Subjects with WHO 1-Level Decrease in Alcohol Consumption (mITT) – Logistic Regression, Weeks 18-25 (last 8 weeks), with Imputation <sup>a</sup> | 56 |
| Table 233: | Percentage of Subjects WHO 2-Level Decrease in Alcohol Consumption Weeks 18-25 with Imputation <sup>a</sup> (last 8 weeks) (mITT) | |
| Table 234: | Subjects with WHO 2-Level Decrease in Alcohol Consumption (mITT) – Logistic | |

| | Regression, Weeks 18-25 (last 8 weeks), with Imputation <sup>a</sup> | 157 |
|---|---|---|
| Table 235: | WHO Shift Baseline to Weeks 18-25 (last 8 weeks), No Imputation <sup>a</sup> (mITT) | 157 |
| Table 236: | Percentage of Subjects WHO 1-Level Decrease in Alcohol Consumption Weeks 18-25 Imputation (last 8 weeks) (mITT) | |
| Table 237: | Subjects with WHO 1-Level Decrease in Alcohol Consumption (mITT) – Logistic Regression, Weeks 18-25 (last 8 weeks), No Imputation | 157 |
| Table 238: | Percentage of Subjects WHO 2-Level Decrease in Alcohol Consumption Weeks 18-25 Imputation (last 8 weeks) (mITT) | |
| Table 239: | Subjects with WHO 2-Level Decrease in Alcohol Consumption (mITT) – Logistic Regression, Weeks 18-25 (last 8 weeks), No Imputation | 157 |
| Table 240: | WHO Shift Baseline to Weeks 14-25 (last 12 weeks), with Imputation <sup>a</sup> (mITT) | 157 |
| Table 241: | Percentage of Subjects WHO 1-Level Decrease in Alcohol Consumption Weeks 14-25 with Imputation <sup>a</sup> (last 12 weeks) (mITT) | |
| Table 242: | Subjects with WHO 1-Level Decrease in Alcohol Consumption (mITT) – Logistic Regression, Weeks 14-25 (last 12 weeks), with Imputation <sup>a</sup> | 157 |
| Table 243: | Percentage of Subjects WHO 2-Level Decrease in Alcohol Consumption Weeks 14-25 with Imputation <sup>a</sup> (last 12 weeks) (mITT) | |
| Table 244: | Subjects with WHO 2-Level Decrease in Alcohol Consumption (mITT) – Logistic Regression, Weeks 14-25 (last 12 weeks), with Imputation <sup>a</sup> | 157 |
| Table 245: | WHO Shift Baseline to Weeks 14-25 (last 12 weeks), No Imputation <sup>a</sup> (mITT) | 157 |
| Table 246: | Percentage of Subjects WHO 1-Level Decrease in Alcohol Consumption Weeks 14-25 Imputation (last 12 weeks) (mITT) | |
| Table 247: | Subjects with WHO 1-Level Decrease in Alcohol Consumption (mITT) – Logistic Regression, Weeks 14-25 (last 12 weeks), No Imputation | 157 |
| Table 248: | Percentage of Subjects WHO 2-Level Decrease in Alcohol Consumption Weeks 14-25 Imputation (last 12 weeks) (mITT) | |
| Table 249: | Subjects with WHO 2-Level Decrease in Alcohol Consumption (mITT) – Logistic Regression, Weeks 14-25 (last 12 weeks), No Imputation | 158 |
| Table 250: | WHO Shift Baseline to Weeks 10-25 (last 16 weeks), with Imputation <sup>a</sup> (mITT) | 158 |
| Table 251: | Percentage of Subjects WHO 1-Level Decrease in Alcohol Consumption Weeks 10-25 (last 16 weeks) with Imputation <sup>a</sup> (mITT) | |
| Table 252: | Subjects with WHO 1-Level Decrease in Alcohol Consumption (mITT) – Logistic Regression, Weeks 10-25 (last 16 weeks), with Imputation <sup>a</sup> | 158 |
| Table 253: | Percentage of Subjects WHO 2-Level Decrease in Alcohol Consumption Weeks 10-25 (last 16 weeks) with Imputation <sup>a</sup> (mITT) | |
| Table 254: | Subjects with WHO 2-Level Decrease in Alcohol Consumption (mITT) – Logistic Regression, Weeks 10-25 (last 16 weeks), with Imputation <sup>a</sup> | 158 |

| Table 255: | WHO Shift Baseline to Weeks 10-25 (last 16 weeks), No Imputation <sup>a</sup> (mITT) |
|---|---|
| Table 256: | Percentage of Subjects WHO 1-Level Decrease in Alcohol Consumption Weeks 10-25 (last 16 weeks) No Imputation (mITT) |
| Table 257: | Subjects with WHO 1-Level Decrease in Alcohol Consumption (mITT) – Logistic Regression, Weeks 10-25 (last 16 weeks), No Imputation |
| Table 258: | Percentage of Subjects WHO 2-Level Decrease in Alcohol Consumption Weeks 10-25 (last 16 weeks) No Imputation (mITT) |
| Table 259: | Subjects with WHO 2-Level Decrease in Alcohol Consumption (mITT) – Logistic Regression, Weeks 10-25 (last 16 weeks), No Imputation |
| Table 260: | WHO Shift Baseline to Weeks 6-25 (last 20 weeks), with Imputation <sup>a</sup> (mITT)158 |
| Table 261: | Percentage of Subjects WHO 1-Level Decrease in Alcohol Consumption Weeks 6-25 (last 20 weeks) with Imputation <sup>a</sup> (mITT) |
| Table 262: | Subjects with WHO 1-Level Decrease in Alcohol Consumption (mITT) – Logistic Regression, Weeks 6-25 (last 20 weeks), with Imputation <sup>a</sup> |
| Table 263: | Percentage of Subjects WHO 2-Level Decrease in Alcohol Consumption Weeks 6-25 (last 20 weeks) with Imputation <sup>a</sup> (mITT) |
| Table 264: | Subjects with WHO 2-Level Decrease in Alcohol Consumption (mITT) – Logistic Regression, Weeks 6-25 (last 20 weeks), with Imputation <sup>a</sup> |
| Table 265: | WHO Shift Baseline to Weeks 6-25 (last 20 weeks), No Imputation <sup>a</sup> (mITT) |
| Table 266: | Percentage of Subjects WHO 1-Level Decrease in Alcohol Consumption Weeks 6-25 (last 20 weeks) No Imputation (mITT) |
| Table 267: | Subjects with WHO 1-Level Decrease in Alcohol Consumption (mITT) – Logistic Regression, Weeks 6-25 (last 20 weeks), No Imputation |
| Table 268: | Percentage of Subjects WHO 2-Level Decrease in Alcohol Consumption Weeks 6-25 (last 20 weeks) No Imputation (mITT) |
| Table 269: | Subjects with WHO 2-Level Decrease in Alcohol Consumption (mITT) – Logistic Regression, Weeks 6-25 (last 20 weeks), No Imputation |
| Table 270: | WHO Shift Baseline to Weeks 2-25 (complete maintenance period), with Imputation <sup>a</sup> (mITT) |
| Table 271: | Percentage of Subjects WHO 1-Level Decrease in Alcohol Consumption Weeks 2-25 (complete maintenance period) with Imputation <sup>a</sup> (mITT) |
| Table 272: | Subjects with WHO 1-Level Decrease in Alcohol Consumption (mITT) – Logistic Regression, Weeks 2-25 (complete maintenance period), with Imputation <sup>a</sup> |
| Table 273: | Percentage of Subjects WHO 2-Level Decrease in Alcohol Consumption Weeks 2-25 (complete maintenance period) with Imputation <sup>a</sup> (mITT) |
| Table 274: | Subjects with WHO 2-Level Decrease in Alcohol Consumption (mITT) – Logistic Regression, Weeks 2-25 (complete maintenance period), with Imputation <sup>a</sup> |

| Table 275: | WHO Shift Baseline to Weeks 2-25 (complete maintenance period), No Imputation <sup>a</sup> (mITT) |
|---|---|
| Table 276: | Percentage of Subjects WHO 1-Level Decrease in Alcohol Consumption Weeks 2-25 (complete maintenance period) No Imputation (mITT) |
| Table 277: | Subjects with WHO 1-Level Decrease in Alcohol Consumption (mITT) – Logistic Regression, Weeks 2-25 (complete maintenance period), No Imputation |
| Table 278: | Percentage of Subjects WHO 2-Level Decrease in Alcohol Consumption Weeks 2-25 (complete maintenance period) No Imputation (mITT) |
| Table 279: | Subjects with WHO 2-Level Decrease in Alcohol Consumption (mITT) – Logistic Regression, Weeks 2-25 (complete maintenance period), No Imputation |
| Table 280: | Percentage of Subjects Abstinent from Cigarettes among Smokers Weeks 24 + 26 – No Imputation (mITT) |
| Table 281: | Subjects Abstinent from Cigarettes among Smokers (mITT) – Logistic Regression, Weeks 24 + 26, No Imputation |
| Table 282: | Percentage of Subjects Abstinent from Cigarettes among Smokers Weeks 24 + 26 – with Imputation <sup>a</sup> (mITT) |
| Table 283: | Subjects Abstinent from Cigarettes among Smokers (mITT) – Logistic Regression, Weeks 24 + 26, No Imputation <sup>a</sup> |
| Table 284: | Percentage of Subjects Abstinent from Cigarettes among Smokers Entire Maintenance Period – No Imputation (mITT) |
| Table 285: | Subjects Abstinent from Cigarettes among Smokers (mITT) – Logistic Regression, Entire Maintenance Period, No Imputation |
| Table 286: | Percentage of Subjects Abstinent from Cigarettes among Smokers Entire Maintenance Period – with Imputation (mITT) |
| Table 287: | Subjects Abstinent from Cigarettes among Smokers (mITT) – Logistic Regression, Entire Maintenance Period, with Imputation <sup>a</sup> |
| Table 288: | Blood PEth Levels (ng/mL) (mITT) – Analysis of Covariance, Transformed, Week 26, No Imputation |
| Table 289: | Percentages of Negative Blood PEth Samples at Week 26 – No Imputation (mITT) 163 |
| Table 290: | Samples with No Detectable Blood PEth Levels (mITT) – Logistic Regression, Week 26, No Imputation |
| Table 291: | MINI AUD Number of Symptoms (mITT) – Analysis of Covariance, Week 26, No Imputation |
| Table 292: | Percentage of Heavy Drinking Days per Week (mITT) – Mixed Effects, Transformed, Weeks 22-25, with Imputation <sup>a</sup> |
| Table 293: | Percentage of Heavy Drinking Days per Week (mITT) Mixed Effects, Transformed, Weeks 2-25 No Imputation |
| Table 294: | Percentage of Heavy Drinking Days per Week (mITT) Mixed Effects, Transformed, |
| Statistical A | Analysis Plan: Protocol NCIG-006, Version 2.0 Dated: 22Aug2016 18 |

| | Weeks 2-25, with Imputation |
|---|---|
| Table 295: | Percentage of Days Abstinent per Week (mITT) – Mixed Effects, Transformed, Weeks 22-25, with Imputation |
| Table 296: | Percentage of Days Abstinent per Week (mITT) – Mixed Effects, Transformed, Weeks 2-25, No Imputation |
| Table 297: | Percentage of Days Abstinent per Week (mITT) – Mixed Effects, Transformed, Weeks 2-25, with Imputation |
| Table 298: | Drinks per Week (mITT) - Mixed Effects, Transformed, Weeks 22-25, with Imputation169 |
| Table 299: | Drinks per Week (mITT) - Mixed Effects, Transformed, Weeks 2-25, No Imputation 169 |
| Table 300: | Drinks per Week (mITT) – Mixed Effects, Transformed, Weeks 2-25, with Imputation. 169 |
| Table 301: | Drinks per Drinking Day (mITT) – Mixed Effects, Transformed, Weeks 22-25, with Imputation |
| Table 302: | Drinks per Drinking Day (mITT) – Mixed Effects, Transformed, Weeks 2-25, No Imputation |
| Table 303: | Drinks per Drinking Day (mITT) – Mixed Effects, Transformed, Weeks 2-25, with Imputation |
| Table 304: | ACQ-SR-R Score (mITT) – Mixed Effects, Transformed, Weeks 24 + 26, with Imputation 169 |
| Table 305: | ACQ-SR-R Score (mITT) – Mixed Effects, Transformed, Weeks 2-26, No Imputation 170 |
| Table 306: | ACQ-SR-R Score (mITT) – Mixed Effects, Transformed, Weeks 2-26, with Imputation 170 |
| Table 307: | ImBIBe Score (mITT) – Mixed Effects, Transformed, Weeks 24 + 26, with Imputation 170 |
| Table 308: | ImBIBe Score (mITT) – Mixed Effects, Transformed, Weeks 2-26, No Imputation 170 |
| Table 309: | ImBIBe Score (mITT) – Mixed Effects, Transformed, Weeks 2-26, with Imputation 170 |
| Table 310: | Mean Cigarettes Smoked per Week among Smokers (mITT) – Mixed Effects, Transformed, Weeks 24 + 26 with Imputation |
| Table 311: | Mean Cigarettes Smoked per Week among Smokers (mITT) – Mixed Effects, Transformed, Weeks 2-26, No Imputation |
| Table 312: | Mean Cigarettes Smoked per Week among Smokers (mITT) – Mixed Effects, Transformed, Weeks 2-26, with Imputation |
| Table 313: | PSQI Score (mITT) – Mixed Effects, Transformed, Weeks 24 + 26, with Imputation 170 |
| Table 314: | PSQI Score (mITT) – Mixed Effects, Transformed, Weeks 2-26, No Imputation |
| Table 315: | PSQI Score (mITT) – Mixed Effects, Transformed, Weeks 2-26, with Imputation 171 |
| Table 316: | PSQI Sleep Quality Score (mITT) – Mixed Effects, Transformed, Weeks 24 + 26, with Imputation |
| Table 317: | PSQI Sleep Quality Score (mITT) – Mixed Effects, Transformed, Weeks 2-26, No<br>Imputation |
| Table 318: | PSQI Sleep Quality Score (mITT) – Mixed Effects, Transformed, Weeks 2-26, with |
| Statistical | Analysis Plan: Protocol NCIG-006, Version 2.0 Dated: 22Aug2016 19 |

| | Imputation |
|---|---|
| Table 319: | PSQI Sleep Latency Score (mITT) – Mixed Effects, Transformed, Weeks 24 + 26, with Imputation |
| Table 320: | PSQI Sleep Latency Score (mITT) – Mixed Effects, Transformed, Weeks 2-26, No<br>Imputation |
| Table 321: | PSQI Sleep Latency Score (mITT) – Mixed Effects, Transformed, Weeks 2-26, with Imputation |
| Table 322: | PSQI Sleep Duration Score (mITT) – Mixed Effects, Transformed, Weeks 24 + 26, with Imputation |
| Table 323: | PSQI Sleep Duration Score (mITT) – Mixed Effects, Transformed, Weeks 2-26, No<br>Imputation |
| Table 324: | PSQI Sleep Duration Score (mITT) – Mixed Effects, Transformed, Weeks 2-26, with Imputation |
| Table 325: | PSQI Sleep Disturbance Score (mITT) – Mixed Effects, Transformed, Weeks 24 + 26, with Imputation |
| Table 326: | PSQI Sleep Disturbance Score (mITT) – Mixed Effects, Transformed, Weeks 2-26, No Imputation |
| Table 327: | PSQI Sleep Disturbance Score (mITT) – Mixed Effects, Transformed, Weeks 2-26, with Imputation |
| Table 328: | PSQI Use of Sleep Medication Score (mITT) – Mixed Effects, Transformed, Weeks 24 + 26, with Imputation |
| Table 329: | PSQI Use of Sleep Medication Score (mITT) – Mixed Effects, Transformed, Weeks 2-26, No Imputation |
| Table 330: | PSQI Use of Sleep Medication Score (mITT) – Mixed Effects, Transformed, Weeks 2-26, with Imputation |
| Table 331: | PSQI Daytime Dysfunction Score (mITT) – Mixed Effects, Transformed, Weeks 24 + 26, with Imputation |
| Table 332: | PSQI Daytime Dysfunction Score (mITT) – Mixed Effects, Transformed, Weeks 2-26, No Imputation |
| Table 333: | PSQI Daytime Dysfunction Score (mITT) – Mixed Effects, Transformed, Weeks 2-26, with Imputation |
| Table 334: | BAI Score (mITT) – Mixed Effects, Transformed, Weeks 24 + 26, with Imputation 171 |
| Table 335: | BAI Score (mITT) – Mixed Effects, Transformed, Weeks 2-26, No Imputation |
| Table 336: | BAI Score (mITT) – Mixed Effects, Transformed, Weeks 2-26, with Imputation |
| Table 337: | BDI-II Score (mITT) – Mixed Effects, Transformed, Weeks 24 + 26, with Imputation 171 |
| Table 338: | BDI-II Score (mITT) – Mixed Effects, Transformed, Weeks 2-26, No Imputation 172 |
| Table 339: | BDI-II Score (mITT) – Mixed Effects, Transformed, Weeks 2-26, with Imputation 172 |

| Table 340: | Subjects with No Heavy Drinking Days by MINI Withdrawal (mITT) – Logistic Regression, Weeks 22-25, with Imputation <sup>a</sup> |
|---|---|
| Table 341: | Subjects with No Heavy Drinking Days by BAI (mITT) – Logistic Regression, Weeks 22-25, with Imputation |
| Table 342: | Subjects with No Heavy Drinking Days by BAI (mITT) – Logistic Regression, Weeks 22-25, with Imputation |
| Table 343: | Subjects with No Heavy Drinking Days by PSQI Total Score (mITT) – Logistic Regression, Weeks 22-25, with Imputation |
| Table 344: | Subjects with No Heavy Drinking Days by Smoking Status (mITT) – Logistic Regression, Weeks 22-25, with Imputation |
| Table 345: | Subjects with No Heavy Drinking Days by POMS Total Mood Disturbance (mITT) – Logistic Regression, Weeks 22-25, with Imputation |
| Table 346: | Subjects with No Heavy Drinking Days by POMS Tension-Anxiety (mITT) – Logistic Regression, Weeks 22-25, with Imputation |
| Table 347: | Subjects with No Heavy Drinking Days by POMS Depression-Dejection (mITT) – Logistic Regression, Weeks 22-25, with Imputation |
| Table 348: | Subjects with No Heavy Drinking Days by POMS Confusion-Bewilderment (mITT) – Logistic Regression, Weeks 22-25, with Imputation |
| Table 349: | Subjects with No Heavy Drinking Days by POMS Vigor-Anxiety (mITT) – Logistic Regression, Weeks 22-25, with Imputation |
| Table 350: | Subjects with No Heavy Drinking Days by POMS Anger-Hostility (mITT) – Logistic Regression, Weeks 22-25, with Imputation |
| Table 351: | Subjects with No Heavy Drinking Days by POMS Fatigue-Inertia (mITT) – Logistic Regression, Weeks 22-25, with Imputation |
| Table 352: | Subjects with No Heavy Drinking Days by ACQ-SR-R (mITT) – Logistic Regression, Weeks 22-25, with Imputation |
| Table 353: | Subjects with No Heavy Drinking Days by Number of Days Abstinent from Alcohol (7 Days Prior to Randomization) (mITT) – Logistic Regression, Weeks 22-25, with Imputation |
| Table 354: | Subjects with No Heavy Drinking Days by Years Drinking Regularly (mITT) – Logistic Regression, Weeks 22-25, with Imputation |
| Table 355: | Subjects with No Heavy Drinking Days by Drinks per Week (28 Days Prior to Screening) (mITT) – Logistic Regression, Weeks 22-25, with Imputation |
| Table 356: | Subjects with No Heavy Drinking Days by Reducer Status (Change in Drinks per Day) (mITT) – Logistic Regression, Weeks 22-25, with Imputation |
| Table 357: | Subjects with No Heavy Drinking Days by Drinking Goal (mITT) – Logistic Regression, Weeks 22-25, with Imputation |
| Table 358: | Subjects with No Heavy Drinking Days by Total Dose (mITT) – Logistic Regression, |

| | Weeks 22-25, with Imputation | 174 |
|---|---|---|
| Table 359: | Subjects with No Heavy Drinking Days by BIS (mITT) – Logistic Regression, W 25, with Imputation | |
| | List of Listings | |
| Listing 1. Sul | bject Disposition - All Subjects | 176 |
| Listing 2. En | rollment and Randomization – All Consented Subjects | 176 |
| Listing 3. Re | ason not Eligible – Screen Failures | 177 |
| Listing 4. Pro | otocol Deviations – mITT Subjects | 177 |
| Listing 5. Sul | bjects Excluded from the Efficacy Analysis or Evaluable Set | 178 |
| Listing 6. De | mographics Data – mITT Subjects | 179 |
| Listing 7. Ba | seline Drinking Characteristics – mITT Subjects | 180 |
| Listing 8. Ba | seline Smoking Characteristics – mITT Subjects | 181 |
| Listing 9. Far | mily Members with History of Alcohol Problems | 181 |
| Listing 10. M | IINI DSM5 Disorders – mITT Subjects | 182 |
| Listing 11. M | IINI DSM5 AUD – mITT Subjects | 182 |
| Listing 12. M | Iedical History – mITT Subjects | 183 |
| Listing 13. D | rinking Treatment History mITT | 184 |
| Listing 14. D | rinking Goal - mITT Subjects | 184 |
| Listing 15. S | urgical History – mITT Subjects | 185 |
| Listing 16. Pl | hysical Exam – mITT Subjects | 185 |
| Listing 17. D | aily and Weekly Standard Drink Units (TLFB) During Treatment | 186 |
| Listing 18. D | rinking Question – mITT Subjects | 186 |
| Listing 19. D | rinking Consequences, Craving, Impulsiveness, Anxiety and Depression Scores | 186 |
| Listing 20. P | ittsburg Sleep Quality Index Scores | 187 |

| Listing 21. | Smoking Data-mITT Subjects | 187 |
|---|---|---|
| Listing 22. | PEth Levels – mITT Subjects | 187 |
| Listing 23. | MINI AUD End of Study – mITT Subjects | 188 |
| Listing 24. | Exit Interview – mITT Subjects | 189 |
| Listing 25. | Other Services Use – mITT Subjects | 190 |
| Listing 26. | Blood for DNA and RNA Testing – mITT Subjects | 191 |
| Listing 27. | Drug Exposure – mITT Subjects | 191 |
| Listing 28. | Adverse Events - mITT Subjects | 192 |
| Listing 29. | Serious Adverse Events - mITT Subjects | 193 |
| Listing 30. | POMS Scores | 194 |
| Listing 31. | Columbia-Suicide Severity Scale – mITT Subjects | 195 |
| Listing 32. | Blood Chemistries – mITT Subjects | 197 |
| Listing 33. | Pregnancy Test/Birth Control Data – mITT Subjects | 197 |
| Listing 34. | Blood Alcohol Concentration – mITT Subjects | 198 |
| Listing 35. | Urine Drug Screen | 198 |
| Listing 36. | Vital Signs and Body Weights-mITT Subjects | 199 |
| Listing 37. | ECG – mITT Subjects | 199 |
| Listing 38. | Prior and Concomitant Medications – mITT Subjects | 200 |
| Listing 39. | Comments – mITT Subjects | 200 |
| | List of Figures | |
| Figure 1: | Percentage of Subjects No Heavy Drinking Days Weeks 22-25 with Imputation | 201 |
| Figure 2: | Percentage of Subjects Abstinent Weeks 22-25 No Imputation | 202 |
| Figure 3: | Percentage of Subjects with WHO 1-Level Decrease in Alcohol Consumption Weeks 25 No Imputation | |
| Figure 4: | Percentage of Subjects with WHO 2-Level Decrease in Alcohol Consumption Weeks 25 No Imputation | |
| Figure 5: | Weekly Percentage of Subjects No Heavy Drinking Days with Imputation (mITT) | 203 |
| Figure 6: | Monthly Percentage of Subjects No Heavy Drinking Days with Imputation (mITT) | 203 |
| Figure 7: | Weekly Percentage of Subjects Abstinent with Imputation (mITT) | 203 |
| Figure 8: | Monthly Percentage of Subjects Abstinent with Imputation (mITT) | 203 |

| Figure 9: | Weekly Percentage WHO 1-Level Decrease in Alcohol Consumption No Imputation (mITT) | 204 |
|---|---|---|
| Figure 10: | Monthly Percentage WHO 1-Level Decrease in Alcohol Consumption No Imputation (mITT) | 204 |
| Figure 11: | Weekly Percentage WHO 2-Level Decrease in Alcohol Consumption No Imputation (mITT) | 204 |
| Figure 12: | Monthly Percentage WHO 2-Level Decrease in Alcohol Consumption No Imputation (mITT) | 204 |
| Figure 13: | Cumulative Grace Periods for Percentage of Subjects No Heavy Drinking Days with Imputation (mITT) | 204 |
| Figure 14: | Cumulative Grace Periods for Percentage of Subjects Abstinent No Imputation (mITT) | 204 |
| Figure 15: | Cumulative Grace Periods for Percentage WHO 1-Level Decrease in Alcohol Consumption no Imputation (mITT) | 204 |
| Figure 16: | Cumulative Grace Periods for Percentage WHO 2-Level Decrease in Alcohol Consumption no Imputation (mITT) | 204 |
| Figure 17: | Percentage Days Abstinent per Week Least Squares Means – (Untransformed) no Imputation (mITT) | 205 |
| Figure 18: | Percent Heavy Drinking Days per Week Lease Squares Means – (Untransformed) no Imputation (mITT) | 205 |
| Figure 19: | Mean Drinks per Week Lease Squares Means – (Untransformed) no Imputation (mITT) | 205 |
| Figure 20: | Mean Drinks per Drinking Day by Week Least Squares Means – (Untransformed) no Imputation (mITT) | 205 |
| Figure 21: | Weekly Number of Cigarettes Smoked in Smokers Over Entire Maintenance Period – Least Squares Means no Imputation (mITT) | 205 |
| Figure 22: | ACQ-SR-R Score by Visit Least Squares Means – (Untransformed) no Imputation (mIT | T)205 |
| Figure 23: | ImBIBe Score by Visit Least Squares Means – (Untransformed) no Imputation (mITT) | 205 |
| Figure 24: | PSQI Score by Visit Least Squares Means – (Untransformed) no Imputation (mITT) | 205 |
| Figure 25: | PSQI Sleep Quality Score by Visit Least Squares Means – (Untransformed) no Imputation (mITT) | |
| Figure 26: | PSQI Sleep Latency Score by Visit Least Squares Means – (Untransformed) no Imputat (mITT) | |
| Figure 27: | PSQI Sleep Duration Score by Visit Least Squares Means – (Untransformed) no Imputation (mITT) | 205 |
| Figure 28: | PSQI Sleep Disturbanced Score by Visit Least Squares Means – (Untransformed) no Imputation (mITT) | 205 |
| Figure 29: | PSQI Use of Sleep Medication Score by Visit Least Squares Means – (Untransformed) Imputation (mITT). | |

| Figure 30: | PSQI Daytime Dysfuction Score by Visit Least Squares Means – (Untransformed) no Imputation (mITT) | 205 |
|---|---|---|
| Figure 31: | BAI by Visit Least Squares Means – (Untransformed) no Imputation (mITT) | 205 |
| Figure 32: | BDI-II by Visit Least Squares Means – (Untransformed) no Imputation (mITT) | 205 |
| Figure 33: | ROC BAI by PSNHDD Weeks 22-25 (mITT) | 205 |
| Figure 34: | ROC BDI-II by PSNHDD Weeks 22-25 (mITT) | 205 |
| Figure 35: | ROC PSQI Total Score by PSNHDD Weeks 22-25 (mITT) | 205 |
| Figure 36: | ROC POMS Total Score by PSNHDD Weeks 22-25 (mITT) | 206 |
| Figure 37: | ROC POMS Tension-Anxiety by PSNHDD Weeks 22-25 (mITT) | 206 |
| Figure 38: | ROC POMS Depression-Dejection by PSNHDD Weeks 22-25 (mITT) | 206 |
| Figure 39: | ROC POMS Vigor-Activity by PSNHDD Weeks 22-25 (mITT) | 206 |
| Figure 40: | ROC POMS Fatigue-Inertia by PSNHDD Weeks 22-25 (mITT) | 206 |
| Figure 41: | ROC POMS Anger-Hostility by PSNHDD Weeks 22-25 (mITT) | 206 |
| Figure 42: | ROC POMS Confusion-Bewilderment by PSNHDD Weeks 22-25 (mITT) | 206 |
| Figure 43: | ROC ACQ-SR-R by PSNHDD Weeks 22-25 (mITT) | 206 |
| Figure 44: | ROC Days Abstinent (7 Days Prior to Randomization) by PSNHDD Weeks 22-25 (mI | TT)206 |
| Figure 45: | ROC Years Drinking Regularly by PSNHDD Weeks 22-25 (mITT) | 206 |
| Figure 46: | ROC Drinks per Week by PSNHDD Weeks 22-25 (mITT) | 206 |
| Figure 47: | ROC Reducer by PSNHDD Weeks 22-25 (mITT) | 206 |
| Figure 48: | ROC BIS by PSNHDD Weeks 22-25 (mITT) | 206 |
| Figure 49: | ROC Total Dose by PSNHDD Weeks 22-25 (mITT) | 206 |
| Figure 50: | Clinical Chemistry Values Over Time | 206 |

# 1. ABBREVIATIONS

| Abbreviation | Definition |
|---|---|
| ACQ-SR-R | Alcohol Craving Scale – Short Form |
| AE | Adverse event |
| AICc | Akaike Information Criterion corrected for finite samples |
| ALT | Alanine aminotransferase |
| AST | Aspartate aminotransferase |
| AUC | Area under the concentration time curve |
| AUD | Alcohol Use Disorder |
| BAC | Blood alcohol concentration |
| BAI | Beck Anxiety Inventory |
| BDI-II | Beck Depression Inventory-II |
| BID | Twice daily |
| BIS | Barratt Impulsiveness Scale |
| CFR | Code of Federal Regulations |
| CI | Confidence interval |
| CIWA-AR | Clinical Institute Withdrawal Assessment for Alcohol-revised |
| CrCl | Creatinine clearance |
| C-SSRS | Columbia-Suicide Severity Rating Scale |
| CTCAE | Common terminology criteria for adverse events |
| dL | Deciliter |
| DNA | Deoxyribonucleic acid |
| DSM-5 | Diagnostic and Statistical Manual of Mental Disorders - Fifth Edition |
| DSMB | Data and Safety Monitoring Board |
| ECG | Electrocardiogram |
| eCRF | Electronic Case Report Form |
| EDMS | Electronic Data Management System |
| EOS | End of study |
| F | Fahrenheit |
| FDA | Food and Drug Administration |
| g | Gram |
| GCP | Good Clinical Practice |
| GGT | Gamma-glutamyl transferase |
| hr | Hour |
| ICH | International Conference on Harmonization |
| IRB | Institutional Review Board |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mg | Milligram |
| μg | Microgram |
| min | Minutes |

| Abbreviation | Definition |
|--------------|-----------------------------------------------------|
| MINI | MINI Neuropsychiatric Interview |
| mITT | Modified intention-to-treat |
| mL | Milliliter |
| mm | Millimeter |
| NHDD | No heavy drinking days |
| NIAAA | National Institutes on Alcohol Abuse and Alcoholism |
| OZ | Ounce |
| PD | Pharmacodynamic |
| PEth | Phosphatidylethanol |
| PK | Pharmacokinetic |
| POMS | Profile of Mood State |
| PSNHDD | Percentage of subjects with no heavy drinking days |
| PSQI | Pittsburg Sleep Quality Index |
| PT | Preferred term |
| RNA | Ribonucleic acid |
| ROC | Receiver Operator Curve |
| SAE | Serious adverse event |
| SAP | Statistical analysis plan |
| SD | Standard deviation |
| SDU | Standard drinking unit |
| SOC | System Organ Class |
| THC | Tetrahydrocannabinol |
| TLFB | Timeline followback |
| ULN | Upper limit of normal |
| WHO | World Health Organization |

#### 2. INTRODUCTION

This statistical analysis plan (SAP) for Protocol No. NCIG-006, "Randomized, Double Blind, Placebo-Controlled Trial of the Safety and Efficacy of HORIZANT® (Gabapentin Enacarbil) Extended-Release Tablets for the Treatment of Alcohol Use Disorder" describes and expands upon the analytical plan presented in the protocol.

This document contains all planned analyses, reasons and justifications for these analyses for all study data with the exception of the pharmacokinetics data. The population pharmacokinetic/pharmacodynamic (PK/PD) analysis will be described in a separate population PK/PD analysis plan that will be authored and performed by XenoPort, Inc. This plan also includes sample tables, figures, and listings that will be populated. The SAP will follow the International Conference on Harmonization of Technical Requirements for Registration of Pharmaceuticals for Human Use (ICH) Guidelines as indicated in Topic E3 (Structure and Content of Clinical Study Reports), Topic E8 (General Considerations for Clinical Trials) and Topic E9 (Statistical Principles for Clinical Trials). The structure and content of the SAP provides sufficient detail to meet the requirements identified by the FDA and ICH.

The following sources were used in preparation of this SAP:

- Protocol # NCIG-006, Protocol Version No.: 3.0; Version Date: 18 May 2015
- ICH Guidance Topics E9, E3 and E8

#### 3. PROTOCOL SUMMARY

## 3.1. Study Objectives

### **3.1.1. Primary**

The primary objective of the study is to compare the efficacy of HORIZANT (gabapentin enacarbil) Extended-Release Tablets 600 mg twice daily (BID) with matched placebo on the primary alcohol consumption outcome endpoint, percentage of subjects with no heavy drinking days (PSNHDD) during the last 4 weeks of treatment, among patients with Alcohol Use Disorder (AUD). PSNHDD will also be analyzed during other time periods (i.e., the last 8, 12, 16, 20, and 24 weeks of the maintenance period) in exploratory analyses (see 9.11.4).

# 3.1.2. Secondary

Secondary objectives are separated into two categories: key secondary and supportive secondary. The key secondary objective is to compare HORIZANT to placebo on the percentage of subjects abstinent from alcohol during the last 4 weeks of treatment. The supportive secondary study objectives are to assess other treatment benefits including: reduction in other alcohol consumption endpoints, alcohol-related craving and consequences, mood, sleep quality, smoking quantity and frequency, and safety.

# 3.2. Study Design

This study is a double-blind, randomized, placebo-controlled, parallel group, multi-site study designed to assess the efficacy of HORIZANT Extended-Release Tablets compared with placebo to reduce drinking in 346 subjects (173 in each group) who report 4 or more Diagnostic and Statistical Manual of Mental Disorders – Fifth Edition (DSM-5<sup>TM</sup>) symptoms of AUD and who meet the drinking criteria outlined hereafter. This study will be conducted at 10 clinical sites. If eligible for the study, subjects will be randomized using a stratified permuted block randomization procedure with "clinical site" as the stratification variable in an approximate 1:1 ratio (targeting 173 subjects per group) to receive either HORIZANT Extended-Release Tablets or placebo for 26 weeks (1 week escalation; 24 weeks maintenance; 1 week taper).

Subjects will be seen in the clinic at screening, at randomization and 11 other times during the study. During the Week 1 dose escalation period (midway through the week) and during the maintenance period (Weeks 2 to 25), subjects will be contacted once per week by telephone at non-clinic visit weeks to encourage study drug compliance and to assess withdrawal, adverse events (AEs), and concomitant medications. A final follow-up telephone interview will occur during Weeks 28 to 29 (1 to 2 weeks after the end of dosing).

An overview of the study design is provided in **Figure 1**. Study assessments and procedures will be performed at the visits and time points outlined in the Schedule of Assessments (**Table 1**).

Figure 1: Overview of Study Design



**Table 1:** Schedule of Assessments

| | Scre | een | Ti-<br>trate | | | | | | | | | Mair | itenan | ce | | | | | | | | Taper | | Safety<br>Follow-<br>up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Clinic Visit # | 0 | 1 | | 2 | | 3 | | 4 | | 5 | | 6 | | 7 | | 8 | | 9 | | 10 | | 11 | 12 | |
| Study Week | -2 to -1 | Day<br>-1 | 1 | 2 | Mid<br>week 2<br>& 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 -<br>15 | 16 | 17-<br>19 | 20 | 21-<br>23 | 24 | 25 | 26 | EOS <sup>a</sup> /27 | 28-<br>29 |
| Informed Consent | X | | | | | | | | | | | | | | | | | | | | | | | |
| Alcohol Breathalyzer | X | X | | X | | X | | X | | X | | X | | X | | X | | X | | X | | X | X | |
| Urine Drug Screen <sup>b</sup> | X | X | | X | | X | | X | | X | | X | | X | | X | | X | | X | | X | X | |
| Locator Form | X | | | | | | | | | | | | | | | | | | | | | | | |
| Demographics | X | | | | | | | | | | | | | | | | | | | | | | | |
| Medical History | X | X | | | | | | | | | | | | | | | | | | | | | | |
| Physical Exam | X | X | | | | | | | | | | | | | | | | | | | | | X | |
| MINI V 7.0 | X | | | | | | | | | | | | | | | | | | | | | x | | |
| Clinical Chemistry d | X | | | | | X | | | | X | | | | X | | X | | X | | X | | X | X | |
| Vital Signs | X | X | | | | X | | | | X | | | | X | | X | | X | | X | | X | X | |
| ECG | X | | | | | | | | | | | | | | | | | | | | | | X | |
| Prior and Concomitant<br>Meds | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| CIWA-AR | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | |
| Eligibility Checklist | X | X | | | | | | | | | | | | | | | | | | | | | | |
| Blood for DNA Genomics Testing f | | X | | | | | | | | | | | | | | | | | | | | | | |
| Blood for RNA<br>Expression Testing | | X | | | | | | | | | | | | | | | | | | X | | | | |
| Blood for PK/Medication<br>Compliance | | | | | | | | | | | | | | X | | | | X | | X | | | | |
| Blood spot for PEth | | X | | | | | | | | | | | | | | | | | | | | X | | |
| Drug compliance/<br>accountability | | | | X | | X | | X | | X | | X | | X | | X | | X | | X | | X | X | |

| | Scre | een | Ti-<br>trate | | | | | | | | | Mair | ntenan | ce | | | | | | | | Taper | | Safety<br>Follow-<br>up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Clinic Visit # | 0 | 1 | | 2 | | 3 | | 4 | | 5 | | 6 | | 7 | | 8 | | 9 | | 10 | | 11 | 12 | |
| Study Week | -2 to -1 | Day<br>-1 | 1 | 2 | Mid<br>week 2<br>& 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 -<br>15 | 16 | 17-<br>19 | 20 | 21-<br>23 | 24 | 25 | 26 | EOS <sup>a</sup> /27 | 28-<br>29 |
| Pregnancy Test + birth control | X | X | | | | X | | | | X | | | | X | | X | | X | | X | | | X | |
| Weight | X | ζ. | | | | | | | | | | | | | | X | | | | | | | X | |
| Drinking Goal | | X | | | | | | | | | | | | | | | | | | | | | | |
| AEs | $\mathbf{X}^{\mathrm{h}}$ | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| C-SSRS | | X | | X | | X | | X | | X | | X | | X | 14 | X | 18 | X | 22 | X | | X | X | |
| RANDOMIZATION | | X | | | | | | | | | | | | | | | | | | | | | | |
| Brief Telephone<br>Interview | | | X | | X | | X | | X | | X | | X | | X | | X | | X | | X | | | |
| Take Control | | X | | X | | X | | X | | X | | X | | X | | X | | X | | X | | X | | |
| Exit Interview | | | | | | | | | | | | | | | | | | | | | | | X | |
| Treatment Referral | | | | | | | | | | | | | | | | | | | | | | | X | |
| Follow-Up Telephone<br>Interview | | | 7 | | | | | | | | | | | | | | | | | | | | | X |
| Final Subject Disposition | | | | | | | | | | | | | | | | | | | | | | | | X |
| Subject Reported<br>Outcomes | | | | | | | | | | | | | | | | | | | | | | | | |
| Family History of Alcohol Problems | | X | | | | | | | | | | | | | | | | | | | | | | |
| BIS | | X | | | | | | | | | | | | | | | | | | | | X | | |
| ImBIBe | | X | | | | X | | | | X | | | | X | | X | | X | | X | | X | | |
| TLFB | X | X | | X | | X | | X | | X | | X | | X | | X | | X | | X | | X | X | |
| Drinking question j | | | | X | | X | | X | | X | | X | | X | | X | | X | | X | | X | X | |
| ACQ-SR-R | | X | | X | | X | | X | | X | | X | | X | | X | | X | | X | | X | | |
| Fagerström Test for<br>Nicotine Dependence | | X | | | | | | | | | | | | | | | | | | | | | | |
| Smoking quantity/frequency | | X | | X | | X | | X | | X | | X | | X | | X | | X | | X | | X | X | |

| | Scre | een | Ti-<br>trate | | Maintenance | | | | | | | | | | | | Taper | | Safety<br>Follow-<br>up | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Clinic Visit # | 0 | 1 | | 2 | | 3 | | 4 | | 5 | | 6 | | 7 | | 8 | | 9 | | 10 | | 11 | 12 | |
| Study Week | -2 to -1 | Day<br>-1 | 1 | 2 | Mid<br>week 2<br>& 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 -<br>15 | 16 | 17-<br>19 | 20 | 21-<br>23 | 24 | 25 | 26 | EOS <sup>a</sup> /27 | 28-<br>29 |
| PSQI | | X | | | | X | | | | X | | | | X | | X | | X | | X | | X | | |
| BAI | | X | | | | X | | | | X | | | | X | | X | | X | | X | | X | | |
| BDI-II | | X | | | | X | | | | X | | | | X | | X | | X | | X | | X | | |
| POMS | | X | | | | X | | | | X | | | | X | | X | | X | | X | | X | | |
| Other Services Used for<br>Alcohol Use Problems | | X | | | | X | | | | X | | | | X | | X | | X | | X | | | X | |

<sup>&</sup>lt;sup>a</sup>EOS=end of study. These assessments are to be done at Week 27 or if the subject discontinues early and agrees to a final clinic visit.

<sup>&</sup>lt;sup>b</sup>Test for opioids, cocaine, amphetamines, methamphetamine, tetrahydrocannabinol (THC), buprenorphine, methadone or benzodiazepines.

<sup>&</sup>lt;sup>c</sup>Only the AUD module is performed at Week 26.

<sup>&</sup>lt;sup>d</sup>Aspartate aminotransferase (AST), alanine aminotransferase (ALT), total bilirubin, creatinine, and gamma glutamyltransferase (GGT).

<sup>&</sup>lt;sup>e</sup>Sitting blood pressure and heart rate.

<sup>&</sup>lt;sup>f</sup>Only for subjects who consent to provide this sample.

<sup>&</sup>lt;sup>g</sup>For each subject, blood collections should be scheduled at different times relative to the morning dose at these 3 clinic visits.

<sup>&</sup>lt;sup>h</sup>Only serious adverse events (SAEs) will be reported from the time of signing informed consent until the first dose of investigational product administration. Thereafter, AEs and SAEs will be reported for the duration of the study.

<sup>&</sup>lt;sup>i</sup>AEs, concomitant medications, CIWA-AR, and drug compliance reminder.

<sup>&</sup>lt;sup>j</sup>Only asked to subjects who are no longer participating in clinic visits and not willing to providing TLFB drinking data.

#### 3.3. Study Endpoints

#### 3.3.1. Primary Efficacy Endpoint

The primary efficacy endpoint examines the hypothesis that HORIZANT Extended-Release Tablets will increase the percentage of subjects with no heavy drinking days (PSNHDD) compared to placebo during the last 4 weeks of maintenance period of treatment (Study Weeks 22-25). A "heavy drinking day" is 4 or more drinks per drinking day for women and 5 or more drinks per drinking day for men. PSNHDD will also be analyzed during other time periods (i.e., the last 8, 12, 16, 20, and 24 weeks of the maintenance period) in exploratory analyses (see 9.11.4). In all of these analyses, a different "grace peiod" is being explored.

## 3.3.2. Secondary Efficacy Endpoints

Secondary endpoints will be analyzed over the last 4 weeks of the maintenance phase of treatment.

- 1. Percentage of subjects abstinent from alcohol (key secondary endpoint)
- 2. Percentage of subjects with a World Health Organization (WHO) drinking risk category decrease of:
  - a at least 1-level
  - b. at least 2-levels
- 3. Percentage of days abstinent per week
- 4. Percentage of heavy drinking days per week
- 5. Weekly mean number of drinks per week
- 6. Weekly mean drinks per drinking day
- 7. Cigarettes per week among smokers
- 8. Alcohol craving score [Alcohol Craving Scale Short Form (ACQ-SR-R)]
- 9. Alcohol related consequences (ImBIBe) score
- 10. Pittsburg Sleep Quality Index (PSQI) score
- 11. Beck Anxiety Inventory (BAI) score
- 12. Beck Depression Inventory Scale II (BDI-II) score

#### 3.3.3. Safety Endpoints

- 1. Vital signs
- 2. Blood chemistries
- 3. Urine drug screen results
- 4. Blood alcohol concentration (BAC) by breathalyzer
- 5. AEs

- 6. Electrocardiogram (ECG) results
- 7. Clinical Institute of Withdrawal Alcohol Revised (CIWA-AR) scores
- 8. Profile of Moods States (POMS) scores
- 9. Frequency of subjects with suicidal ideation at any time during the treatment period Columbia-Suicide Severity Rating Scale (C-SSRS)

#### 3.3.4. Compliance

Compliance will be assessed by self report of compliance with investigational products and gabapentin plasma levels. Compliance will be calculated as the percentage of medication taken as prescribed.

#### 3.3.5. Pharmacokinetics

A population PK/PD analysis will be performed using gabapentin plasma levels determined from blood samples collected at Weeks 12, 20, and 24 from subjects in the HORIZANT Extended-Release Tablets group. There will be a separate population PK/PD SAP that addresses this analysis.

#### 3.3.6 Exploratory Endpoints

- 1. Percentage of subjects abstinent from smoking
- 2. Number of symptoms observed in the MINI AUD scale
- 3. Blood PEth levels
- 4. PSNHDD, percentage subjects abstinent from alcohol, percentage of subjects with a WHO- 1-level decrease, and WHO 2-level decrease in alcohol consumption on a weekly and monthly basis, and across all grace periods, with and without imputation (exclusive of the primary endpoint)
- 5. All secondary endpoints with imputation
- 6. Moderators of PSNHDD during Weeks 22-25

#### 4. **DEFINITION OF ANALYSIS SETS**

The study analysis populations will consist of the following:

**Modified Intention-to-Treat (mITT) Analysis Set:** The mITT set is defined as subjects randomized to participate in the study who took at least one dose of investigational product.

**Evaluable Analysis Set:** The evaluable analysis set is defined as those subjects randomized to the study who took at least 80% of the prescribed dose of tablets during the maintenance period (Weeks 2 - 25) and did not have a major protocol violation.

The analysis of the primary and secondary efficacy endpoints will be conducted on both the mITT and evaluable analysis sets. Exploratory analyses will be performed on the mITT analysis set, unless otherwise specified. Safety analyses will be conducted on the mITT analysis set.
#### 5. ASSSESSMENT AND JUSTIFICATION OF STUDY ENDPOINTS

## 5.1. Alcohol Consumption Endpoints

#### 5.1.1. Daily Quantity of Alcohol Consumption

Drinking will be assessed using the TLFB methodology and Form 90 structured assessment pattern chart. The TLFB is a semi-structured interview that provides estimates of the daily quantity of alcohol consumption during specified time periods. It uses a calendar prompt and a number of other memory aids (e.g., holidays, payday, and other personally relevant dates) to facilitate accurate recall of drinking or other drug use during the target period. The procedure has been widely used in clinical and research contexts. It has demonstrated adequate levels of reliability and validity when administered as an in-person interview, over the telephone, and when administered via computer (Carey-1997, Sobell et al-1988, Sobell et al-1996).

If a subject is withdrawn from the study early and is no longer participating in clinic visits or providing TLFB drinking data but is willing to be contacted by phone at the week most proximal to dropout, then they will be asked about any drinking and heavy drinking during the time since last contact. Phone calls will continue until the end of the treatment period, as deemed acceptable by the patient. The two questions cover whether the subject had any heavy drinking days or drinking days during the period covered.

## 5.1.2. Drinking Days

A drinking day is one calendar day in which the subject reported any alcohol consumption (i.e., > 0 standard drinking units [SDUs]). A standard drink contains approximately 0.6 fluid ounces (oz) of pure alcohol. The data given by the subjects on amount and type of alcoholic beverage(s) consumed will be converted to SDUs. Standard drink unit definitions are provided in **Table 2**.

#### **Table 2:** Standard Drink Unit Definitions

For Beer (~ 5% alcohol), the approximate number of SDUs in:

- 12 oz = 1.0
- 16 oz = 1.3
- 22 oz = 2.0
- 40 oz = 3.3

For malt liquor ( $\sim 7\%$  alcohol), the approximate number of SDUs in:

- 12 oz = 1.4
- 16 oz = 1.9
- 22 oz = 2.6
- 40 oz = 4.7

For table wine (~ 12% alcohol), the approximate number of SDUs in:

- 750 mL bottle = 250z = 5.0
- 5 oz glass = 1.0
- 10 oz glass = 2.0

### **Table 2:** Standard Drink Unit Definitions (Continued)

For 80 proof spirits ( $\sim 40\%$  alcohol), or hard liquor, the approximate number of SDUs in:

- 1.5 oz (mixed drink) = 1.0
- 16 oz (pint) = 11.0
- 25 oz ( a fifth)= 17.0
- 1.75 L (59 oz) = 39.0

## 5.1.3. Heavy Drinking Day

A heavy drinking day is defined as a day with 5 or more drinks (SDUs) for males and 4 or more drinks (SDUs) for females.

#### 5.1.4. Days at Risk

If a subject is being treated at an inpatient facility, is incarcerated, or otherwise under confinement, the days spent in under these conditions is considered a reduction in the days at risk for drinking and is deducted from the denominator in calculations of rates of drinking days.

# 5.1.5. Percentage of Subjects with No Heavy Drinking Days and Percentage of Subjects Abstinent from Alcohol

The percentage of subjects with no heavy drinking days is the number of subjects that have no heavy drinking days during the period of interest divided by the number of subjects with at least one day of non-missing drinking data during the period of interest, multiplied by 100.

The percentage of subjects abstinent from alcohol is calculated similarly, except the numerator is the number of subjects that have no drinking days during the period of interest.

## 5.1.6. Weekly Percentage of Heavy Drinking Days and Weekly Percentage of Days Abstinent

Weekly percentage of heavy drinking days is the number of heavy drinking days in a 7-day period divided by 7 then multiplied by 100. The TLFB permits capturing data in a subsequent visit if a visit is missed; however, if fewer than 7 days are observed then the denominator is the number of days observed in the 7-day period. At least 3 days in a week must be observed; otherwise, the week is considered missing.

Weekly percentage of days abstinent is similarly calculated by using the number of days abstinent instead of the number of heavy drinking days.

# 5.1.7. Weekly Mean Number of Drinks and Weekly Mean Number of Drinks per Drinking Day

Weekly mean number of drinks is the sum of SDUs calculated to the tenths over 7 calendar days divided by the number of days with non-missing data. The quotient is multiplied by 7. At least 3 days in a week must be observed; otherwise, the week is considered missing.

Weekly mean number of drinks per drinking days utilizes the same numerator, and the denominator is the number of days with greater than 0 SDUs. Weeks where all days within the week are abstinent are assigned a value of 0 for weekly drinks per drinking day.

## 5.1.8. World Health Organization Drinking Risk Categorical Scale

The WHO has developed a drinking risk categorical scale that can be used in a responder analysis approach to assess clinically relevant decreases in alcohol consumption (<u>Aubin et al-2015</u>). Two dichotomous endpoints will be analyzed: WHO 1-level and WHO 2-level decrease in alcohol consumption. The WHO 1-level and 2-level decrease endpoints are the percentage of subjects experiencing at least a 1-level or 2-level decrease in WHO levels of alcohol consumption, respectively, from the level at baseline (the period including the 28 days before screening) to the level during the last 4 weeks of the maintenance phase (Study Weeks 22-25). The WHO levels of average alcohol consumption per day are as follows:

| | Males | Females |
|----------------|------------|-----------|
| Low Risk | 1 to 40g | 1 to 20g |
| Medium Risk | 41 to 60g | 21 to 40g |
| High Risk | 61 to 100g | 41 to 60g |
| Very High Risk | 101+g | 61+g |

where 14g = 1 SDU (<u>WHO-2000</u>). In computing the alcohol consumption level, average drinks per day will be used, computed as the sum of all drinking in the 28 day period divided by the number of days with non-missing drinking data in that period. Abstinent subjects will be included in a separate "Abstinent" category. A subject must have at least 1 week of data during the last 4 weeks of the maintenance phase to be considered non-missing.

## 5.2. Alcohol-Related Craving, Consequences, and Withdrawal

Alcohol-related craving is measured using the ACQ-SR-R scale and alcohol-related consequences are measured using the ImBIBe and CIWA-AR scales.

The ACQ-SR-R contains 12-items adapted from the 47-item ACQ-NOW developed by Singleton et al (1994) to assess craving for alcohol among alcohol users in the current context (right now). There are 4 subscale scores for compulsivity, expectancy, purposefulness and emotionality. Each subscale has 3 items with each item having a 1 to 7 raw score (from strongly disagree to strongly agree). A subscale score is obtained by summing the raw scores for the 3 items and dividing by 3. Items 3, 8, and 11 are reverse keyed. A general craving index is derived by summing all items and dividing by 12. If an item is missing, then the number of items is reduced by the number missing, and the sum is only the sum of the answered items. At least 10 items must be endorsed for the general craving index of ACQ-SR-R to be considered non-missing (i.e., scored). Any subscale with a missing item will be considered missing.

ImBIBe is a 15-item questionnaire in which the subject responds on a 5-point scale responses to questions on the consequences of alcohol use. This scale was adapted from the Drinker Inventory of Consequences questionnaire based on FDA recommendations on patient reported outcomes (Miller & Tonigen-1995). The total score is the sum of the individual item scores. In order to account for missing items, the sum is the sum of the responses times 15 divided by the number of items endorsed.

The CIWA-AR modified telephone version is an adaptation for telephone administration of the CIWA-AR a brief 10-item measure used to provide a quantitative index of the severity of the alcohol withdrawal syndrome (Sullivan et al-1989). The CIWA-AR has been used both in clinical and research applications and has demonstrated both reliability and validity (Sellers et al-1992, Stuppaeck et al-1994). The total score is the sum of the individual item scores. Since this is an interview scale, no missing items are anticipated. A score  $\geq$  10 is considered an indication that the subject is undergoing alcohol withdrawal.

#### **5.3.** Mood

Mood will be measured with the POMS, BDI-II, and BAI.

The POMS measures dimensions of affect or mood (McNair and Heuchert-2005). It consists of 65 adjectives to which the subject responds according to a 5-point scale ranging from "not at all (0)" to "extremely (5)." Six subscale scores will be computed for items grouped as follows: Tension-Anxiety, Depression-Dejection, Anger-Hostility, Vigor-Activity, Fatigue-Inertia, and Confusion-Bewilderment. A Total Mood Disturbance score will also be computed which consists of the sum of Tension-Anxiety, Depression-Dejection, Anger-Hostility, Fatigue-Inertia, and Confusion-Bewilderment scores then subtracting the Vigor-Activity subscale score. A missing value within a subscale will be replaced by the average score of the answered items within the subscale; if 2 or more items within a subscale are missing then the entire subscale is missing (Macefield et al-2010).

The BDI-II is a 21-item multiple choice questionnaire that is used for measuring the severity of depression (Beck et al-1966). Each item is scored on a scale value of 0 to 3. The BDI-II score is computed by summing all items. If fewer than 4 items are missing, then the missing items are replaced by the average value of the answered items, rounded to the nearest whole number (Lipps et al-2010). If 4 or more items are missing then the BDI-II is not scored. The standardized cutoffs for depression severity are:

0–13: minimal depression

14–19: mild depression

20–28: moderate depression

29-63: severe depression

The BAI consists of 21 questions about how the subject has been feeling in the last week, expressed as common symptoms of anxiety (such as numbness and tingling, sweating not due to heat, and fear of the worst happening). This inventory was designed to minimize the overlap with depression scales (Beck et al-1988). Missing responses to items will be treated the same as the BDI-II. Each question has the same set of four possible answer choices. These are:

Not at all. (0 points)

Mildly: It did not bother me much. (1 point)

Moderately: It was very unpleasant, but I could stand it. (2 points)

Severely: I could barely stand it. (3 points)

The BAI score is computed by summing all items. The standardized cutoffs for anxiety severity are:

0-7: minimal level of anxiety

8-15: mild anxiety

16-25: moderate anxiety 26-63: severe anxiety

## 5.4. Sleep Quality

Sleep quality will be measured using the PSQI. The PSQI is a 19-item questionnaire with 6 subscales (subjective sleep quality, sleep latency, sleep duration, habitual sleep disturbances, use of sleep medication and day time dysfunction) (Buysse et al-1989). Each subscale is rated from 0 to 3 with the higher scores reflecting more severe sleep complaints. The addition of all the scores permits an analysis of the subject's overall sleep experience in the past 30 days. The lower the overall score, the better the person sleeps. The scale and scoring instructions from Buysse et al-1989 are provided in Appendix A. A score  $\geq 5$  is indictive of a sleep disturbance. If any of the items is missing, then the entire form is missing (i.e, overall score and subscale scores) for that evaluation (PSQI website).

#### 5.5. Alcohol Use Disorder (MINI Version 7 – DSM5)

The AUD module of the MINI specifies the severity of AUD into 3 categories based on the total number of symptoms to which the subject is coded "Yes" as follows:

Mild = 2 to 3 symptoms

Moderate = 4 to 5 symptoms

Severe = 6 or more symptoms

Subjects must have at least 4 symptoms to be eligible to participate in the study. The total number of symptoms being scored is 11. No imputation for missing values will be used.

## 5.6. Smokers and Cigarettes per Week

A quantity frequency interview at baseline and during treatment will include two questions to assess cigarette smoking behavior: 1) Over the past week, on how many days did you smoke cigarettes?, 2) On the days you smoked during the past week, how many cigarettes did you smoke on average?. At baseline subjects that answer "0" to question #1 are considered non-smokers for the study. Cigarettes per week is the answer to question #1 multiplied by the answer to question #2. No imputation for missing values will be used.

#### 6. HYPOTHESES TO BE TESTED

#### 6.1. Primary Efficacy Endpoint

It is hypothesized that HORIZANT Extended-Release Tablets, as compared to placebo, will increase the PSNHDD during Study Weeks 22 to 25 (last 4 weeks of the maintenance period). This hypothesis will be explored using other time periods (see 9.11.4).

## 6.2. Secondary Efficacy Endpoints

Over the last 4 weeks of the maintenance period, it is hypothesized that the HORIZANT Extended-Release Tablets group, as compared to the placebo group, will:

- 1. Increase the percentage of subjects abstinent from alcohol (key secondary endpoint)
- 2. Increase the percentage of subjects with a WHO drinking risk category decrease of::
  - a. at least 1-level
  - b. at least 2-levels
- 3. Increase the percentage of days abstinent per week
- 4. Decrease the percentage of heavy drinking days per week
- 5. Decease the weekly mean number of drinks per week
- 6. Decrease the weekly mean drinks per drinking day
- 7. Decrease the cigarettes per week among smokers
- 8. Decrease the alcohol craving score (ACQ-SR-R) per visit
- 9. Decrease the alcohol related consequences (ImBIBe) score per visit
- 10. Decrease PSQI score
- 11. Decrease the BAI score
- 12. Decrease the BDI-II score

## 6.3 Exploratory Efficacy Endpoints

The following exploratory endpoints will be examined to generate hypotheses or perform sensitivity analyses for hypotheses that the HORIZANT Extended-Release Tablets group, as compared to the placebo group, will:

- 1. Increase the percentage of subjects abstinent from smoking in subjects that were smokers at the start of the study
- 2. Decrease the number of symptoms observed in the MINI AUD scale
- 3. Decrease the blood PEth levels
- 4. Increase the PSNHDD, percentage of subjets abstinent from alcohol, percentage of subjects with a WHO- 1-level decrease, and a WHO 2-level decrease in alcohol consumption on a weekly and monthly basis, and across all grace periods, with and without imputation (exclusive of the primary endpoint)

- 5. Change all secondary endpoints, with imputation, in the direction listed in Section 6.2
- 6. Have a greater treatment effect on the primary endpoint during Weeks 22-25, among moderators suggestive of alcohol withdrawal and increased severity of alcohol use disorder.

#### 7. SAMPLE SIZE CONSIDERATIONS

The sample size was based on a conservative approach to the results of the randomized, placebo-controlled trial reported by Mason et al (2014). Mason et al (2014) found an effect size for PSNHDD of odds ratio = 2.8 (Cohen's h = 0.48). However, this study was a single site trial and single site trials are known to have greater effect sizes than multi-site trials (Feinn and Kranzler, 2005). Taking a conservative approach, we assumed a smaller effect size for the current multi-site trial, an odds ratio = 2.5; (Cohen's h=.34, that occurs given a placebo PSNHDD during Study Weeks 22-25 of 13% and an active study drug PSNHDD of 27%). To achieve 91% power for this trial, given a two-tailed alpha of 0.05, then a sample size of 173 per group (346 total) is needed (Fleiss et al-2003). The estimates of 13% and 27% for placebo and gabapentin, respectively, assumes 15% of the randomized subjects in each treatment group will dropout prior to or during the last 4 weeks of the Maintenance Period, and consequently, these dropouts will be imputed as subjects with heavy drinking days (i.e., treatment failures).

#### 8. DATA QUALITY ASSURANCE

Data quality assurance will start with training of clinical investigative staff on data collection and assessment procedures including a Manual of Operations that describes what data to collect and procedures for completion of eCRFs. Completed eCRFs will be reviewed by Fast-Track Drugs and Biologics clinical monitors on a regular basis throughout the trial by comparison against the source documents.

All study data will come from the eCRFs and no other source data. eCRFs for this study were created using an electronic data management system (EDMS) based on Merge eClinicalOS. eCRFs were created using an established data dictionary for each variable including the field name, field type, field attributes, and coding for variables. Range checks, alpha-numeric requirements, and null/not null parameters were programmed as applicable. The back end database application is Oracle. Data entered into the EDMS system will be reviewed by Fast-Track clinical monitors and data managers. If incomplete or inaccurate data are found, the data will be queried in the system for site staff to address. The site will resolve data inconsistencies and errors using the EDMS with full audit trail of corrections being maintained within the system. Corrections and changes to the data will be reviewed by Fast-Track clinical monitors and data managers.

Additional edit checks will be written to detect anomalies in the database. These checks will address inconsistencies (within visits, across visits), invalid/unusual values, missing values, and protocol violations. Edit checking will be validated on test data or actual clinical trial data. In addition to programmed edit checks, quality control examination of data will also be performed on reviews of data listings.

#### 9. STATISTICAL CONSIDERATIONS

#### 9.1. General Considerations

For descriptive purposes, dichotomous and categorical variables will be presented as number of observations and percentages; continuous variables will be given as means, standard deviations (SD), median, miniumum (min) and maximum(max). Statistical tests will be two-tailed at a 0.05 Type I error rate. P-values for the primary and secondary endpoints of < 0.05 will be considered statistically significant. Endpoint data will also be screened for outliers and skewness. Appropriate non-parametric tests will be used to compare treatment groups on continuous baseline characteristics that are not normally distributed. Continuous endpoint data that are not normally distributed will be transformed using either a square root, logarithmic, or inverse transformation, the selection of which is determined by skewness and kurtosis statistics with values closest to zero. Cohen's d will be used to calculate the effect size for means and Cohen's h will be used to calculate the effect size for proportions. Odds ratios will be provided for all dichotomous outcomes and coverted to Cohen's d when appropriate. Descriptive statistics — mean, SD, median, min and max — of all endpoint data will be presented in listings.

## 9.2. Participant Accountability and Protocol Deviations

A summary will be prepared to show dropouts/retention over time in each group, along with the reason for early termination. The number of missing observations will be presented between groups. Protocol deviations will be presented as summaries by type of deviation.

## 9.3. Demographics and Other Baseline Characteristics

Summaries of the characteristics of the subjects in each of the study groups at baseline will be prepared for the mITT, and evaluable analysis sets. Demographic characteristics (e.g., age, gender, race, ethnicity, marital status, employment, and education) and other baseline characteristics including Family History of Alcohol Problems, Barratt Impulsiveness scale (BIS), mood scales (e.g., Beck Anxiety Inventory (BAI), Beck Depression Inventory – II (BDI-II), Profile of Mood States (POMS) total and subscale scores), Pittsburg Sleep Quality Index (PSQI), and drinking goal (multiple choices and dichotomized total abstinence or not total abstinence) will be summarized by treatment group for the mITT and evaluable subjects.

Baseline drinking parameters in the 28-days prior to the start of screening, age started drinking regularly, medical treatments for drinking in the past year, and other services used for alcohol problems in the past 4 weeks prior to consent will be summarized by treatment group for the mITT subjects. The number and percentage of subjects with mild, moderate and severe symptoms of AUD and summary statistics for total number of symptoms will also be presented.

Nicotine dependence will be assessed using the modified Fagerstrom Test for Nicotine Dependence with responses to each question will be presented. A summary nicotine dependence score will be tabulated. The quantity of cigarettes smoked per week in the week prior to randomization will be presented for those subjects who reported any smoking. The numbers and percentages of subjects who test positive for THC will also be presented.

Baseline drinking-associated consequences (CIWA-AR and ImBIBe scores) and drinking-associated-craving (ACQ-SR-R) total score and subscales will be summarized in the tables.

Continuous variables will be summarized using means, standard deviations, medians, min, and maximum values. Categorical variables will be summarized using counts and percentages.

The comparability among the treatment groups with respect to the demographic and baseline variables will be evaluated by appropriate statistical methods. These will include t-tests for continuous variables, chi-square tests for categorical variables, and Fisher's exact test for binary variables. If a continuous variable is skewed, then the Wilcoxon rank sum test will be used on the raw data or a t-test on an appropriately transformed variable.

## 9.4. Efficacy Analysis

## 9.4.1. Primary Analysis of the Primary Efficacy Endpoint

The primary analysis of the primary efficacy endpoint will be conducted via a fully covaried logistic regression of PSNHDD during Study Weeks 22 to 25 (last 4 weeks of the maintenance period on the mITT population). The Wald statistic from the fully covaried logistic regression will be used to test for treatment differences. A two-tailed p-value < 0.05 will be considered statistically significant. A bar graph will present the results. Exploratory analyses will examine other timeframes beyond the last 4 weeks (see Section 9.11.4).

# 9.4.2. Covariate Adjustment for the Primary Analysis of the Primary Efficacy Endpoint

The logistic regression model will include treatment group, clinical site, pre-randomization drinking goal (abstinence versus not abstinent), and baseline percent heavy drinking days. Clinical site was deemed a covariate because it was chosen as a stratification variable to account for between site variability in outcome. Prior to conducting the logistic regression, a blinded analysis of site by treatment group by PSNHDD outcome will be performed to determine if every site has an outcome. Clinical sites with fewer than 3 events will be be combined for the purpose of conducting the logistic regression. The subject's pre-randomization goal for drinking outcome has been observed in prior studies as a predictor of reducing the frequency of heavy drinking days and will be included in this study as a dichotomized covariate. Baseline drinking is a strong predictor of drinking outcome, and thus will be included as a covariate. Since all subjects will have at least one heavy drinking day at baseline (thus preclusing the possibility of between subject variability on baseline PSNHDD), it was not possible to use baseline PSNHDD as a covariate of PSNHDD outcome. Thus, baseline percent heavy drinking days was chosen to be the covariate as a near-analgous measure of PSNHDD outcome.

## 9.4.3. Analysis of the Secondary Efficacy Endpoints

Secondary efficacy endpoints will also be analyzed based on data collected during the last 4 weeks of the maintenance period (Weeks 22 through 25), including TLFB and other questionnaire data assessed at Week 26 that reflect data collected during this period.

In general, every continuous secondary efficacy endpoint is analyzed using a repeated measures mixed effects model where subjects are random effects; factors and covariates are fixed effects. The analyses will be performed using SAS PROC MIXED procedure with the categorical or

dichotomous fixed effects variable having values ordered per the data. The information criterion is requested from every mixed effects model. Subjects are treated as a class variable and not continuous. The week (Weeks 22 through 25), treatment group, and clinical site are also treated as class variables.

The primary analysis model for all continuous endpoints is:

• Appropriately transformed endpoint = treatment + week + treatment\*week + clinical site + baseline equivalent of endpoint + other covariates (identified in Section 9.4.4)

This model will also be created for the untransformed endpoint. The solution statement from SAS PROC MIXED is requested to provide the solution for the fixed effects parameters. A REPEATED statement specifies that values are repeated each week and subjects are nested within treatment group. The covariance structure is specified.

The selection of the covariance structure is performed using a simple repeated mixed effects model that includes treatment group as the only fixed effect and subject nested within treatment group as the only random effect. The covariance structure for each continuous secondary endpoint is selected from autoregressive, compound symmetry, Toeplitz, and unstructured. The Akaike Information Criterion (AICc) corrected for a finite sample is obtained from each of the four models for the four possible covariance structures to determine model fit. The smallest (minimum) AICc associated with one of the covariance structurs is selected and the difference for each of the other three covariance structurs is calculated. A graph is produced of the model fit statistics and relative difference for the four possible covariance structures. The graphs across the continuous endpoints are compared to determine which covariance structure will be selected for all continuous endpoints or if one or more models need different covariance structures.

Results based on the primary analysis model and the model of the untransformed endpoint will be presented in tabular form. The overall least squares means and least square means for each time point along with the 95% confidence intervals will be presented for the untransformed endpoint only, while two-tailed p-values and Cohen's d will be presented for both the untransformed and transformed data. Inference and Cohen's d will be based upon the results using appropriately transformed data. Graphs of all secondary endpoints will be produced.

#### 9.4.3.1. Key Secondary Endpoint: Percentage of Subjects Abstinent

Percentage of subjects abstinent during Weeks 22 to 25 is the key secondary endpoint. The analysis will be performed as indicated in Section 9.4.4 and the two-tailed p-value from the fully covaried logistic regression will be evaluated if and only if the primary endpoint (PSNHDD) is statistically significant (p<0.05 [Section 9.4.1]). The testing procedure utilizes the serial gatekeeping methodology (Dmitrienko and Tamhane 2009). The key secondary endpoint can only be evaluated for statistical significance after the primary endpoint has been identified as statistically significant. In this situation, percentage of subjects abstinent will be evaluated using the Wald statistic from the logistic regression model at p<0.05 after PSNHDD is found to have p<0.05. If PSNHDD is not statistically significant at the 0.05 level then no significance testing of percentage of subjects abstinent will be performed. This analysis will be performed on mITT subjects with a drinking day imputed for missing data. However, if drinking data are missing by TLFB, but the subject reports any drinking during Weeks 22 to 25 using the Drinking Question

eCRF, then the subject will be considered not abstinent. An analysis of percent subjects abstinent without imputation for missing data will be performed as an exploratory analysis

## 9.4.3.2. Secondary Drinking Endpoints

Percentage of days abstinent per week, percentage of heavy drinking days per week, weekly mean number of drinks per week, and weekly mean number of drinks per drinking day will be analyzed using the mixed effects model specified in Section 9.4.3. Covariates for these models will be identified as in Section 9.4.4.

Percentage of subjects with a WHO 1-level decrease, and WHO 2-level decrease in alcohol consumption risk category will be analyzed during the last 4 weeks of the maintenance period (Weeks 22 through 25) using the same logistic regression model method and contingency table as defined for the primary endpoint in Sections 9.4.1 and 9.4.2. Covariates for these models will be identified as in Section 9.4.4.

## 9.4.3.3. Alcohol Consequences and Craving Scales

The ImBIBe and ACQ-SR-R scales are assessed at Study Weeks 24 and 26 which will be used for the secondary endpoints. Mixed effects models as stated in Section 9.4.3 will be generated for the total score for each of these scales and for the 4 subscales for the ACQ-SR-R. Covariates for these models will be identified as in Section 9.4.4.

#### 9.4.3.4. Smoking Quantity

The mean number of cigarettes smoked in the past week is measured at Study Weeks 24 and 26. The sample is the mITT subjects who smoked at baseline. The data will be analyzed as described in Section 9.4.3. Covariates for this endpoint will be identified in Section 9.4.4.

## 9.4.3.5. Depression, Anxiety, and Sleep Scales

The BDI-II total score, BAI total score, and PSQI total score (and subscale scores) are continuous variables. The secondary endpoints for the BDI-II, BAI, and PSQI subscales are assessed at Study Weeks 24 and 26. The data will be analyzed as described in Section 9.4.3. Covariates for these models will be identified as in Section 9.4.4.

#### 9.4.4. Covariate Adjustment for the Analysis of Secondary Efficacy Endpoints

Covariates for continuous secondary efficacy endpoints include the baseline equivalent of the endpoint, clinical site, treatment, time and the treatment by time interaction. Additional covariates for the secondary efficacy endpoints may include baseline characteristics with a theoretical and/or empirical basis for a relationship with a particular secondary endpoint. Such characteristics may include, but are not limited to, drinking goal (total abstinence versus less than total abstinence), age, years of regular drinking (age minus age first started drinking alcohol regularly), baseline alcohol craving scale total score. Prior to the unblinding of the data, matrices of correlations between these baseline characteristics and each of the secondary efficacy endpoints, pooled across blinded treatment assignment, will be produced (using Pearson for continuous variables, Spearman for categorical outcomes). Selection of baseline variables to include as covariates in the models will be based on consideration of the following criteria: at least modest correlation with outcome (i.e., r>0.20), and clinical expertise. Each endpoint may

have a unique set of covariates. Care is taken to only select a limited number of covariates such that the models are not over fitted.

Covariates for the dichotomous secondary endpoints, percentage of subjects abstinent, WHO 1-level risk category decrease, and WHO 2-level risk category decrease in alcohol consumption, will be the same as those used for the primary endpoint PSNHDD as described in Section 9.4.2. Fewer covariates for the logistic regression may be used depending upon the number of events. If the number of events permits the inclusion of a baseline drinking covariate, the percentage of days abstinent will be used as the covariate for the percent subjects abstinent endpoint; however, no baseline drinking covariate will be employed for the endpoint, percent subjects with a WHO decrease in alcohol consumption, as this endpoint already adjusts for baseline drinking in its calculation.

## 9.5. Handling of Missing Data

## 9.5.1. Primary Analysis of the Primary Efficacy Endpoint

The primary efficacy analysis of the PSNHDD endpoint will use all mITT subjects and will employ imputation for missing drinking data such that any subject with any missing drinking data during the evaluation period for this endpoint will be imputed as a subject with a heavy drinking day.

Prior to the subject dropping out of the study, every attempt will be made to continue to collect TLFB data; however, if the subject does not want to participate in the collection of the TLFB they will be asked to participate in a periodic follow-up phone call to collect a summary of drinking information. If the subject agrees to be contact then they will be asked about any drinking and heavy drinking during the time since last contact. Phone calls will continue until the end of the treatment period, as deemed acceptable by the patient. The two questions cover whether the subject had any heavy drinking days or drinking days during the period covered. This summary drinking data will be used for the primary endpoint.

If the subject does not agree to participate with phone contact thus no summary drinking data nor TLFB data is available then imputation as indicated above will be used.

## 9.5.2. Analysis of the Secondary Efficacy Endpoints

The primary efficacy analysis of the percentage of subjects abstinent endpoint will use all mITT subjects and will employ imputation for missing drinking data such that any subject with any missing drinking data during the evaluation period for this endpoint will be imputed as a subject with a drinking day. Analyses of supportive secondary efficacy endpoints will use all mITT subjects with no imputation for missing data. Analyses will also be performed in evaluable subjects.

#### 9.6. Safety Analysis

#### 9.6.1. Adverse Events

AEs will be coded using the most recent version of the Medical Dictionary for Regulatory Activities (MedDRA) and will be grouped by system, organ, and class (SOC) and preferred term (PT) designation. The severity, frequency, and relationship of AEs to investigational product will

be presented by SOC and PT groupings. Listings of each individual AE including start date, stop date, severity, relationship, outcome, and duration will be provided. Each AE (based on PT) will be counted once only for a given study subject. If the same AE occurred on multiple occasions, the highest severity will be assumed. Thus, study subjects are not counted multiple times in a given numerator in the calculation of frequencies for a specific AE. C-SSRS reports of suicidality or suicidal ideation will be reported as AEs and analyzed as AEs if the investigator determines after an interview with the subject, that the responses are consistent with suicidal ideation or attempt.

### 9.6.2. Clinical Laboratory and Point of Care Tests

For clinical laboratory data, descriptive statistics will be generated for all tests performed at screening and at each clinic visit. If a laboratory analysis is repeated, the last measurement performed prior to the clinic visit will be used in the summary statistics for that clinic visit. If an unscheduled clinical laboratory visit occurs prior to a scheduled visit that is missed due to dropout, then the unscheduled visit will be used in the summary statistics for the missed scheduled clinical visit. If an unscheduled clinical laboratory visit occurs between two scheduled clinical visits, then the data from the unscheduled visit only be presented in the listings and not in summary statistics. In addition, at each post-randomization clinic visit descriptive statistics for change from baseline will be generated. Laboratory values will be plotted as mean ± standard error over time. All laboratory measurements will be presented in the listings.

Number and percentage of positive urine drug tests and pregnancy tests for screening visits and all treatment and follow-up visits will be tabulated. Results of all urine drug tests and pregnancy tests will be presented in the listings. The percentage of subjects with a positive urine drug test at any time post start of treatment will also be presented by test type and treatment group.

#### 9.6.3. Vital Signs, ECG, and Body Weight

Vital signs will be presented as summary statistics and change from baseline. The percentage of ECG results considered abnormal and clinically significant will be provided. Body weight will be presented as summary statistics and change from screening. Vital signs, ECG results, and weight measurements for all visits will be presented in the listings.

#### 9.6.4. CIWA-AR Scores

The number and percentage of subjects who reported CIWA-AR scores  $\geq 10$  at any time after the start of dosing will be presented.

#### 9.6.5. Profile of Mood States

The POMS has 6 subscales and total disturbance score. Each subscale and summary score are continuous data and will be analyzed over the entire maintenance period using the same repeated measures mixed effects model as specified in Section 9.4.3. Treatment group, clinical site, study week, the treatment group by study week interaction, and baseline value of the subscale or summary score will be the only covariates in the mixed effects models for this endpoint. The entire maintenance period will be used for this endpoint. No imputation will be utilized for this safety endpoint.

## 9.7. Drug Exposure and Retention Analyses

Drug exposure will be presented for both groups as the mean number of tablets taken per week by subject self report during the entire treatment phase, mean total exposure over the entire maintenance period, and number of days that at least one dose was taken over the maintenance period. Self-reported compliance with HORIZANT Extended-Release Tablets will be compared against plasma samples having detectable levels of gabapentin by using 2 x 2 contingency tables. In addition, the percentage of subjects discontinuing medication and a listing of the reasons for discontinuation will be provided.

## 9.8. Other Services Used Analysis

Weekly days of attendance at self-help meetings or other professional service providers to help reduce/quit drinking will be presented as summary statistics by treatment group. All other services used data will be presented in the listings.

## 9.9. Blood Alcohol Content

The number and percent of subjects at any clinic visit that have a BAC > 0 will be tabulated. All BAC measurements will be presented in the listings.

## 9.10. PK Analysis

Plasma levels of gabapentin will be presented as descriptive statistics including mean, SD, coefficient of variation, geometric mean, 95% CI, minimum and maximum levels and mean  $\pm$  SD will be presented graphically over time. Population PK analyses will be conducted in accordance with a separate PK/PD SAP.

#### 9.11. Exploratory Analyses

#### 9.11.1. Exploratory Endpoint: Percentage of Subjects Abstinent from Smoking

The percentage of subjects abstinent from smoking is the number of subjects that have consumed no cigarettes per week during the weeks included in period of interest divided by the number of subjects with at least one week of non-missing smoking data during the period of interest, multiplied by 100. This endpoint will be analyzed only among subjects who smoked at baseline. Analysis will include two treatment time periods of interest: during the last 4 weeks of the maintenance period and over the entire maintenance period. The analysis will follow the plan in Section 9.4.1. The covariate selection plan will follow the plan in Section 9.4.2; however, if the number of events permits the inclusion of a baseline smoking covariate, the mean number of cigarettes smoked per week will be used. All analyses of this endpoint will be conducted on both a nonimputed and imputed endpoint. Imputation will proceed such that any subject with any missing cigarettes per week data during the evaluation periods for this endpoint will be imputed as a smoker.

#### 9.11.2. Exploratory Endpoint: MINI AUD Number of Symptoms

The MINI AUD total number of symptoms at Week 26 (covering the last 4 weeks of the maintenance period) will be modeled using analysis of covariance with the following variables

included in the model: treatment group, clinical site, and baseline MINI AUD total number of symptoms. No imputation will be performed.

## 9.11.3. Exploratory Endpoint: Blood PEth Levels

Blood PEth levels are measured at baseline and Week 26. Analysis of Week 26 blood PEth levels will be modeled using analysis of covariance with the following variables included in the model: treatment group, clinical site, and baseline blood PEth level. No imputation will be performed for this analysis.

The proportion of positive samples [a test result > 8 ng/mL - the lower limit of quantitation (LLOQ) of the test] at Week 26 data will be modeled using logistic regression with treatment group, clinical site, and baseline PEth level as covariates provided there are sufficient events. No imputation will be performed for this analysis.

# 9.11.4. Primary and Secondary Endpoints With or Without Imputation over Different Study Periods

Treatment group differences will be analyzed on a weekly and monthly basis for the imputed and nonimputed versions of the following three dichotomous drinking endpoints: PSNHDD, percentage of subjects abstinent from alcohol, percentage of subjects with a WHO 1-level decrease, and a WHO 2-level decrease in alcohol consumption. These analyses will use 2x2 contingency table. The Wald statistic from the fully covaried logistic regression will be used to test for treatment group differences. The adjusted prevalence rates are obtained from the logistic regression model. These rates along with the SD, 95% CI, difference between adjusted prevalence rates for the treatment groups, and Cohen's h. Graphs will present the weekly and monthly prevalence rates. These three dichotomous endpoints (both imputed and nonimputed) will further be analyzed by grace period, over: Weeks 22-25 (last 4 weeks), Weeks 18-25 (last 8 weeks), Weeks 14-25 (last 12 weeks), Weeks 10-25 (last 16 weeks), Weeks 6-25 (last 20 weeks) and Weeks 2-25 (last 24 weeks; i.e., entire maintenance phase) using 2x2 contagency tables. The Wald statistic from the fully covaried logistic regression will be used to test for treatment group differences. Graphs of the prevalence rates will be presented over the grace periods.

Covariates used in the exploratory analyses of these endpoints may be excluded if there are insufficient numbers of events. The imputation of PSNHDD and percentage of subjects abstinent from alcohol will proceed such that subjects with missing endpoint data will considered treatment failures. Since the WHO 1-level and WHO 2-level decrease in alcohol consumption utilizes average drinks per day in its calculation, multiple imputation (described below) will be used to impute weekly drinks per day data prior to computing this endpoint. The last 4 weeks (Weeks 22-25) for these three endpoints will be analyzed within the evaluable analysis set using imputed data for PSNHDD and non-imputed data for Percentage of Subjects abstinent from alcohol and WHO 1-level and WHO 2-level decrease in alcohol consumption.

Continuous secondary endpoints will be imputed via multiple imputation analyzed over the last 4 weeks of the maintenance period, and both imputed and nonimputed endpoints will be analyzed over the entire maintenance period, using repeated measures mixed effects described in Section 9.4 and using the same covariates selected for the primary analyses of these endpoints. Graphs will present the least squares means of the untransformed endpoints without imputation. The multiple imputation method for handling missing data will use the mITT population and will

replace each missing value with a set of "m" plausible values that represent the uncertainty about the right value to impute (<u>Hopke et al-2001</u>, <u>Rubin-1976</u>, <u>Rubin-1996</u>, <u>Schafer-1997</u>). The data are assumed to have monotone missingness, and the regression method will be used. The same variables used in the mixed effects model will be included in the multiple imputation models with the addition of time-related variables such as the values of the endpoint prior to dropout. The "m" imputed datasets each will be analyzed using mixed effects models then SAS PROC MIANALYZE will be used to combine the parameter estimates.

#### 9.11.5. Moderators of Drinking Outcomes

A number of variables will be tested as potential moderators of the medication treatment effect on the imputed PSNHDD primary endpoint. The time period of interest is the last 4 weeks of the maintenance period (Weeks 22-25). The models identified in Section 9.4 will be amended to include the potential moderator variable and the moderator by treatment group interaction. For the logistic regression models of PSNHDD, two covariates may need to be dropped from the final model of Section 9.4.2 to accommodate the moderator variable and interaction term. To aid with interpretation, continuous moderator variables will be dichotomized based on clinically accepted levels available from the literature. In the event a clinically meaningful cutoff is not available, receiver operator curves (ROC) (Harris-2010, Lambert and Lipkovich-2008) will be used. In all approaches, an appropriate cutoff will be one that ensures a sufficient sample size in all resultant subgroups. The potential moderator variables that will be examined include measures suggestive of alcohol withdrawal (i.e., withdrawal question on the MINI for alcohol use disorder, BAI, BDI-II, PSQI total score, POMS total and subscales, ACQ-SR-R total score, and number of days abstinent prior to randomization), severity of alcohol use disorder (i.e., drinks per week [28] days prescreen] and years of regular drinking), reducer status (change in baseline drinks per day), alcohol-related treatment goal (total abstinence vs. less than total abstinence), Barratt Impulsiveness Scale score, total dose of medication taken, and baseline smoking status.

#### 10. VALIDATION OF PROGRAMMING CODE

All SAS codes used to generate tables and listings will be validated and reviewed before being finalized. The validation process will be used to determine that the numbers are produced by a statistically valid method and that the execution of the computations is correct. Qualified personnel who have not previously been involved in the production of the original programming codes will perform the validation procedures. Methods of validation include independent programming and comparison to data listings. Tables will be reviewed for accuracy, consistency with this plan, consistency within tables, and consistency with corresponding output. Once validation is complete, a quality control reviewer will perform a final review of the documents for accuracy and consistency. Upon completion of validation and quality review procedures, all documentation will be collected and filed in the study documentation files at Fast-Track.

#### 11. REFERENCES

Aubin HJ, Reimer J, Nutt DJ, Bladstrom A, Torup L, Francois C, Chick J. Clinical relevance of as-needed treatment with nalmefene in alcohol dependent patients. Eur Addict Res. 2015;21:160–68.

Beck AT, Steer RA, Ball R, Ranieri W. Comparison of Beck Depression Inventories -IA and -II in psychiatric outpatients. J Personality Assess. 1966;67: 588-97.

Beck AT, Epstein N, Brown G, Steer RA. "An inventory for measuring clinical anxiety: Psychometric properties. J Consult Clinical Psych. 1988;56:893-897.

Buysse, D. J., Reynolds, C. F., 3rd, Monk, T. H., et al. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989;28:193-213.

Carey KB. Reliability and validity of the time-line follow-back interview among psychiatric outpatients: a preliminary report. Psych Addic Behav. 1997;11, 26-33.

Dmitrienko A, Tamhane AC. Gatekeeping procedures in clinical trials. Multiple Testing Problems in Pharmaceutical Statistics. Dmitrienko, A., Tamhane, A.C., Bretz, F. (editors). Chapman and Hall/CRC Press, New York. 2009.

Feinn R, Kranzler HR. Does effect size in naltrexone trials for alcohol dependence differ for single-site vs. multi-center studies? Alcohol Clin Exp Res. 2005;29:963-988.

Fleiss JL, Levin B., Paik MC. Statistical Methods for Rates and Proportions. Third Edition. John Wiley & Sons. New York. 2003.

Harris K. ROC Hard? No, ROC made easy. *Proc 2010 SAS Global Forum*. http://support.sas.com/resources/.../proceedings10/222-2010.pdf

Hopke PK, Liu C, Rubin DB. Multiple imputation for multivariate data with missing and below-threshold measurements: time-series concentrations of pollutants in the Arctic. Biometrics. 2001;57:22-33.

Lambert J, Lipkovich I. A Macro For Getting More Out Of Your ROC Curve." *Proc 2008 SAS Global Forum*. http://www2.sas.com/proceedings/forum2008/231-2008.pdf

Lipps GE, Lowe GA, De La Haye W, Longman-Mills S, Clarke TR, Banton EM, Bain B. Validation of the Beck Depression Inventory II in HIV-positive patients. West Ind Med J 2010;59:374-379.

Macefield RC, Metcalfe C, Lane JA, Donovan JL, Avery KNL, Blazeby JM, Down L, Neal DE, Hamdy FC, Vedhara K. Impact of prostate cance testing: evaluation of the emotional consequences of a negative biopsy result. Br J Cancer 2010;102:1335-1340.

Mason BJ, Light JM, Williams LD, Drobes DJ. Proof-of-concept human laboratory study for protracted abstinence in alcohol dependence: Effects of gabapentin. Addict Biol. 2009;14:73-83.

Mason BJ, Quello S, Goodell V, Shadan F. Gabapentin treatment for alcohol dependence. JAMA. 2014;174:70-77.

McNair DM, Heuchert JWP. Profile of Mood States (POMS) Multi-Health Systems, Tonawanda, NY. 2005.

Miller WR, Tonigan JS. The Drinker Inventory of Consequences (DrInC): an instrument for assessing adverse consequences of alcohol abuse. In Mattson, M. E., and Marshall, L. A. (Eds.) NIAAA Project MATCH Monograph Series, Vol. 4. Rockville, MD: National Institute on Alcohol Abuse and Alcoholism. 1995.

Peduzzi P, Concato J, Kemper E, Holford TR, Feinstein AR. A simulation study of the number of events per variable in logistic regression analysis. 1996;49:1373-1379.

Rubin DB. Inference and Missing Data. Biometrika. 1976;63:581–592.

Rubin DB. Multiple Imputation After 18+ Years. J Amer Statistical Assoc. 1996;91:473–489.

Schafer JL. Analysis of Incomplete Multivariate Data, New York: Chapman and Hall. 1997.

Sellers EM, Sullivan JT, Somer G, Sykora K. Characterization of DSM-III-R criteria for uncomplicated alcohol withdrawal: proposal for a diagnostic inventory and revised withdrawal scale. In Naranjo, C. A. and Sellers, E. M. (Eds.) Novel pharmacological interventions for alcoholism. New York (pp. 369-71). 1992.

Singleton EG, Tiffany, ST, Henningfield JE. Development and validation of a new questionnaire to assess craving for alcohol. In: Harris LS (ed) *Problems of Drug Dependence, 1994; Proceedings of the 56<sup>th</sup> Annual Scientific Meeting, The College on Problems of Drug Dependence, Inc.* National Institute of Drug Abuse Research Monograph Series. Vol. 153. Rockville, MD 1995. p. 289.

Sobell LC, Sobell MB, Leo GI, Cancilla A. Reliability of a timeline method: assessing normal drinkers' reports of recent drinking and a comparative evaluation across several populations. Br J Addict. 1988;83:393-402.

Sobell LC, Brown J, Leo GI, Sobell MB. The reliability of the Alcohol Timeline Followback when administered by telephone and by computer. Drug Alcohol Depend 1996;42:49-54.

Stuppaeck CH, Barnas C, Falk M, Guenther V, Hummer M, Oberbauer H, Pycha R, Whitworth AB, Fleischhacker WW. Assessment of the alcohol withdrawal syndrome--validity and reliability of the translated and modified Clinical Institute Withdrawal Assessment for Alcohol scale (CIWA-A). Addiction. 1994;89:1287-92.

Sullivan JT, Sykora K, Schneiderman J, Naranjo CA, Sellers EM. Assessment of alcohol withdrawal: the revised clinical institute withdrawal assessment for alcohol scale (CIWA-AR). Br J Addict. 1989;84:1353-7.

World Health Organization (WHO): International Guide for Monitoring Alcohol Consumption and Related Harm. Geneva, WHO, 2000. Available at: http://whqlibdoc.who.int/hq/2000/who msd msb 00.4.pdf.

- 12. TABLE, LISTING, AND FIGURE SHELLS
- 12.1. Tables
- 12.1.1. Subject Disposition, Participation, Compliance

**Table 1:** Subject Disposition - All Randomized Subjects

| | Treatment | Group | | |
|---|---|---|---|---|
| | Placebo<br>(N=xx)<br>n (%) | HORIZANT (N=xx) n (%) | Total<br>(N=xxx)<br>n (%) | p-value |
| | | , | | • |
| Number of Subjects Randomized not Receiving Study Drug | x (xx.x%) | x (xx.x%) | x (xx.x%) | |
| Number of mITT Subjects | xx (xx.x%) | xx (xx.x%) | xxx (xx.x%) | 0.xxx |
| Number of Completed Subjects | xx (xx.x%) | xx (xx.x%) | xxx (xx.x%) | 0.xxx |
| Number of Evaluable Subjects | xx (xx.x%) | xx (xx.x%) | xxx (xx.x%) | 0.xxx |
| Number of Subjects Discontinuing Medication, Remain in Study | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | 0.xxx |
| Number of Subjects Discontinuing Medication, Drop out of Study | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | 0.xxx |
| Reason for Any Discontinuation | | | | |
| Lost to follow up | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Died | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | |
| Adverse Event | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | |
| Logistical or practical reasons | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | |
| Lack of perceived efficacy | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | |
| Absent from the protocol due to confinement in a controlled environment | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | |
| Other reason | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | |

Notes: A subject might have more than one reason for discontinuation. .

Programmer Notes: The discontinuation reasons are as given on the CRF. Include only the reasons actually used for the subjects in the study. If a subject discontinued, but the specific reason is missing, include 'Missing' as a row in the table. Use the order of discontinuation reasons as presented on the CRF page.

<sup>&</sup>lt;sup>1</sup> p-value from chi-square test (c), and Fisher's exact test for binary (f)

**Table 2:** Exposure to Investigational Products – mITT Subjects

| | | | Plac | cebo | | | | | HORIZ | ZANT | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Period | N | Mean | SD | Med | Min | Max | n | Mean | SD | Med | Min | Max | p-value <sup>1</sup> |
| Escalation | | | | | | | | | | | | | |
| Dose <sup>2</sup> | | | | | | | | | | | | | |
| Week 1 | XX | XX.X | XX.X | XX.X | XX.X | XX.X | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx |
| Maintenance (Weeks 2-25) | | | | | | | | | | | | | |
| Total Dose | XX | XX.X | XX.X | XX.X | XX.X | XX.X | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx |
| Dose per Day | XX | XX.X | XX.X | XX.X | XX.X | XX.X | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx |
| Dose | | | | | | | | | | | | | |
| Week 2 | XX | XX.X | XX.X | XX.X | XX.X | XX.X | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx |
| Week 3 | XX | XX.X | XX.X | XX.X | XX.X | XX.X | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx |
| Week 4 | XX | XX.X | XX.X | XX.X | XX.X | XX.X | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx |
| Week 5 | XX | XX.X | XX.X | XX.X | XX.X | XX.X | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx |
| Week 6 | XX | XX.X | XX.X | XX.X | XX.X | XX.X | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx |
| Week 7 | XX | XX.X | XX.X | XX.X | XX.X | XX.X | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx |
| Week 8 | XX | XX.X | XX.X | XX.X | XX.X | XX.X | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx |
| Week 9 | XX | XX.X | XX.X | XX.X | XX.X | XX.X | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx |
| Week 10 | XX | XX.X | XX.X | XX.X | XX.X | XX.X | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx |
| Week 11 | XX | XX.X | XX.X | XX.X | XX.X | XX.X | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx |
| Week 12 | XX | XX.X | XX.X | XX.X | XX.X | XX.X | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx |
| Week 13 | XX | XX.X | XX.X | XX.X | XX.X | XX.X | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx |
| Week 14 | XX | XX.X | XX.X | XX.X | XX.X | XX.X | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx |
| Week 15 | XX | XX.X | XX.X | XX.X | XX.X | XX.X | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx |
| Week 16 | XX | XX.X | XX.X | XX.X | XX.X | XX.X | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx |
| Week 17 | XX | XX.X | XX.X | XX.X | XX.X | XX.X | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx |
| Week 18 | XX | XX.X | XX.X | XX.X | XX.X | XX.X | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx |
| Week 19 | XX | XX.X | XX.X | XX.X | XX.X | XX.X | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx |
| Week 20 | XX | XX.X | XX.X | XX.X | XX.X | XX.X | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx |
| Week 21 | XX | XX.X | XX.X | XX.X | XX.X | XX.X | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx |
| Week 22 | XX | XX.X | XX.X | XX.X | XX.X | XX.X | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx |
| Week 23 | XX | XX.X | XX.X | XX.X | XX.X | XX.X | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx |
| Week 24 | XX | XX.X | XX.X | XX.X | XX.X | XX.X | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx |
| Week 25 | XX | XX.X | XX.X | XX.X | XX.X | XX.X | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx |
| Taper | | | | | | | | | | | | | |
| Dose | | | | | | | | | | | | | |
| Week 26 | XX | XX.X | XX.X | XX.X | XX.X | XX.X | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx |

| | | | Plac | cebo | | | | | HORIZ | ZANT | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Period | N | Mean | SD | Med | Min | Max | n | Mean | SD | Med | Min | Max | p-value <sup>1</sup> |
| Overall (Weeks 1-26) | | | | | | | | | | | | | |
| Total dose | XX | XX.X | XX.X | XX.X | XX.X | XX.X | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx |
| Total dose per day | XX | XX.X | XX.X | XX.X | XX.X | XX.X | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx |

<sup>&</sup>lt;sup>1</sup> p-value from t-test for continuous variables (t) – skewed continuous data uses the Wilcoxon rank-sum test (w).
<sup>2</sup> Dose is expressed in number of capsules of HORIZANT or placebo.

Table 3: **Exposure to Investigational Products – Evaluable Subjects** 

Same as Table 2 only using Evaluable subjects.

**Drug Compliance – mITT Subjects** Table 4:

| | | | Plac | cebo | | | | | HORIZ | ZANT | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Period | n | Mean | SD | Med | Min | Max | n | Mean | SD | Med | Min | Max | p-value <sup>1</sup> |
| Escalation | | | | | | | | | | | | | |
| Compliance <sup>2</sup> | | | | | | | | | | | | | |
| Week 1 | XX | XX.X | XX.X | XX.X | XX.X | XX.X | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx |
| Maintenance (Weeks 2-25) | | | | | | | | | | | | | |
| Compliance | | | | | | | | | | | | | |
| Total Dose | XX | XX.X | XX.X | XX.X | XX.X | XX.X | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx |
| Week 2 | XX | XX.X | XX.X | XX.X | XX.X | XX.X | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx |
| Week 3 | XX | XX.X | XX.X | XX.X | XX.X | XX.X | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx |
| Week 4 | XX | XX.X | XX.X | XX.X | XX.X | XX.X | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx |
| Week 5 | XX | XX.X | XX.X | XX.X | XX.X | XX.X | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx |
| Week 6 | XX | XX.X | XX.X | XX.X | XX.X | XX.X | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx |
| Week 7 | XX | XX.X | XX.X | XX.X | XX.X | XX.X | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx |
| Week 8 | XX | XX.X | XX.X | XX.X | XX.X | XX.X | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx |
| Week 9 | XX | XX.X | XX.X | XX.X | XX.X | XX.X | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx |
| Week 10 | XX | XX.X | XX.X | XX.X | XX.X | XX.X | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx |
| Week 11 | XX | XX.X | XX.X | XX.X | XX.X | XX.X | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx |
| Week 12 | XX | XX.X | XX.X | XX.X | XX.X | XX.X | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx |
| Week 13 | XX | XX.X | XX.X | XX.X | XX.X | XX.X | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx |
| Week 14 | XX | XX.X | XX.X | XX.X | XX.X | XX.X | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx |
| Week 15 | XX | XX.X | XX.X | XX.X | XX.X | XX.X | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx |
| Week 16 | XX | XX.X | XX.X | XX.X | XX.X | XX.X | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx |
| Week 17 | XX | XX.X | XX.X | XX.X | XX.X | XX.X | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx |
| Week 18 | XX | XX.X | XX.X | XX.X | XX.X | XX.X | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx |
| Week 19 | XX | XX.X | XX.X | XX.X | XX.X | XX.X | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx |

| | | | Plac | cebo | | | | | HORIZ | ZANT | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Period | n | Mean | SD | Med | Min | Max | n | Mean | SD | Med | Min | Max | p-value <sup>1</sup> |
| Week 20 | XX | XX.X | XX.X | XX.X | XX.X | XX.X | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx |
| Week 21 | XX | XX.X | XX.X | XX.X | XX.X | XX.X | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx |
| Week 22 | XX | XX.X | XX.X | XX.X | XX.X | XX.X | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx |
| Week 23 | XX | XX.X | XX.X | XX.X | XX.X | XX.X | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx |
| Week 24 | XX | XX.X | XX.X | XX.X | XX.X | XX.X | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx |
| Week 25 | XX | XX.X | XX.X | XX.X | XX.X | XX.X | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx |
| <b>Taper</b> Compliance | | | | | | | | | | | | | |
| Week 26 | XX | XX.X | XX.X | XX.X | XX.X | XX.X | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx |
| Overall (Weeks 1-26) Compliance | | | | | | | | | | | | | |
| Total dose | XX | XX.X | XX.X | XX.X | XX.X | XX.X | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx |

<sup>&</sup>lt;sup>1</sup>p-value from t-test for continuous variables (t) – skewed continuous data uses the Wilcoxon rank-sum test (w).

**Table 5:** Drug Compliance – Evaluable Subjects

Same as Table 4 only using evaluable subjects.

**Table 6:** Summary of HORIZANT Blood Levels – HORIZANT Group (mITT Subjects)

| | | | | | | | | 95% | CI |
|---|---|---|---|---|---|---|---|---|---|
| Study Week | N | Mean | SD | % CV <sup>1</sup> | Min | Max | GeoMean | Upper CI | Lower CI |
| 12 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 20 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 24 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |

<sup>&</sup>lt;sup>1</sup>CV=Coefficient of variation

## Table 7: Summary of HORIZANT Blood Levels – HORIZANT Group (Evaluable Subjects)

Same as Table 6 only using evaluable subjects.

<sup>&</sup>lt;sup>2</sup>Compliance is expressed in number of capsules of HORIZANT or placebo.

Table 8: Self Report of HORIZANT Use (within 24 hours prior to PK sample) Versus Positive Gabapentin Blood Level – mITT Subjects

| | | Pill Count In<br>Tal | _ | |
|---|---|---|---|---|
| Timing | Blood Level Indicates Drug Taken <sup>1</sup> | Yes | No | p-value |
| Week 12 | | | | |
| | Yes | xx (xx.x%) | xx (xx.x%) | X.XXX |
| Week 20 | No | xx (xx.x%) | xx (xx.x%) | |
| WCCK 20 | Yes | xx (xx.x%) | xx (xx.x%) | X.XXX |
| Week 24 | No | xx (xx.x%) | xx (xx.x%) | |
| week 24 | Yes | xx (xx.x%) | xx (xx.x%) | X.XXX |
| Owanall | No | xx (xx.x%) | xx (xx.x%) | |
| Overall | Yes | xx (xx.x%) | xx (xx.x%) | x.xxx |
| | No | xx (xx.x%) | xx (xx.x%) | |

Blood level of  $\geq$ 80 ng/mL (lower limit of quantitation) indicates drug taken

Table 9: Self Report of HORIZANT Use (within 24 hours prior to PK sample) Versus Positive Gabapentin Blood Level – Evaluable Subjects

Same as Table 8 only using evaluable subjects.

Table 10: Exit Interview – mITT Subjects

| | Placebo | HORIZANT | Total | |
|---|---|---|---|---|
| Question | (N=xx) | (N=xx) | (N=xxx) | p-value <sup>1</sup> |
| What medication do you believe you were taking? | | | | 0.xxx |
| Placebo | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | |
| Active | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Both Active & Placebo | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| No Idea | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | |
| Other | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Missing | xx | XX | XX | |
| Why did you answer above? | | | | 0.xxx |
| Had side effects | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | |
| Had no side effects | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Staff treated me different | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| No improvement | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | |
| Had improvement | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | |
| Had a hunch | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | |
| I just felt different | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | |
| Other | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Missing | XX | XX | XX | |
| Do you feel the medication helped you to reduce drinking? | | | | 0.xxx |
| Very Much | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | |
| Much | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | |
| Moderately | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| A little | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | |
| Not at all | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Missing | XX | XX | XX | |
| How would you describe your experience taking the medication | n? | | | 0.xxx |
| Experienced no unwanted side effects and benefited | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | |
| Experienced some unwanted side effects but benefited | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Experienced a lot unwanted side effects but benefited | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | |
| Experienced no unwanted side effects but did not benefit | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Experienced some unwanted side effects and did not benefit | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Experienced a lot of unwanted side effects and did not benefit | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Missing | XX | XX | XX | |

| | Placebo | HORIZANT | Total | |
|---|---|---|---|---|
| Question | (N=xx) | (N=xx) | (N=xxx) | p-value <sup>1</sup> |
| If a friend were in need of help for a drink | ing problem, would you recommend tak | ing the medication to h | nim/her? | 0.xxx |
| Yes, definitely | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | |
| Yes, generally | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Neither yes nor no | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | |
| No, not really | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | |
| No, definitely not | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | |
| Missing | XX | Xx | XX | |
| If you were to need treatment in the future<br>Definitely yes<br>Probably yes | xx (xx.x%)<br>xx (xx.x%) | on again?<br>xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%) | 0.xxx |
| Maybe | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Probably not | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Definitely not | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Missing | xx | Xx | XX | |
| How much do you think of yourself as wan | ting to please other people (people pleas | er)? | | 0.xxx |
| More than average | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | |
| Average | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | |
| Less than average | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | |
| Missing | XX | Xx | XX | |

<sup>&</sup>lt;sup>1</sup> p-value from t-test for continuous variables (t) – skewed continuous data uses the Wilcoxon rank-sum test (w) - chi-square test for categorical variables (c).

## **Table 11:** Exit Interview – Evaluable Subjects

Same as Table 10 only using evaluable subjects.

**Table 12:** Dropouts by Treatment Group and Week – mITT Subjects

| | | Placebo (N=x | x) | | HORIZANT (N=x | xx) | |
|---|---|---|---|---|---|---|---|
| Study Week <sup>2</sup> | n | <b>Cumulative</b> n | <b>Cumulative %</b> | n | Cumulative n | <b>Cumulative %</b> | p-value <sup>1</sup> |
| Week 1 | XX | XX | XX.X% | XX | XX | XX.X <sup>0</sup> / <sub>0</sub> | 0.xxx |
| Week 2 | XX | XX | XX.X% | XX | XX | xx.x% | 0.xxx |
| Week 3 | XX | XX | XX.X% | XX | XX | xx.x% | 0.xxx |
| Week 4 | XX | XX | XX.X% | XX | XX | xx.x% | 0.xxx |
| Week 5 | XX | XX | XX.X% | XX | XX | xx.x% | 0.xxx |
| Week 6 | XX | XX | XX.X% | XX | XX | xx.x% | 0.xxx |
| Week 7 | XX | XX | XX.X% | XX | XX | xx.x% | 0.xxx |
| Week 8 | XX | XX | XX.X% | XX | XX | xx.x% | 0.xxx |
| Week 9 | XX | XX | XX.X <sup>0</sup> / <sub>0</sub> | XX | XX | xx.x% | 0.xxx |
| Week 10 | XX | XX | XX.X <sup>0</sup> / <sub>0</sub> | XX | XX | xx.x% | 0.xxx |
| Week 11 | XX | XX | $XX.X^{0}/_{0}$ | XX | XX | xx.x% | 0.xxx |
| Week 12 | XX | XX | XX.X <sup>0</sup> / <sub>0</sub> | XX | XX | xx.x% | 0.xxx |
| Week 13 | XX | XX | XX.X% | XX | XX | xx.x% | 0.xxx |
| Week 14 | XX | XX | $XX.X^{0}/_{0}$ | XX | XX | xx.x% | 0.xxx |
| Week 15 | XX | XX | XX.X <sup>0</sup> / <sub>0</sub> | XX | XX | xx.x% | 0.xxx |
| Week 16 | XX | XX | $XX.X^{0}/_{0}$ | XX | XX | xx.x% | 0.xxx |
| Week 17 | XX | XX | $XX.X^{0}/_{0}$ | XX | XX | xx.x% | 0.xxx |
| Week 18 | XX | XX | XX.X% | XX | XX | xx.x% | 0.xxx |
| Week 19 | XX | XX | $XX.X^{0}/_{0}$ | XX | XX | xx.x% | 0.xxx |
| Week 20 | XX | XX | XX.X <sup>0</sup> / <sub>0</sub> | XX | XX | xx.x% | 0.xxx |
| Week 21 | XX | XX | $XX.X^{0}/_{0}$ | XX | XX | xx.x% | 0.xxx |
| Week 22 | XX | XX | XX.X% | XX | XX | xx.x% | 0.xxx |
| Week 23 | XX | XX | $XX.X^{0}/_{0}$ | XX | XX | xx.x% | 0.xxx |
| Week 24 | XX | XX | XX.X% | XX | XX | xx.x% | 0.xxx |
| Week 25 | XX | XX | XX.X <sup>0</sup> / <sub>0</sub> | XX | XX | xx.x% | 0.xxx |
| Week 26 | XX | XX | XX.X% | XX | XX | xx.x% | 0.xxx |
| Week 27 | XX | XX | XX.X <sup>0</sup> / <sub>0</sub> | XX | XX | xx.x% | 0.xxx |

<sup>&</sup>lt;sup>1</sup> Fisher's exact test

**Table 13:** Dropouts by Treatment Group and Week – Evaluable Subjects

Same as Table 12 only using evaluable subjects.

<sup>&</sup>lt;sup>2</sup>Subjects are considered dropouts when they stop providing TLFB and other data. Subjects that discontinue study drug but provide data are not considered dropouts.

Table 14: Number and Percent of Subjects Using Summary Drinking Questions after Discontinuing TLFB – mITT Subjects

| | P | Placebo | HOR | IZANT | |
|------------|----|---------|-----|-------|----------------------|
| Study Week | n | % | n | % | p-value <sup>1</sup> |
| Week 3 | XX | XX.X% | XX | XX.X% | 0.xxx |
| Week 4 | XX | xx.x% | XX | XX.X% | 0.xxx |
| Week 5 | XX | xx.x% | XX | XX.X% | 0.xxx |
| Week 6 | XX | xx.x% | XX | XX.X% | 0.xxx |
| Week 7 | XX | xx.x% | XX | XX.X% | 0.xxx |
| Week 8 | XX | xx.x% | XX | xx.x% | 0.xxx |
| Week 9 | XX | xx.x% | XX | XX.X% | 0.xxx |
| Week 10 | XX | xx.x% | XX | xx.x% | 0.xxx |
| Week 11 | XX | xx.x% | XX | xx.x% | 0.xxx |
| Week 12 | XX | xx.x% | XX | xx.x% | 0.xxx |
| Week 13 | XX | xx.x% | XX | xx.x% | 0.xxx |
| Week 14 | XX | xx.x% | XX | xx.x% | 0.xxx |
| Week 15 | XX | xx.x% | XX | xx.x% | 0.xxx |
| Week 16 | XX | xx.x% | XX | XX.X% | 0.xxx |
| Week 17 | XX | xx.x% | XX | XX.X% | 0.xxx |
| Week 18 | XX | xx.x% | XX | XX.X% | 0.xxx |
| Week 19 | XX | xx.x% | XX | xx.x% | 0.xxx |
| Week 20 | XX | xx.x% | XX | XX.X% | 0.xxx |
| Week 21 | XX | xx.x% | XX | XX.X% | 0.xxx |
| Week 22 | XX | xx.x% | XX | xx.x% | 0.xxx |
| Week 23 | XX | xx.x% | XX | xx.x% | 0.xxx |
| Week 24 | XX | xx.x% | XX | XX.X% | 0.xxx |
| Week 25 | XX | XX.X% | XX | xx.x% | 0.xxx |
| Week 26 | XX | xx.x% | XX | xx.x% | 0.xxx |
| Week 27 | XX | xx.x% | XX | xx.x% | 0.xxx |
| Overall | XX | xx.x% | XX | xx.x% | 0.xxx |

<sup>&</sup>lt;sup>1</sup>Fisher's exact test

Note only rows with values above 0 will be presented

Table 15: Number and Percent of Subjects Using Summary Drinking Questions after Discontinuing TLFB – Evaluable Subjects

Same as Table 14 only using evaluable subjects.

| 12.1.2. | Demographic and Baseline Characteristics |
|---------|------------------------------------------|

 Table 16:
 Demographic Characteristics - mITT Subjects

| | Placebo | HORIZANT | Total | |
|---|---|---|---|---|
| Characteristic | (N=xx) | (N=xx) | (N=xxx) | p-value <sup>1</sup> |
| Age (years) | | | | 0.xxx |
| N | XX | XX | XX | |
| Mean | XX.X | XX.X | XX.X | |
| SD | XXX.XX | XXX.XX | XXX.XX | |
| Median | XX | XX | XX | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Gender | | | | 0.xxx |
| N | | | | |
| Male | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Female | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | |
| Race | | | | 0.xxx |
| N | XX | XX | XX | |
| White | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| African-American or Black | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | |
| Asian | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Native Hawaiian or Other Pacific Islander | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | |
| American Indian or Alaskan Native | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Other | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | |
| Ethnicity | | | | 0.xxx |
| N | XX | XX | XX | |
| Hispanic or Latino | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | |
| Not Hispanic or Latino | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | |
| Race/Ethnicity | | | | 0.xxx |
| N | XX | XX | XX | |
| White | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | |
| Black | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | |
| Hispanic | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | |
| Other | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | |

<sup>1</sup> p-value from chi-square test (c), t-test for continuous data, and Fisher's exact test for binary categories (f)

 Table 16:
 Demographic and Baseline Characteristics - mITT Subjects (Continued)

| | Placebo<br>(N=xx) | HORIZANT | Total<br>(N=xxx) | p-value <sup>1</sup> |
|---|---|---|---|---|
| Characteristic | | (N=xx) | | |
| Education (years) | | ` ' | , , | 0.xxx |
| N | XX | XX | XX | |
| Mean | XX.X | XX.X | XX.X | |
| SD | XXX.XX | XXX.XX | XXX.XX | |
| Median | XX | XX | XX | |
| Education | | | | 0.xxx |
| ≤ High School | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | |
| > High School | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | |
| Marital Status | | | | 0.xxx |
| Legally Married | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | |
| Living with Partner / Cohabitating | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | |
| Widowed | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | |
| Separated | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | |
| Divorced | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | |
| Never Married | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Marital Status | | | | 0.xxx |
| Married | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | |
| Not Married | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | |
| Employment | | | | 0.xxx |
| Full-time > 35 hrs /week | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | |
| Part-time regular | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | |
| Part-time irregular | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | |
| Student | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | |
| Military Service | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | |
| Unemployed | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | |
| Retired/Disabled | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | |
| Homemaker | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | |
| In controlled environment | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Employment | | | | 0.xxx |
| Employed | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | |
| Unemployed | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |

## Table 17: Demographic Characteristics - Evaluable Subjects

Same as Table 16 only using evaluable subjects.

 Table 18:
 Psychiatric Baseline Characteristics – mITT Subjects

| | Placebo | HORIZANT | Total | |
|---|---|---|---|---|
| Characteristic | (N=xx) | (N=xx) | (N=xxx) | p-value <sup>1</sup> |
| BIS First Order Factors | | | | |
| Attention | | | | 0.xxx |
| N | XX | XX | XX | |
| Mean | XX.X | XX.X | XX.X | |
| SD | XXX.XX | XXX.XX | XXX.XX | |
| Median | XX | XX | XX | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Scale Min-Max | | | (xx-xx) | |
| Motor | | | | 0.xxx |
| N | XX | XX | XX | |
| Mean | XX.X | XX.X | XX.X | |
| SD | XXX.XX | XXX.XX | XXX,XX | |
| Median | XX | XX | XX | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Scale Min-Max | , , | , , | (xx-xx) | |
| Self Control | | | | 0.xxx |
| Ň | XX | XX | XX | |
| Mean | XX.X | XX.X | XX.X | |
| SD | XXX.XX | XXX.XX | XXX.XX | |
| Median | XX | XX | XX | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Scale Min-Max | , , | , , | (xx-xx) | |
| Cognitive Complexity | | | | 0.xxx |
| N | XX | XX | XX | |
| Mean | XX.X | XX.X | XX.X | |
| SD | XXX.XX | XXX.XX | XXX.XX | |
| Median | XX | XX | XX | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Scale Min-Max | , | ` ' | (xx-xx) | |
| | Placebo | HORIZANT | Total | |
|---|---|---|---|---|
| Characteristic | (N=xx) | (N=xx) | (N=xxx) | p-value <sup>1</sup> |
| Perseverance | | | | 0.xxx |
| N | XX | XX | XX | |
| Mean | XX.X | XX.X | XX.X | |
| SD | XXX.XX | xxx.xx | XXX.XX | |
| Median | XX | XX | XX | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Scale Min-Max | | | (xx-xx) | |
| Cognitive Instability | | | | 0.xxx |
| N | XX | XX | XX | |
| Mean | XX.X | XX.X | XX.X | |
| SD | XXX.XX | XXX.XX | XXX.XX | |
| Median | XX | XX | XX | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Scale Min-Max | | | (xx-xx) | |
| BIS Second-order Factors | | | | |
| Attentional | | | | 0.xxx |
| N | XX | XX | XX | |
| Mean | XX.X | XX.X | XX.X | |
| SD | XXX.XX | XXX.XX | XXX.XX | |
| Median | XX | XX | XX | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Scale Min-Max | | | (xx-xx) | |
| Motor | | | | 0.xxx |
| N | XX | XX | XX | |
| Mean | XX.X | XX.X | XX.X | |
| SD | XXX.XX | xxx.xx | XXX.XX | |
| Median | XX | XX | XX | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Scale Min-Max | | | (xx-xx) | |

| | Placebo | HORIZANT | Total | |
|---|---|---|---|---|
| Characteristic | (N=xx) | (N=xx) | (N=xxx) | p-value <sup>1</sup> |
| Non planning | | | | 0.xxx |
| N | XX | XX | XX | |
| Mean | XX.X | XX.X | XX.X | |
| SD | XXX.XX | XXX.XX | XXX.XX | |
| Median | XX | XX | XX | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Scale Min-Max | | | (xx-xx) | |
| BAI | | | | |
| N | XX | XX | XX | 0.xxx |
| Mean | XX.X | XX.X | XX.X | |
| SD | XXX.XX | XXX.XX | XXX.XX | |
| Median | XX | XX | XX | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Scale Range | | | (xx-xx) | |
| Minimal anxiety | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | 0.xxx |
| Mild anxiety | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | |
| Moderate anxiety | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | |
| Severe anxiety | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| BDI-II | | | | 0.xxx |
| N | XX | XX | XX | |
| Mean | XX.X | XX.X | XX.X | |
| SD | XXX.XX | XXX.XX | XXX.XX | |
| Median | XX | XX | XX | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Scale Min-Max | | | (xx-xx) | |
| Minimal depression | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | 0.xxx |
| Mild depression | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Moderate depression | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | |
| Severe depression | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |

| | Placebo | HORIZANT | Total | |
|---|---|---|---|---|
| Characteristic | (N=xx) | (N=xx) | (N=xxx) | p-value <sup>1</sup> |
| DSM-5 Disorders | | | | |
| Depression | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | |
| Suicidality | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | |
| Manic | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | |
| Hypomanic | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | |
| Bipolar | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | |
| Panic | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | |
| Agoraphobia | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | |
| Social Phobia | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | |
| Obsessive Compulsive | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | |
| Posttraumatic Stress | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Substance Abuse | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | |
| Psychotic | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Mood | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | |
| Anorexia | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Bulemia | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | |
| Binge-eating | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Generalized Anxiety | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | |
| Medical Organic | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | |
| Antisocial Personality | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | |

<sup>1</sup> p-value from chi-square test (c), t-test (t), and Fisher's exact test for binary categories (f)

 Table 19:
 Psychiatric Baseline Characteristics – Evaluable Subjects

Same as Table 18 only using evaluable subjects.

 Table 20:
 Baseline POMS – mITT Subjects

| | Placebo | HORIZANT | Total | |
|----------------------|---------|----------|---------|----------------------|
| Characteristic | (N=xx) | (N=xx) | (N=xxx) | p-value <sup>1</sup> |
| Tension-Anxiety | | | | 0.xxx |
| N | XX | XX | XX | |
| Mean | XX.X | XX.X | XX.X | |
| SD | XXX.XX | XXX.XX | XXX.XX | |
| Median | XX | XX | XX | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Scale Min-Max | | | (xx-xx) | |
| Depression-Dejection | | | | 0.xxx |
| N | XX | XX | XX | |
| Mean | XX.X | XX.X | XX.X | |
| SD | XXX.XX | XXX.XX | XXX.XX | |
| Median | XX | XX | XX | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Scale Min-Max | | | (xx-xx) | |
| Anger-Hostility | | | | 0.xxx |
| N | XX | XX | XX | |
| Mean | XX.X | XX.X | XX.X | |
| SD | XXX.XX | XXX.XX | XXX.XX | |
| Median | XX | XX | XX | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Scale Min-Max | | | (xx-xx) | |
| Fatigue-Inertia | | | | 0.xxx |
| N | XX | XX | XX | |
| Mean | XX.X | XX.X | XX.X | |
| SD | XXX.XX | xxx.xx | XXX.XX | |
| Median | XX | XX | XX | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Scale Min-Max | | | (xx-xx) | |

| | Placebo | HORIZANT | Total | |
|---|---|---|---|---|
| Characteristic | (N=xx) | (N=xx) | (N=xxx) | p-value <sup>1</sup> |
| Confusion-Bewilderment | · | | | 0.xxx |
| N | XX | XX | XX | |
| Mean | XX.X | XX.X | XX.X | |
| SD | XXX.XX | XXX.XX | XXX.XX | |
| Median | XX | XX | XX | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Scale Min-Max | | | (xx-xx) | |
| Vigor-Activity | | | | 0.xxx |
| N | XX | XX | XX | |
| Mean | XX.X | XX.X | XX.X | |
| SD | XXX.XX | XXX.XX | XXX.XX | |
| Median | XX | XX | XX | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Scale Min-Max | | | (xx-xx) | |
| Total Mood Disturbance | | | | 0.xxx |
| N | XX | XX | XX | |
| Mean | XX.X | XX.X | XX.X | |
| SD | XXX.XX | XXX.XX | XXX.XX | |
| Median | XX | XX | XX | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Scale Min-Max | , | , , | (xx-xx) | |

Note: 1 p-value from t-test for continuous variables (t) – skewed continuous data uses the Wilcoxon rank-sum test (w)

 Table 21:
 Baseline POMS – Evaluable Subjects

Same as Table 20 only using evaluable subjects.

 Table 22:
 Baseline PSQI – mITT Subjects

| | Placebo | HORIZANT | Total | |
|-------------------|---------|----------|---------|----------------------|
| Characteristic | (N=xx) | (N=xx) | (N=xxx) | p-value <sup>1</sup> |
| Sleep Quality | | | | 0.xxx |
| N | XX | XX | XX | |
| Mean | XX.X | XX.X | XX.X | |
| SD | XXX.XX | XXX.XX | XXX.XX | |
| Median | XX | XX | XX | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Scale Min-Max | | | (xx-xx) | |
| Sleep Latency | | | | 0.xxx |
| N | XX | XX | XX | |
| Mean | XX.X | XX.X | XX.X | |
| SD | XXX.XX | XXX.XX | XXX.XX | |
| Median | XX | XX | XX | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Scale Min-Max | | | (xx-xx) | |
| Sleep Duration | | | | 0.xxx |
| N | XX | XX | XX | |
| Mean | XX.X | XX.X | XX.X | |
| SD | XXX.XX | XXX.XX | XXX.XX | |
| Median | XX | XX | XX | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Scale Min-Max | | | (xx-xx) | |
| Sleep Disturbance | | | | 0.xxx |
| N | XX | XX | XX | |
| Mean | XX.X | XX.X | XX.X | |
| SD | XXX.XX | XXX.XX | XXX.XX | |
| Median | XX | XX | XX | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Scale Min-Max | | | (xx-xx) | |

| | Placebo | HORIZANT | Total | |
|---|---|---|---|---|
| Characteristic | (N=xx) | (N=xx) | (N=xxx) | p-value <sup>1</sup> |
| Use of Sleep Medication | , , | ` , | | 0.xxx |
| N | XX | XX | XX | |
| Mean | XX.X | XX.X | XX.X | |
| SD | XXX.XX | XXX.XX | XXX.XX | |
| Median | XX | XX | XX | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Scale Min-Max | | | (xx-xx) | |
| Daytime Dysfunction | | | | 0.xxx |
| N | XX | XX | XX | |
| Mean | XX.X | XX.X | XX.X | |
| SD | XXX.XX | XXX.XX | XXX.XX | |
| Median | XX | XX | XX | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Scale Min-Max | | | (xx-xx) | |
| Overall Sleep Experience | | | | 0.xxx |
| N | XX | XX | XX | |
| Mean | XX.X | XX.X | XX.X | |
| SD | XXX.XX | XXX.XX | XXX.XX | |
| Median | XX | XX | XX | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Scale Min-Max | | , , | (xx-xx) | |

Note: 1 p-value from t-test for continuous variables (t) – skewed continuous data uses the Wilcoxon rank-sum test (w)

**Table 23:** Baseline PSQI – Evaluable Subjects

Same as Table 22 only using evaluable subjects.

Table 24: Drinking-related Behavior and Characteristics – mITT Subjects

| | Placebo | HORIZANT | Total | |
|---|---|---|---|---|
| Characteristic | (N=xx) | (N=xx) | (N=xxx) | p-value <sup>1</sup> |
| Family Members with History of Alcohol | | | | 0.xxx |
| Problems | | | | |
| None | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Father | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Mother | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | |
| 1 Sibling | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | |
| >1 Sibling | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| 1 Child | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | |
| >1 Child | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Parental History of Alcohol Problems | | | | 0.xxx |
| Father and/or Mother | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| None | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | |
| Drinking Goal (n, %) | | | | 0.xxx |
| Controlled Use | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | |
| Temporary Abstinence | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | |
| Occasional Drinking | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | |
| Total Abstinence with Slip | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Total Abstinence | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| No Goal | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | |
| Abstinence Goal | | | | 0.xxx |
| <total abstinence<="" td=""><td>xx (xx.x%)</td><td>xx (xx.x%)</td><td>xx(xx.x%)</td><td></td></total> | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | |
| Total Abstinence | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | |
| Motivation to Reach Goal | , , | | · · · | 0.xxx |
| N | XX | XX | XX | |
| Mean | XX.X | XX.X | XX.X | |
| SD | XXX.XX | XXX.XX | XXX.XX | |
| Median | XX | XX | XX | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Scale Min-Max | , | ` , | (xx - xx) | |
| Confidence to Reach Goal | | | , | |
| N | XX | XX | XX | 0.xxx |
| Mean | XX.X | XX.X | XX.X | |
| SD | XXX.XX | XXX.XX | XXX.XX | |
| Median | XX | XX | XX | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Scale Min-Max | • / | • • • | (xx - xx) | |

| | Placebo | HORIZANT | Total | |
|---|---|---|---|---|
| Characteristic | (N=xx) | (N=xx) | (N=xxx) | p-value <sup>1</sup> |
| AUD C 4 C 4 | | | | 0 |
| AUD Symptom Severity | ( 0/) | ( 0() | ( 0/) | 0.xxx |
| Moderate (4 or 5 symptoms) | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | |
| Severe (6 or more symptoms) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | |
| AUD Number of Symptoms | | | | 0.xxx |
| 4 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| 5 | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | |
| 6 | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | |
| 7 | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | |
| 8 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| 9 | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | |
| 10 | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | |
| 11 | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | |
| AUD Number of Symptoms (continuous) | | | | 0.xxx |
| N | XX | XX | XX | |
| Mean | XX.X | XX.X | XX.X | |
| SD | XXX.XX | XXX.XX | XXX.XX | |
| Median | XX | XX | XX | |
| Age First Started Drinking Regularly (years) | | | | |
| N | XX | XX | XX | 0.xxx |
| Mean | XX.X | XX.X | XX.X | |
| SD | XXX,XX | XXX.XX | XXX.XX | |
| Median | XX | XX | XX | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| | (M. M.) | (int int) | (M. M.) | |
| Number Lifetime Hospitalizations to | | | | |
| Reduce/Quit Drinking | | | | 0 |
| N | XX | XX | XX | 0.xxx |
| Mean | XX.X | XX.X | XX.X | |
| SD | XXX.XX | XXX.XX | XXX.XX | |
| Median | XX | XX | XX | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |

| | Placebo | HORIZANT | Total | |
|---|---|---|---|---|
| Characteristic | (N=xx) | (N=xx) | (N=xxx) | p-value <sup>1</sup> |
| Number Lifetime Hospitalizations for Illness/ | | | | |
| Injuries due to Drinking | | | | |
| N | XX | XX | XX | 0.xxx |
| Mean | XX.X | XX.X | XX.X | |
| SD | XXX.XX | XXX.XX | XXX.XX | |
| Median | XX | XX | XX | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Number Outpatient Visits to Reduce/Quit | | | | |
| Drinking in Last 12 Months | | | | |
| N | XX | XX | XX | 0.xxx |
| Mean | XX.X | XX.X | XX.X | |
| SD | XXX.XX | XXX.XX | XXX.XX | |
| Median | XX | XX | XX | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Number Lifetime Medical Detoxifications | | | | |
| N | XX | XX | XX | 0.xxx |
| Mean | XX.X | XX.X | XX.X | |
| SD | XXX.XX | XXX.XX | XXX.XX | |
| Median | XX | XX | XX | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Past Year Number of Support Group Meetings | | | | |
| N | XX | XX | XX | 0.xxx |
| Mean | XX.X | XX.X | XX.X | |
| SD | XXX.XX | xxx.xx | XXX.XX | |
| Median | XX | XX | XX | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |

Note: Percentages are based on the number of non-missing values in each variable.

## Table 25: Drinking-related Behavior and Characteristics – Evaluable Subjects

Same subjects as Table 24 only using evaluable subjects.

<sup>&</sup>lt;sup>1</sup> p-value from t-test for continuous variables (t) – skewed continuous data uses the Wilcoxon rank-sum test (w) - chi-square test for categorical variables (c) – Fisher's exact test for dichotomous variables (f)

 Table 26:
 Baseline Drinking by TLFB – mITT Subjects

| | Placebo | HORIZANT | Total | |
|---|---|---|---|---|
| Parameter | (N=xx) | (N=xx) | (N=xxx) | p-value <sup>1</sup> |
| Drinks/Week (Pre-screening Days -1 to -28) | | | | 0.xxx |
| Mean | XX.X | XX.X | XX.X | |
| SD | XX.X | XX.X | XX.X | |
| Median | XX.X | XX.X | XX.X | |
| Minimum | XX.X | XX.X | XX.X | |
| Maximum | XX.X | XX.X | XX.X | |
| Drinks/Week (7 Days Prior to Randomization) | | | | 0.xxx |
| Mean | XX.X | XX.X | XX.X | |
| SD | XX.X | XX.X | XX.X | |
| Median | XX.X | XX.X | XX.X | |
| Minimum | XX.X | XX.X | XX.X | |
| Maximum | XX.X | XX.X | XX.X | |
| Drinks/Week (Percent Change Pre-screening Days -1 to -28 to 7 Days Prior to Randomization) | | | | 0.xxx |
| Mean | XX.X | XX.X | XX.X | |
| SD | XX.X | XX.X | XX.X | |
| Median | XX.X | XX.X | XX.X | |
| Minimum | XX.X | XX.X | XX.X | |
| Maximum | XX.X | XX.X | XX.X | |
| Drinks/Drinking Day (Pre-screening Days -1 to -28) | | | | 0.xxx |
| Mean | XX.X | XX.X | XX.X | |
| SD | XX.X | XX.X | XX.X | |
| Median | XX.X | XX.X | XX.X | |
| Minimum | XX.X | XX.X | XX.X | |
| Maximum | XX.X | XX.X | XX.X | |
| Drinks/Drinking Day (7Days Prior to Randomization) | | | | 0.xxx |
| Mean | XX.X | XX.X | XX.X | |
| SD | XX.X | XX.X | XX.X | |
| Median | XX.X | XX.X | XX.X | |
| Minimum | XX.X | XX.X | XX.X | |
| Maximum | XX.X | XX.X | XX.X | |

| | Placebo | HORIZANT | Total | |
|---|---|---|---|---|
| Parameter | (N=xx) | (N=xx) | (N=xxx) | p-value <sup>1</sup> |
| Drinks/Drinking Day (Percent Change Pre-screening Days - | | | | 0.xxx |
| 1 to -28 to 7 Days Prior to Randomization) | | | | U.XXX |
| Mean | XX.X | XX.X | XX.X | |
| SD | XX.X | XX.X | XX.X | |
| Median | XX.X | XX.X | XX.X | |
| Minimum | XX.X | XX.X | XX.X | |
| Maximum | XX.X | XX.X | XX.X | |
| Percentage of Heavy Drinking Days | | | | 0.xxx |
| (Pre-screening Days -1 to -28) | | | | |
| Mean | $XX.X^{0}/_{0}$ | xx.x% | $xx.x^{0}/_{0}$ | |
| SD | $XX.X^{0}/_{0}$ | xx.x% | $xx.x^{0}/_{0}$ | |
| Median | $XX.X^{0}/_{0}$ | xx.x% | $xx.x^{0}/_{0}$ | |
| Minimum | XX.X% | xx.x% | XX.X% | |
| Maximum | XX.X <sup>0</sup> / <sub>0</sub> | XX.X <sup>0</sup> / <sub>0</sub> | xx.x% | |
| Percentage Days Abstinent | | | | 0.xxx |
| (Pre-screening Days -1 to -28) | | | | |
| Mean | XX.X% | xx.x% | XX.X% | |
| SD | XX.X% | xx.x% | XX.X% | |
| Median | XX.X% | xx.x% | XX.X% | |
| Minimum | XX.X% | xx.x% | XX.X% | |
| Maximum | XX.X <sup>0</sup> / <sub>0</sub> | XX.X <sup>0</sup> / <sub>0</sub> | xx.x% | |
| WHO Risk Level | | | | 0.xxx |
| High Risk | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | |
| Very High Risk | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |

## **Table 27:** Baseline Drinking by TLFB - Evaluable Subjects

Same as Table 26 only using evaluable subjects.

Note: Percentages are based on the number of non-missing values in each variable.

1 p-value from t-test for continuous variables (t) – skewed continuous data uses the Wilcoxon rank-sum test (w) - chi-square test for categorical variables (c)

Table 28: Baseline Alcohol-Related Craving, Consequences, and Withdrawal – mITT Subjects

| | Placebo | HORIZANT | Total | |
|----------------|---------|----------|---------------|----------------------|
| Parameter | (N=xx) | (N=xx) | (N=xxx) | p-value <sup>1</sup> |
| ACQ-SR-R | | | | |
| Total Score | | | | 0.xxx |
| Mean | XX.X | XX.X | XX.X | |
| SD | XX.X | XX.X | XX.X | |
| Median | XX.X | XX.X | XX.X | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Scale Min-Max | | | (xx.x - xx.x) | |
| Compulsivity | | | | 0.xxx |
| Mean | XX.X | XX.X | XX.X | |
| SD | XX.X | XX.X | XX.X | |
| Median | XX.X | XX.X | XX.X | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Scale Min-Max | | | (xx.x - xx.x) | |
| Expectancy | | | | 0.xxx |
| Mean | XX.X | XX.X | XX.X | |
| SD | XX.X | XX.X | XX.X | |
| Median | XX.X | XX.X | XX.X | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Scale Min-Max | | | (xx.x - xx.x) | |
| Purposefulness | | | | 0.xxx |
| Mean | XX.X | XX.X | XX.X | |
| SD | XX.X | XX.X | XX.X | |
| Median | XX.X | XX.X | XX.X | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Scale Min-Max | | | (xx.x - xx.x) | |
| Emotionality | | | | 0.xxx |
| Mean | XX.X | XX.X | XX.X | |
| SD | XX.X | XX.X | XX.X | |
| Median | XX.X | XX.X | XX.X | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | |
| Scale Min-Max | | | (xx.x - xx.x) | |

| | Placebo | HORIZANT | Total | |
|---|---|---|---|---|
| Parameter | (N=xx) | (N=xx) | (N=xxx) | p-value <sup>1</sup> |
| ImBIBe | · | | | |
| Total Score | | | | 0.xxx |
| Mean | XX.X | XX.X | XX.X | |
| SD | XX.X | XX.X | XX.X | |
| Median | XX.X | XX.X | XX.X | |
| Minimum | XX.X | XX.X | XX.X | |
| Maximum | XX.X | XX.X | XX.X | |
| Scale Min-Max | | | (xx.x - xx.x) | |
| CIWA-AR | | | | 0.xxx |
| Mean | XX.X | XX.X | XX.X | |
| SD | XX.X | XX.X | XX.X | |
| Median | XX.X | XX.X | XX.X | |
| Minimum | XX.X | XX.X | XX.X | |
| Maximum | XX.X | XX.X | XX.X | |
| Scale Min-Max | | | (xx.x - xx.x) | |
| Withdrawal Symptoms (CIWA $\geq$ 10) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | 0.xxx |

Note: 1 p-value from t-test for continuous variables (t) – skewed continuous data uses the Wilcoxon rank-sum test (w); chi-squared test for symptoms (c)

Programmer's note: Place the parenthesis and character after each p-value to denote the test

 Table 29:
 Baseline Alcohol-Related Craving, Consequences, and Withdrawal – Evaluable Subjects

Same as Table 28 only using evaluable subjects.

 Table 30:
 Baseline Other Substance Use – mITT Subjects

| | Placebo | HORIZANT | Total | |
|---|---|---|---|---|
| Parameter | (N=xx) | (N=xx) | (N=xxx) | p-value <sup>1</sup> |
| Fagerstrom Test for Nicotine Dependence | | | | |
| How often do you smoke? | | | | |
| Not at all | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | 0.xxx |
| Occasionally | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | |
| Daily | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | |
| How soon upon waking smoke? | | | | 0.xxx |
| <= 5 min | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | |
| 6-30 min | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| 31-60 min | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| After 1 hr | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | |
| Difficult to refrain from smoking? | | | | 0.xxx |
| No | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | |
| Yes | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Which eigarette do you hate to give up the most? | | | | 0.xxx |
| First morning | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | |
| All others | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | |
| How many cigarettes per day? | | | | 0.xxx |
| 10 or less | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | |
| 11-20 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| 21-30 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| 31 or more | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Smoke more frequently during 1st hours of waking? | | | | 0.xxx |
| No | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | |
| Yes | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Do you smoke if you are ill and in bed? | ( ) | ( / | | 0.xxx |
| No | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Yes | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |

| | Placebo | HORIZANT | Total | |
|---|---|---|---|---|
| Parameter | (N=xx) | (N=xx) | (N=xxx) | p-value <sup>1</sup> |
| Nicotine Dependence Score | | | | 0.xxx |
| Mean | XX.X | XX.X | XX.X | |
| SD | XX.X | XX.X | XX.X | |
| Median | XX.X | XX.X | XX.X | |
| Minimum | XX.X | XX.X | XX.X | |
| Maximum | XX.X | XX.X | XX.X | |
| <b>Days Smoked in the Past Week</b> | | | | 0.xxx |
| Mean | XX.X | XX.X | XX.X | |
| SD | XX.X | XX.X | XX.X | |
| Median | XX.X | XX.X | XX.X | |
| Minimum | XX.X | XX.X | XX.X | |
| Maximum | XX.X | XX.X | XX.X | |
| Average Cigarettes Smoked Per Week | | | | 0.xxx |
| Mean | XX.X | XX.X | XX.X | |
| SD | XX.X | XX.X | XX.X | |
| Median | XX.X | XX.X | XX.X | |
| Minimum | XX.X | XX.X | XX.X | |
| Maximum | XX.X | XX.X | XX.X | |
| THC | | | | 0.xxx |
| Negative | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Positive | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |

Note: Percentages are based on the number of non-missing values in each variable. <sup>1</sup> p-value from t-test for continuous variables (t) – skewed continuous data uses the Wilcoxon rank-sum test (w) - chi-square test for categorical (c), Fisher's exact test for binary variables (f) *Programmer's note: Place the parenthesis and character after each p-value to denote the test* 

**Table 31:** Baseline Other Substance Use – Evaluable Subjects

Same as Table 30 only using evaluable subjects.

## 12.1.3. Primary Efficacy Endpoint

Table 32: Subjects with No Heavy Drinking Days (mITT) – Full Model, Logistic Regression, Weeks 22-25, with Imputation<sup>a</sup>

| | | | | | | | | | 95% | 6 CI |
|---|---|---|---|---|---|---|---|---|---|---|
| Parameter | | DF | Estimate | Standard<br>Error | | _ | Cohen's<br>h | OR | Upper CI | Lower CI |
| Intercept | | 1 | XX.XXX | XX.XXX | XX.XXX | 0.xxx | | | | |
| Treatment | Horizant | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | 0.xxx | XX.XXX | XX.XXX | XX.XXX |
| Site | Overall | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | | | | |
| Site | 1 | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | | XX.XXX | XX.XXX | XX.XXX |
| Site | 210 | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | | XX.XXX | XX.XXX | XX.XXX |
| Cov | | X | XX.XXX | xx.xxx | XX.XXX | 0.xxx | | XX.XXX | XX.XXX | XX.XXX |

<sup>&</sup>lt;sup>a</sup>Missing day imputed as a heavy drinking day

Table 33: Subjects with No Heavy Drinking Days (Evaluable) – Full Model, Logistic Regression, Weeks 22-25, with Imputation

Same as Table 32 only using evaluable subjects.

| 12.1.4. Secondary | Efficacy | <b>Endpoints</b> |
|-------------------|----------|------------------|
|-------------------|----------|------------------|

Table 34: Percent Subjects Abstinent from Alcohol (mITT) – Weeks 22-25, With Imputation<sup>a</sup>

| | Placebo (N=xx) | HORIZANT (N=xx) | Total (N=xxx) |
|------------|----------------|-----------------|---------------|
| Completely | | | |
| Abstinent | | | |
| Yes | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| No | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |

<sup>&</sup>lt;sup>a</sup> Missing data imputed as a drinking day

Table 35: Subjects Abstinent from Alcohol (mITT) – Full Model, Logistic Regression, Weeks 22-25, With Imputation<sup>a</sup>

| | | | | | | | | | 95% | 6 CI |
|---|---|---|---|---|---|---|---|---|---|---|
| Parameter | | DF | Estimate | Standard<br>Error | Wald Chi-<br>Square | Pr > Chi-<br>Square | Cohen's<br>h | OR | Upper CI | Lower CI |
| Intercept | | 1 | XX.XXX | XX.XXX | XX.XXX | 0.xxx | | | | |
| Treatment | Horizant | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | 0.xxx | XX.XXX | XX.XXX | XX.XXX |
| Site | Overall | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | | | | |
| Site | 1 | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | | XX.XXX | XX.XXX | XX.XXX |
| Site | 210 | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | | xx.xxx | XX.XXX | XX.XXX |
| Cov | | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | | xx.xxx | XX.XXX | XX.XXX |

<sup>&</sup>lt;sup>a</sup> Missing data imputed as a drinking day

Table 36: Percent Subjects Abstinent from Alcohol (Evaluable) – Weeks 22-25, With Imputation<sup>a</sup> Same as Table 36 only using evaluable subjects.

Table 37: Subjects Abstinent from Alcohol (Evaluable) – Full Model, Logistic Regression, Weeks 22-25, with Imputation<sup>a</sup> Same as Table 37 only using evaluable subjects.

**Table 38:** WHO Shift Baseline to Weeks 22-25, No Imputation

| Baseline | | V | Week 22-25 Category mITT Subjects | / <sup>a</sup> | |
|---|---|---|---|---|---|
| Category | Abstinent | Abstinent Low Risk Medium Risk High Risk Very High Risk | | | |
| | n (%) | n (%) | n (%) | n (%) | n (%) |
| High Risk | | | | | |
| Very High Risk | | | | | |

<sup>&</sup>lt;sup>a</sup> Percent is based upon row denominator (eg # subjects with High Risk at baseline)

Same table for Horizant subjects only

Same table for Placebo subjects only

Table 39: WHO 1-Level Decrease in Alcohol Consumption (mITT) – Weeks 22-25, No Imputation

| Placebo<br>(N=xx) | HORIZANT (N=xx) | Total<br>(N=xxx) |
|---|---|---|
| xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | (N=xx)<br>xx (xx.x%) | (N=xx) (N=xx) xx (xx.x%) xx (xx.x%) |

Table 40: WHO 1-Level Decrease in Alcohol Consumption (mITT) – Full Model, Logistic Regression, Weeks 22-25, No Imputation

| | | | | | | | | | 95% | ∕₀ CI |
|---|---|---|---|---|---|---|---|---|---|---|
| Parameter | | DF | Estimate | Standard<br>Error | Wald Chi-<br>Square | Pr > Chi-<br>Square | Cohen's<br>h | OR | Upper CI | Lower CI |
| Intercept | | 1 | XX.XXX | XX.XXX | XX.XXX | 0.xxx | | | | |
| Treatment | Horizant | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | 0.xxx | XX.XXX | XX.XXX | XX.XXX |
| Site | Overall | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | | | | |

| | | | | | | | | | 95% | 6 CI |
|---|---|---|---|---|---|---|---|---|---|---|
| Paramet | er | DF | Estimate | Standard<br>Error | Wald Chi-<br>Square | Pr > Chi-<br>Square | Cohen's<br>h | OR | Upper CI | Lower CI |
| Site | 1 | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | | XX.XXX | XX.XXX | XX.XXX |
| Site | 210 | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | | XX.XXX | XX.XXX | XX.XXX |
| Cov | | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | | XX.XXX | XX.XXX | XX.XXX |

Table 41: WHO 1-Level Decrease in Alcohol Consumption (Evaluable) – Weeks 22-25, No Imputation Same as Table 39 only using evaluable subjects.

Table 42: WHO 1-Level Decrease in Alcohol Consumption (Evaluable) – Full Model, Logistic Regression, Weeks 22-25, No Imputation

Same as Table 40 only using evaluable subjects.

Table 43: WHO 2-Level Decrease in Alcohol Consumption (mITT) – Weeks 22-25, No Imputation

| | Placebo<br>(N=xx) | HORIZANT (N=xx) | Total<br>(N=xxx) |
|---|---|---|---|
| WHO 2-Level Decrease | | | |
| Yes | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| No | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |

Table 44: WHO 2-Level Decrease in Alcohol Consumption (mITT) – Full Model, Logistic Regression, Weeks 22-25, No Imputation

| | | | | | | | | | | 95% CI |
|---|---|---|---|---|---|---|---|---|---|---|
| Parameter | | DF | Estimate | Standard<br>Error | Wald Chi-<br>Square | Pr > Chi-<br>Square | Cohen's<br>h | OR | Upper CI | Lower CI |
| Intercept | | 1 | XX.XXX | XX.XXX | XX.XXX | 0.xxx | | | | |
| Treatment | Horizant | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | 0.xxx | XX.XXX | XX.XXX | XX.XXX |
| Site | Overall | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | | | | |
| Site | 1 | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | | XX.XXX | XX.XXX | XX.XXX |
| Site | 210 | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | | XX.XXX | XX.XXX | XX.XXX |
| Cov | | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | | XX.XXX | XX.XXX | XX.XXX |

Table 45: WHO 2-Level Decrease in Alcohol Consumption (Evaluable) – Weeks 22-25, No Imputation

Same as Table 43 only using evaluable subjects.

Table 46: WHO 2-Level Decrease in Alcohol Consumption (Evaluable) – Full Model, Logistic Regression, Weeks 22-25, No Imputation

Same as Table 44 only using evaluable subjects.

Table 47: Percentage of Days Abstinent per Week (mITT) -- Full Model, Mixed Effects, Transformed, Weeks 22-25, No Imputation

**Type III Wald Tests** 

| Parameter | Num DF | Den DF | F Value | p-value |
|-----------|--------|--------|---------|---------|
| ARM | 1 | XXX | XXX.XX | 0.xxx |
| Week | 3 | XXX | XXX.XX | 0.xxx |
| Site | 9 | XXX | XXX.XX | 0.xxx |
| Cov | X | XXX | XXX.XX | 0.xxx |
| ARM*Week | 3 | XXX | XXX.XX | 0.xxx |

**Least Squares Means** 

| | | | | 95% CI | | 95% CI | | | | | sformed | Transformed |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Arm | Week | Estimate | SE | Lower CI | Upper CI | Difference | SE | p-value | Cohen's d | p-value | Cohen's d | |
| HORIZANT | 22 | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | X.XXX | 0.xxx | XX.XXX | 0.xxx | XX.XXX | |
| Placebo | 22 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | | | | |
| HORIZANT | 23 | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | x.xxx | 0.xxx | XX.XXX | 0.xxx | XX.XXX | |
| Placebo | 23 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | | | | |
| HORIZANT | 24 | xx.xx | 0.xxx | 0.xxx | 0.xxx | X.XXX | x.xxx | 0.xxx | XX.XXX | 0.xxx | XX.XXX | |
| Placebo | 24 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | | | | |
| HORIZANT | 25 | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | x.xxx | 0.xxx | XX.XXX | 0.xxx | XX.XXX | |
| Placebo | 25 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | | | | |
| HORIZANT | Overall | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | X,XXX | 0.xxx | XX.XXX | 0.xxx | XX.XXX | |
| Placebo | Overall | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | | | | |

Table 48: Percentage of Days Abstinent per Week (Evaluable) -- Full Model, Mixed Effects, Transformed, Weeks 22-25, No Imputation

Same as Table 47 only using evaluable subjects.

Table 49: Percentage of Days Abstinent per Week (mITT) – Untransformed, Weeks 2-25, No Imputation

| | HORIZANT | | | | | | | | Pl | acebo | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Week | N | Mean | SD | Median | Min | Max | N | Mean | SD | Median | Min | Max |
| 2 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 3 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 4 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 5 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 6 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 7 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 8 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 9 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 10 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 11 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 12 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 13 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 14 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 15 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 16 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 17 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 18 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 19 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 20 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 21 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 22 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 23 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 24 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 25 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |

Table 50: Percentage of Days Abstinent per Week (Evaluable) – Untransformed, Weeks 2-25, No Imputation Same as Table 49 only using evaluable subjects.

Table 51: Percentage of Heavy Drinking Days per Week (mITT) – Full Model, Mixed Effects, Transformed, Weeks 22-25, No Imputation

**Type III Wald Tests** 

| Parameter | Num DF | Den DF | F Value | p-value |
|-----------|--------|--------|---------|---------|
| ARM | 1 | XXX | XXX.XX | 0.xxx |
| Week | 3 | XXX | XXX.XX | 0.xxx |
| Site | 9 | XXX | XXX.XX | 0.xxx |
| Cov | X | XXX | XXX.XX | 0.xxx |
| ARM*Week | 3 | XXX | XXX.XX | 0.xxx |

**Least Squares Means** 

| | | | | 95% CI | | 95% CI | | | | | sformed | Transformed |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Arm | Week | Estimate | SE | Lower CI | Upper CI | Difference | SE | p-value | Cohen's d | p-value | Cohen's d | |
| HORIZANT | 22 | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | X.XXX | 0.xxx | XX.XXX | 0.xxx | XX.XXX | |
| Placebo | 22 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | | | | |
| HORIZANT | 23 | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | x.xxx | 0.xxx | XX.XXX | 0.xxx | XX.XXX | |
| Placebo | 23 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | | | | |
| HORIZANT | 24 | xx.xx | 0.xxx | 0.xxx | 0.xxx | X.XXX | x.xxx | 0.xxx | XX.XXX | 0.xxx | XX.XXX | |
| Placebo | 24 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | | | | |
| HORIZANT | 25 | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | x.xxx | 0.xxx | XX.XXX | 0.xxx | XX.XXX | |
| Placebo | 25 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | | | | |
| HORIZANT | Overall | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | X,XXX | 0.xxx | XX.XXX | 0.xxx | XX.XXX | |
| Placebo | Overall | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | | | | |

Table 52: Percentage of Heavy Drinking Days per Week (Evaluable) – Full Model, Mixed Effects, Transformed, Weeks 22-25, No Imputation

Same as Table 51 only with evaluable subjects.

Table 53: Percentage of Heavy Drinking Days per Week (mITT) – Untransformed, Weeks 2-25, No Imputation

| | HORIZANT | | | | | | | | Pl | acebo | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Week | N | Mean | SD | Median | Min | Max | N | Mean | SD | Median | Min | Max |
| 2 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 3 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 4 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 5 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 6 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 7 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 8 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 9 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 10 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 11 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 12 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 13 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 14 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 15 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 16 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 17 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 18 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 19 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 20 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 21 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 22 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 23 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 24 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 25 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |

Table 54: Percentage of Heavy Drinking Days per Week (Evaluable) – Untransformed, Weeks 2-25, No Imputation Same as Table 53 only using evaluable subjects.

Table 55: Drinks per Week (mITT) – Full Model, Mixed Effects, Transformed, Weeks 22-25, No Imputation
Type III Wald Tests

| Parameter | Num DF | Den DF | F Value | p-value |
|-----------|--------|--------|---------|---------|
| ARM | 1 | XXX | XXX.XX | 0.xxx |
| Week | 3 | XXX | XXX.XX | 0.xxx |
| Site | 9 | XXX | XXX.XX | 0.xxx |
| Cov | X | XXX | XXX.XX | 0.xxx |
| ARM*Week | 3 | XXX | XXX.XX | 0.xxx |

**Least Squares Means** 

| | | | | 95% CI | | | | Untransformed | | Transformed | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Arm | Week | Estimate | SE | Lower CI | Upper CI | Difference | SE | p-value | Cohen's d | p-value | Cohen's d |
| HORIZANT | 22 | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | X,XXX | 0.xxx | XX.XXX | 0.xxx | XX.XXX |
| Placebo | 22 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | | | |
| HORIZANT | 23 | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | x.xxx | 0.xxx | XX.XXX | 0.xxx | XX.XXX |
| Placebo | 23 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | | | |
| HORIZANT | 24 | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | x.xxx | 0.xxx | XX.XXX | 0.xxx | XX.XXX |
| Placebo | 24 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | | | |
| HORIZANT | 25 | xx.xx | 0.xxx | 0.xxx | 0.xxx | X.XXX | x.xxx | 0.xxx | XX.XXX | 0.xxx | XX.XXX |
| Placebo | 25 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | | | |
| HORIZANT | Overall | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | x.xxx | 0.xxx | XX.XXX | 0.xxx | XX.XXX |
| Placebo | Overall | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | | | |

Table 56: Drinks per Week (Evaluable) – Full Model, Mixed Effects, Transformed, Weeks 22-25, No Imputation Same as Table 55 only using evaluable subjects.

Table 57: Drinks per Week (mITT) – Untransformed, Weeks 2-25, No Imputation

| | | | Н | ORIZANT | | | Placebo | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Week | N | Mean | SD | Median | Min | Max | N | Mean | SD | Median | Min | Max |
| 2 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 3 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 4 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 5 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 6 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 7 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 8 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 9 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 10 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 11 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 12 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 13 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 14 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 15 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 16 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 17 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 18 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 19 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 20 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 21 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 22 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 23 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 24 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 25 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |

Table 58: Drinks per Week (Evaluable) – Untransformed, Weeks 2-25, No Imputation

Same as Table 57 only using evaluable subjects.

Table 59: Drinks per Drinking Day (mITT) – Full Model, Mixed Effects, Transformed, Weeks 22-25, No Imputation
Type III Wald Tests

| Parameter | Num DF | Den DF | F Value | p-value |
|-----------|--------|--------|---------|---------|
| ARM | 1 | XXX | XXX.XX | 0.xxx |
| Week | 3 | XXX | XXX.XX | 0.xxx |
| Site | 9 | XXX | XXX.XX | 0.xxx |
| Cov | X | XXX | XXX.XX | 0.xxx |
| ARM*Week | 3 | XXX | XXX.XX | 0.xxx |

**Least Squares Means** 

| | | | | 95% | 95% CI | | | Untransformed | | Transformed | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Arm | Week | Estimate | SE | Lower CI | Upper CI | Difference | SE | p-value | Cohen's d | p-value | Cohen's d |
| HORIZANT | 22 | xx.xx | 0.xxx | 0.xxx | 0.xxx | X.XXX | X.XXX | 0.xxx | XX.XXX | 0.xxx | XX.XXX |
| Placebo | 22 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | | | |
| HORIZANT | 23 | xx.xx | 0.xxx | 0.xxx | 0.xxx | X.XXX | x.xxx | 0.xxx | XX.XXX | 0.xxx | XX.XXX |
| Placebo | 23 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | | | |
| HORIZANT | 24 | xx.xx | 0.xxx | 0.xxx | 0.xxx | X.XXX | x.xxx | 0.xxx | XX.XXX | 0.xxx | XX.XXX |
| Placebo | 24 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | | | |
| HORIZANT | 25 | xx.xx | 0.xxx | 0.xxx | 0.xxx | X.XXX | X.XXX | 0.xxx | XX.XXX | 0.xxx | XX.XXX |
| Placebo | 25 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | | | |
| HORIZANT | Overall | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | X.XXX | 0.xxx | XX.XXX | 0.xxx | XX.XXX |
| Placebo | Overall | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | | | |

Table 60: Drinks per Drinking Day (Evaluable) – Full Model, Mixed Effects, Transformed, Weeks 22-25, No Imputation Same as Table 59 only using evaluable subjects.

Table 61: Drinks per Drinking Day (mITT) – Untransformed, Weeks 2-25, No Imputation

| HORIZANT | | | | | | | | | Pl | acebo | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Week | N | Mean | SD | Median | Min | Max | N | Mean | SD | Median | Min | Max |
| 2 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 3 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 4 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 5 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 6 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 7 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 8 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 9 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 10 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 11 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 12 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 13 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 14 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 15 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 16 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 17 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 18 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 19 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 20 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 21 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 22 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 23 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 24 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 25 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |

**Table 62: Drinks per Drinking Day (Evaluable) – Untransformed, Weeks 2-25, No Imputation** Same as Table 61 only using evaluable subjects.

Table 63: ACQ-SR-R Score (mITT) – Full Model, Mixed Effects, Transformed, Weeks 24 + 26 (covering last 4 weeks of maintenance phase), No Imputation

**Type III Wald Tests** 

| Parameter | Num DF | Den DF | F Value | p-value |
|-----------|--------|--------|---------|---------|
| ARM | 1 | XXX | XXX.XX | 0.xxx |
| Week | 1 | XXX | XXX.XX | 0.xxx |
| Site | 9 | XXX | XXX.XX | 0.xxx |
| Cov | X | XXX | XXX.XX | 0.xxx |
| ARM*Week | 1 | XXX | XXX.XX | 0.xxx |

**Least Squares Means** 

| | | | | 95% | | | Untransformed | | Transformed | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Arm | Week | Estimate | SE | Lower CI | Upper CI | Difference | SE | p-value | Cohen's d | p-value | Cohen's d |
| HORIZANT | 24 | xx.xx | 0.xxx | 0.xxx | 0.xxx | X.XXX | x.xxx | 0.xxx | XX.XXX | 0.xxx | XX.XXX |
| Placebo | 24 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | | | |
| HORIZANT | 26 | xx.xx | 0.xxx | 0.xxx | 0.xxx | X.XXX | x.xxx | 0.xxx | XX.XXX | 0.xxx | XX.XXX |
| Placebo | 26 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | | | |
| HORIZANT | Overall | xx.xx | 0.xxx | 0.xxx | 0.xxx | X.XXX | x.xxx | 0.xxx | XX.XXX | 0.xxx | XX.XXX |
| Placebo | Overall | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | | | |

Table 64: ACQ-SR-R Score (Evaluable) – Full Model, Mixed Effects, Transformed, Weeks 24 + 26 (covering last 4 weeks of maintenance phase), No Imputation

Same as Table 63 only using evaluable subjects.

Table 65: ACQ-SR-R Score (mITT) – Untransformed, Each Evaluation During Maintenance Period, No Imputation

| | HORIZANT | | | | | | | Placebo | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Week | N | Mean | SD | Median | Min | Max | N | Mean | SD | Median | Min | Max |
| 2 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 4 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 6 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 8 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 10 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 12 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 16 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 20 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 24 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 26 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |

Table 66: ACQ-SR-R Score (Evaluable) – Untransformed, Each Evaluation During Maintenance Period, No Imputation Same as Table 65 only using evaluable subjects.

Table 67: ImBIBe Score (mITT) – Full Model, Mixed Effects, Transformed, Weeks 24 + 26 (covering last 4 weeks of maintenance phase), No Imputation

**Type III Wald Tests** 

| Parameter | Num DF | Den DF | F Value | p-value |
|-----------|--------|--------|---------|---------|
| ARM | 1 | XXX | XXX.XX | 0.xxx |
| Week | 1 | XXX | XXX.XX | 0.xxx |
| Site | 9 | XXX | XXX.XX | 0.xxx |
| Cov | X | XXX | XXX.XX | 0.xxx |
| ARM*Week | 1 | XXX | XXX.XX | 0.xxx |

**Least Squares Means** 

| | | | | 95% CI | | | | Untransformed | | Transformed | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Arm | Week | Estimate | SE | Lower CI | Upper CI | Difference | SE | p-value | Cohen's d | p-value | Cohen's d |
| HORIZANT | 24 | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | X.XXX | 0.xxx | XX.XXX | 0.xxx | XX.XXX |
| Placebo | 24 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | | | |
| HORIZANT | 26 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | XX.XXX | 0.xxx | XX.XXX |
| Placebo | 26 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | | | |
| HORIZANT | Overall | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | XX.XXX | 0.xxx | XX.XXX |
| Placebo | Overall | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | | | |

Table 68: ImBIBe Score (Evaluable) – Full Model, Mixed Effects, Transformed, Weeks 24 + 26 (covering last 4 weeks of maintenance phase), No Imputation

Same as Table 67 only using evaluable subjects.

Table 69: ImBIBe Score (mITT) – Untransformed, Each Evaluation During Maintenance Period, No Imputation

HORIZANT Placebo Study Week Max N Median N Mean SD Median Min Mean SD Min Max XXXXX XXXXXXXXXXXX XXX XXXXXXXXXXXX XXX8 XXXXX XXXXXXXXX XXX XXXXXXXXXXXX XXXXXX12 XXXXXXXXXXXXXXXXXXXX XXXXXXXXXXXXXXX16 XXXXXXXXXXXXXXXXXXXX XXXXXXXXXXXXXXX20 XXXXX XXXXXXXXXXXXXXX XXXXXXXXXXXXXXX24 XX XXXXXXXXXXXXXXXXXX XXXXXXXXXXXXXXX26 XX XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX

Table 70: ImBIBe Score (Evaluable) – Untransformed, Each Evaluation During Maintenance Period, No Imputation Same as Table 69 only using evaluable subjects.

Table 71: Mean Cigarettes Smoked (mITT) – Full Model, Mixed Effects, Transformed, Weeks 24 + 26 (covering last 4 weeks of maintenance phase), No Imputation

**Type III Wald Tests** 

| Parameter | Num DF | Den DF | F Value | p-value |
|-----------|--------|--------|---------|---------|
| ARM | 1 | XXX | XXX.XX | 0.xxx |
| Week | 1 | XXX | XXX.XX | 0.xxx |
| Site | 9 | XXX | XXX.XX | 0.xxx |
| Cov | X | XXX | XXX.XX | 0.xxx |
| ARM*Week | 1 | XXX | XXX.XX | 0.xxx |

**Least Squares Means** 

| | | | | 95% CI | | | | Untransformed | | Transformed | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Arm | Week | Estimate | SE | Lower CI | Upper CI | Difference | SE | p-value | Cohen's d | p-value | Cohen's d |
| HORIZANT | 24 | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | X.XXX | 0.xxx | XX.XXX | 0.xxx | XX.XXX |
| Placebo | 24 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | | | |
| HORIZANT | 26 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | XX.XXX | 0.xxx | XX.XXX |
| Placebo | 26 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | | | |
| HORIZANT | Overall | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | XX.XXX | 0.xxx | XX.XXX |
| Placebo | Overall | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | | | |

Table 72: Mean Cigarettes Smoked (Evaluable) – Full Model, Mixed Effects, Transformed, Weeks 24 + 26 (covering last 4 weeks of maintenance phase), No Imputation

Same as Table 71 only using evaluable subjects.
Table 73: Mean Cigarettes Smoked (mITT) – Untransformed, Each Evaluation During Maintenance Period, No Imputation

| | | | H | ORIZANT | | | | | Pla | acebo | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Week | N | Mean | SD | Median | Min | Max | N | Mean | SD | Median | Min | Max |
| 2 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 4 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 6 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 8 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 10 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 12 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 16 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 20 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 24 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 26 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |

Table 74: Mean Cigarettes Smoked (Evaluable) – Untransformed, Each Evaluation During Maintenance Period, No Imputation

Same as Table 73 only using evaluable subjects.

Table 75: PSQI Score (mITT) – Full Model, Mixed Effects, Transformed, Weeks 24 + 26 (covering last 4 weeks of maintenance phase), No Imputation

**Type III Wald Tests** 

| Parameter | Num DF | Den DF | F Value | p-value |
|-----------|--------|--------|---------|---------|
| ARM | 1 | XXX | XXX.XX | 0.xxx |
| Week | 1 | XXX | XXX.XX | 0.xxx |
| Site | 9 | XXX | XXX.XX | 0.xxx |
| Cov | X | XXX | XXX.XX | 0.xxx |
| ARM*Week | 1 | XXX | XXX.XX | 0.xxx |

**Least Squares Means** 

| | | | | 95% CI | | 95% CI | | Untran | sformed | Tran | sformed |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Arm | Week | Estimate | SE | Lower CI | Upper CI | Difference | SE | p-value | Cohen's d | p-value | Cohen's d |
| HORIZANT | 24 | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | X.XXX | 0.xxx | XX.XXX | 0.xxx | XX.XXX |
| Placebo | 24 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | | | |
| HORIZANT | 26 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | XX.XXX | 0.xxx | XX.XXX |
| Placebo | 26 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | | | |
| HORIZANT | Overall | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | XX.XXX | 0.xxx | XX.XXX |
| Placebo | Overall | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | | | |

Table 76: PSQI Score (Evaluable) – Full Model, Mixed Effects, Transformed, Weeks 24 + 26 (covering last 4 weeks of maintenance phase), No Imputation

Same as Table 75 using only evaluable subjects.

Table 77: PSQI Score (mITT) – Untransformed, Each Evaluation During Maintenance Period, No Imputation

| | HORIZANT | | | | | | | Placebo | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Week | N | Mean | SD | Median | Min | Max | N | Mean | SD | Median | Min | Max |
| 4 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 8 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 12 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 16 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 20 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 24 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 26 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |

Table 78: PSQI Score (Evaluable) – Untransformed, Each Evaluation During Maintenance Period, No Imputation Same as Table 77 using only evaluable subjects.

Table 79: PSQI Sleep Quality Score (mITT) – Full Model, Mixed Effects, Transformed, Weeks 24 + 26 (covering last 4 weeks of maintenance phase), No Imputation

Same method as Table 75.

- Table 80: PSQI Sleep Quality Score (Evaluable) Full Model, Mixed Effects, Transformed, Weeks 24 + 26 (covering last 4 weeks of maintenance phase), No Imputation
- Table 81: PSQI Sleep Quality Score (mITT) Untransformed, Each Evaluation During Maintenance Period, No Imputation
- Table 82: PSQI Sleep Quality Score (Evaluable) Untransformed, Each Evaluation During Maintenance Period, No Imputation
- Table 83: PSQI Sleep Latency Score (mITT) Full Model, Mixed Effects, Transformed, Weeks 24 + 26 (covering last 4 weeks of maintenance phase), No Imputation
- Table 84: PSQI Sleep Latency Score (Evaluable) Full Model, Mixed Effects, Transformed, Weeks 24 + 26 (covering last 4 weeks of maintenance phase), No Imputation
- Table 85: PSQI Sleep Latency Score (mITT) Untransformed, Each Evaluation During Maintenance Period, No Imputation
- Table 86: PSQI Sleep Latency Score (Evaluable) Untransformed, Each Evaluation During Maintenance Period, No Imputation
- Table 87: PSQI Sleep Duration Score (mITT) Full Model, Mixed Effects, Transformed, Weeks 24 + 26 (covering last 4 weeks of maintenance phase), No Imputation
- Table 88: PSQI Sleep Duration Score (Evaluable) Full Model, Mixed Effects, Transformed, Weeks 24 + 26 (covering last 4 weeks of maintenance phase), No Imputation
- Table 89: PSQI Sleep Duration Score (mITT) Untransformed, Each Evaluation During Maintenance Period, No Imputation
- Table 90: PSQI Sleep Duration Score (Evaluable) Untransformed, Each Evaluation During Maintenance Period, No Imputation
- Table 91: PSQI Sleep Disturbance Score (mITT) Full Model, Mixed Effects, Transformed, Weeks 24 + 26 (covering last 4 weeks of maintenance phase), No Imputation
- Table 92: PSQI Sleep Disturbance Score (Evaluable) Full Model, Mixed Effects, Transformed, Weeks 24 + 26 (covering last 4 weeks of maintenance phase), No Imputation

Table 93: PSQI Sleep Disturbance Score (mITT) – Untransformed, Each Evaluation During Maintenance Period, No Imputation

Table 94: PSQI Sleep Disturbance Score (Evaluable) – Untransformed, Each Evaluation During Maintenance Period, No Imputation

- Table 95: PSQI Use of Sleep Medication Score (mITT) Full Model, Mixed Effects, Transformed, Weeks 24 + 26 (covering last 4 weeks of maintenance phase), No Imputation
- Table 96: PSQI Use of Sleep Medication Score (Evaluable) Full Model, Mixed Effects, Transformed, Weeks 24 + 26 (covering last 4 weeks of maintenance phase), No Imputation
- Table 97: PSQI Use of Sleep Medication Score (mITT) Untransformed, Each Evaluation During Maintenance Period, No Imputation
- Table 98: PSQI Use of Sleep Medication Score (Evaluable) Untransformed, Each Evaluation During Maintenance Period, No Imputation
- Table 99: PSQI Daytime Dysfunction Score (mITT) Full Model, Mixed Effects, Transformed, Weeks 24 + 26 (covering last 4 weeks of maintenance phase), No Imputation
- Table 100: PSQI Daytime Dysfunction Score (Evaluable) Full Model, Mixed Effects, Transformed, Weeks 24 + 26 (covering last 4 weeks of maintenance phase), No Imputation
- Table 101: PSQI Daytime Dysfunction Score (mITT) Untransformed, Each Evaluation During Maintenance Period, No Imputation
- Table 102: PSQI Daytime Dysfunction Score (Evaluable) Untransformed, Each Evaluation During Maintenance Period, No Imputation
- Table 103: BAI Score (mITT) Full Model, Mixed Effects, Transformed, Weeks 24 + 26 (covering last 4 weeks of maintenance phase), No Imputation
- Table 104: BAI Score (Evaluable) Full Model, Mixed Effects, Transformed, Weeks 24 + 26 (covering last 4 weeks of maintenance phase), No Imputation
- Table 105: BAI Score (mITT) Untransformed, Each Evaluation During Maintenance Period, No Imputation
- Table 106: BAI Score (Evaluable) Untransformed, Each Evaluation During Maintenance Period, No Imputation
- Table 107: BDI-II Score (mITT) Full Model, Mixed Effects, Transformed, Weeks 24 + 26 (covering last 4 weeks of maintenance phase), No Imputation
- Table 108: BDI-II Score (Evaluable) Full Model, Mixed Effects, Transformed, Weeks 24 + 26 (covering last 4 weeks of maintenance phase), No Imputation
- Table 109: BDI-II Score (mITT) Untransformed, Each Evaluation During Maintenance Period, No Imputation

| Table 110: | BDI-II Score (Evaluable) – Untransformed, Each Evaluation During Maintenance Period, No Imputation |
|---|---|

## 12.1.5. Safety Analyses

Overall Summary of Adverse Events – mITT Subjects **Table 111:** 

| Disposition | Placebo<br>(N=xx) | HORIZANT (N=xx) | Total<br>(N=xxx) | p-value <sup>1</sup> |
|---|---|---|---|---|
| Subjects reporting at least one Adverse Event | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | 0.xxx |
| Subjects reporting at least one Severe Adverse Event | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | 0.xxx |
| Subjects reporting at least one Treatment–Related <sup>2</sup> Adverse Event | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | 0.xxx |
| Subjects reporting at least one Treatment–Related Severe Adverse Event | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | 0.xxx |
| Subjects reporting at least one Serious Adverse Event | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | 0.xxx |
| Subjects reporting at least one Treatment–Related Serious Adverse Event | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | 0.xxx |
| Subjects who Discontinued Medication due to an Adverse Event | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | 0.xxx |
| Subjects who Died due to an Adverse Event | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | 0.xxx |

**Table 112:** Number and Percentage of Subjects with Adverse Events - mITT Subjects

| MedDRA System Organ Class/<br>Preferred Term | Placebo<br>(N=xx) | HORIZANT (N=xx) | p-value <sup>1</sup> |
|---|---|---|---|
| - Any Adverse Events - | xx (xx.x%) | xx (xx.x%) | 0.xxx |
| SOC | | | |
| - Overall - | xx (xx.x%) | xx (xx.x%) | 0.xxx |
| Preferred term 1 | xx (xx.x%) | xx (xx.x%) | |
| Preferred term 2 | xx (xx.x%) | xx (xx.x%) | |

Notes: Percentages are based on the total number of subjects, as given in the column heading.

Multiple occurrences of a specific adverse event for a subject are counted once in the frequency for the adverse event. Likewise, multiple occurrences of adverse events within a specific preferred term for a subject are counted once in the frequency for the preferred term.

<sup>&</sup>lt;sup>1</sup> p-value from chi-square test (c), unless a row has fewer than 5 in a cell then Fisher's exact test (f)
<sup>2</sup> Treatment related is defined as an adverse event that is possibly, probably, or definitely related to treatment

<sup>&</sup>lt;sup>1</sup> Fisher's exact test

Table 113: Summary of Subjects with Adverse Events by Severity and Relationship – HORIZANT

| Number of Subjects (%) (N=x) | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Mild Moderate Severe Life-threatening All Grades | | | | | | | | | | | | |
| SOC | MedDRA<br>PT | R | NR | R | NR | R | NR | R | NR | R | NR | R + NR |
| | | XX<br>(XX.X%) | xx<br>(xx.x%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | xx<br>(xx.x%) | xx<br>(xx.x%) | xx<br>(xx.x%) | XX<br>(XX.X%) | XX<br>(XX.X%) |

Notes: Events are counted once per subject at the highest severity grade and closest relationship to the investigational product. R= related to investigational product (possibly, probably, definitely). NR = not related to investigational product (unrelated, unlikely).

Table 114: Summary of Subjects with Adverse Events by Severity and Relationship – Placebo

| Number of Subjects (%) (N=x) | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Mild Moderate Severe Life-threatening All Grades | | | | | | | | | | | | |
| SOC | MedDRA<br>PT | R | NR | R | NR | R | NR | R | NR | R | NR | R + NR |
| | | XX<br>(XX.X%) | xx<br>(xx.x%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | XX<br>(XX.X%) | xx<br>(xx.x%) | XX<br>(XX.X%) | XX<br>(XX.X%) | xx<br>(xx.x%) |

Notes: Events are counted once per subject at the highest severity grade and closest relationship to the investigational product. R= related to investigational product (possibly, probably, definitely). NR = not related to investigational product (unrelated, unlikely).

Table 115: Number and Percentage of Subjects with Adverse Events by Maximum Severity - mITT Subjects

MedDRA SOC/<br/>Preferred TermPlacebo<br/>(N=xx)HORIZANT<br/>(N=xx)

| | Mild | Moderate | Severe | Life-<br>threatening | Mild | Moderate | Severe | Life-<br>threatening |
|---|---|---|---|---|---|---|---|---|
| | | Moderate | Bevere | till catelling | TVIIIG | Moderate | Severe | tilleatening |
| - Any Adverse Events - SOC | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| - Overall - | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Preferred term 1 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Preferred term 2 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |

Notes: Percentages are based on the total number of subjects, as given in the column heading.

Multiple occurrences of a specific adverse event for a subject are counted once in the frequency for the adverse event. Likewise, multiple occurrences of adverse events within a specific preferred term for a subject are counted once in the frequency for the preferred term.

Table 116: Number and Percentage of Subjects Adverse Events by Relatedness - mITT Subjects

| MedDRA SOC/<br>Preferred Term | | cebo<br>=xx) | HORIZANT<br>(n=xx) | |
|---|---|---|---|---|
| | Related <sup>1</sup> | Not-Related <sup>2</sup> | Related | Not-Related |
| SOC<br>- Overall - | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Preferred term 1 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Preferred term 2 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn(xx.x%) |

<sup>&</sup>lt;sup>1</sup>Related are possibly, probably or definitely related to investigational product

<sup>&</sup>lt;sup>2</sup> Not Related to investigational product (not related or unlikely)

Table 117: Number and Percentage of Subjects with Treatment-Related Adverse Events by Maximum Severity- mITT Subjects

| MedDRA SOC/ | Placebo | HORIZANT |
|----------------|---------|----------|
| Preferred Term | (N=xx) | (N=xx) |

| | | | | Life- | | | | Life- |
|---|---|---|---|---|---|---|---|---|
| | Mild | Moderate | Severe | threatening | Mild | Moderate | Severe | threatening |
| SOC<br>- Overall - | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Preferred term 1 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Preferred term 2 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |

Notes: Percentages are based on the total number of subjects, as given in the column heading.

Multiple occurrences of a specific adverse event for a subject are counted once in the frequency for the adverse event. Likewise, multiple occurrences of adverse events within a specific preferred term for a subject are counted once in the frequency for the preferred term.

Programmer's Notes: Order System Organ Class alphabetically and preferred term alphabetically within System Organ Class.

Table 118: Number and Percentage of Subjects with Adverse Events Occurring in >= 5% - mITT Subjects

| MedDRA SOC/ | Placebo | HORIZANT | p-value <sup>1</sup> |
|--------------------|------------|------------|----------------------|
| Preferred Term | (N=xx) | (N=xx) | |
| SOC<br>- Overall - | nn (xx.x%) | nn (xx.x%) | 0.xxx |
| Preferred term 1 | nn (xx.x%) | nn (xx.x%) | 0.xxx |
| Preferred term 2 | nn (xx.x%) | nn (xx.x%) | 0.xxx |

Notes: Percentages are based on the total number of subjects, as given in the column heading.

Multiple occurrences of a specific adverse event for a subject are counted once in the frequency for the adverse event. Likewise, multiple occurrences of adverse events within a specific preferred term for a subject are counted once in the frequency for the preferred term. At least 5% occurring in either arm to be included in the table.

1 Fisher's Exact test

Table 119: Number and Percentage of Subjects with Adverse Events Leading to Discontinuation of Study - mITT Subjects

| MedDRA SOC/<br>Preferred Term | Placebo<br>(N=xx) | HORIZANT (N=xx) |
|-------------------------------|-------------------|-----------------|
| SOC<br>- Overall - | nn (xx.x%) | nn (xx.x%) |
| Preferred term 1 | nn (xx.x%) | nn (xx.x%) |
| Preferred term 2 | nn (xx.x%) | nn (xx.x%) |
| | nn (xx.x%) | nn (xx.x%) |
| | nn (xx.x%) | nn (xx.x%) |
| | nn (xx.x%) | nn (xx.x%) |
| | nn (xx.x%) | nn (xx.x%) |

Notes: Percentages are based on the total number of subjects, as given in the column heading.

Multiple occurrences of a specific adverse event for a subject are counted once in the frequency for the adverse event. Likewise, multiple occurrences of adverse events within a specific preferred term for a subject are counted once in the frequency for the preferred term.

Programmer's Notes: Order System Organ Class alphabetically and preferred term alphabetically within System Organ Class.

Table 120: Number and Percentage of Subjects with Adverse Events Leading to Discontinuation of Study Medication—mITT Subjects

| MedDRA SOC/<br>Preferred Term | Placebo<br>(N=xx) | HORIZANT<br>(N=xx) |
|---------------------------------|-------------------|--------------------|
| SOC<br>- Overall - | nn (xx.x%) | nn (xx.x%) |
| - Overall -<br>Preferred term 1 | nn (xx.x%) | nn (xx.x%) |
| Preferred term 2 | nn (xx.x%) | nn (xx.x%) |
| | nn(xx.x%) | nn (xx.x%) |
| | nn (xx.x%) | nn (xx.x%) |
| | nn (xx.x%) | nn (xx.x%) |
| | nn (xx.x%) | nn (xx.x%) |

Notes: Percentages are based on the total number of subjects, as given in the column heading.

Multiple occurrences of a specific adverse event for a subject are counted once in the frequency for the adverse event. Likewise, multiple occurrences of adverse events within a specific preferred term for a subject are counted once in the frequency for the preferred term.

Table 121: Number and Percentage of Subjects with Somnolence or Dizziness AEs that Started on a Drinking Day – mITT Subjects

| Adverse Event | Placebo<br>(N=xx) | HORIZANT<br>(N=xx) |
|---------------|-------------------|--------------------|
| Somnolence | nn (xx.x%) | nn (xx.x%) |
| Dizziness | nn (xx.x%) | nn (xx.x%) |

**Table 122:** CIWA-AR Score ≥ 10 at Least Once During Treatment – mITT Subjects

| | Placebo | HORIZANT | Total | | | | 95% | o CI |
|---|---|---|---|---|---|---|---|---|
| | (N=xx) | (N=xx) | (N=xxx) | p-value <sup>1</sup> | Cohen's h | Odds Ratio | OR Lower CI | OR Upper CI |
| CIWA-AR Score >= 10 | | | | | | | | |
| Never | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | | | | | |
| At Least Once | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) | 0.xxx | 0.xx | XX.XXX | XX.XXX | XX.XXX |

1 Chi-squared test

Table 123: Summary of Vital Signs and Body Weights – mITT Subjects

| Parameter | N | Mean | SD | Med | Max | Min |
|---------------------------------|----|------|------|------|------|------|
| Vital Sign (units) | | | | | | |
| Screening | | | | | | |
| Placebo | XX | XX.X | XX.X | XX.X | XX.X | XX.X |
| HORIZANT | XX | XX.X | XX.X | XX.X | XX.X | XX.X |
| Week 4 | | | | | | |
| Placebo | XX | XX.X | XX.X | XX.X | XX.X | XX.X |
| HORIZANT | XX | XX.X | XX.X | XX.X | XX.X | XX.X |
| Change from baseline | | | | | | |
| Placebo | XX | XX.X | XX.X | XX.X | XX.X | XX.X |
| HORIZANT | XX | XX.X | XX.X | XX.X | XX.X | XX.X |
| Weeks 8, 12, 16, 20, 24, 26, 27 | | | | | | |

Programmers note: vital signs include pulse rate, systolic blood pressure, and diastolic blood pressure. Body weight (kg) will also be presented.

**Table 124:** Summary of Other Services Used During Treatment Period – mITT Subjects

| | Placebo | HORIZANT | |
|---|---|---|---|
| Services | (N=xx) | (N=xx) | p-value <sup>1</sup> |
| Self Help Meetings | | | 0.xxx |
| N | XX | XX | |
| Mean | XX.X | XX.X | |
| SD | XXX.XX | XXX.XX | |
| Median | XX | XX | |
| Min-Max | (xx-xx) | (xx-xx) | |
| Have you visited another health professional to | | | |
| get help reducing drinking? | | | |
| N | Xx | XX | |
| Yes n (%) | xx (xx) | xx (xx) | |
| Type of Professional | | | |
| A | xx(xx) | xx (xx) | |
| В | xx (xx) | xx (xx) | |
| C | xx (xx) | xx (xx) | |
| Other | xx (xx) | xx (xx) | |

Programmer note: categorize type of professional for those categories reaching 5%

**Table 125:** Summary of ECG Results - mITT Subjects

| Result | Placebo<br>(N=xx) | HORIZANT<br>(N=xx) |
|---|---|---|
| Screening | | |
| Normal | nn(xx.x%) | nn (xx.x%) |
| Abnormal, Not Clinically Significant | nn(xx.x%) | nn (xx.x%) |
| Abnormal, Clinically Significant | nn (xx.x%) | nn (xx.x%) |
| Week 27 | | |
| Normal | nn (xx.x%) | nn (xx.x%) |
| Abnormal, Not Clinically Significant | nn (xx.x%) | nn (xx.x%) |
| Abnormal, Clinically Significant | nn (xx.x%) | nn (xx.x%) |

**Table 126:** Summary of Blood Chemistries – mITT Subjects

| | Placebo | | | HORIZANT | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Test | N | Mean | SD | Med | Min | Max | N | Mean | SD | Med | Min | Max |
| Test Name (units) | | • | | | | | | • | | | | |
| Screening | | | | | | | | | | | | |
| Week 4 | | | | | | | | | | | | |
| Change from baseline | | | | | | | | | | | | |
| Weeks 8, 12, 16, 20, 24, 26, 27 | _ | | _ | | | | | | | _ | | |

Programmers note: table will include creatinine, ALT, AST, total bilirubin, and GGT.

Table 127: Summary of Positive Urine Drug Tests, Preganancy Test or BAC > 0.000 Any Time During the Study– mITT Subjects

| | Number ( | % Positive) |
|-----------------|----------|-------------|
| Test | Placebo | HORIZANT |
| TIMO | ( 0() | ( 0() |
| THC | xx (xx%) | xx (xx%) |
| Cocaine | xx (xx%) | xx (xx%) |
| Opioids | xx (xx%) | xx (xx%) |
| Methamphetamine | xx (xx%) | xx (xx%) |
| Amphetamine | xx (xx%) | xx (xx%) |
| Benzodiazapines | xx (xx%) | xx (xx%) |
| Buprenorphine | xx (xx%) | xx (xx%) |
| Methadone | xx (xx%) | xx (xx%) |
| Pregnancy | xx (xx%) | xx (xx%) |
| BAC > 0.000 | xx (xx%) | xx (xx%) |

Table 128: POMS Total Mood Disturbance Score (mITT) -- Full Model, Mixed Effects, Transformed, Entire Maintenance Period, No Imputation

**Type III Wald Tests** 

| Parameter | Num DF | Den DF | F Value | p-value |
|-------------------------|--------|--------|---------|---------|
| ARM | 1 | XXX | XXX.XX | 0.xxx |
| Week | 6 | XXX | XXX.XX | 0.xxx |
| Site | 9 | XXX | XXX.XX | 0.xxx |
| Baseline<br>Total Score | X | XXX | XXX.XX | 0.xxx |
| ARM*Week | 6 | XXX | xxx.xx | 0.xxx |

**Least Squares Means** 

| | | | | 95% CI | | _ | _ | Untransformed | | Transformed | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Arm | Week | Estimate | SE | Lower CI | Upper CI | Difference | SE | p-value | Cohen's d | p-value | Cohen's d |
| HORIZANT | 4 | xx.xx | 0.xxx | 0.xxx | 0.xxx | X.XXX | X.XXX | 0.xxx | XX.XXX | 0.xxx | XX.XXX |
| Placebo | 4 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | | | |
| HORIZANT | 8 | xx.xx | 0.xxx | 0.xxx | 0.xxx | X.XXX | X.XXX | 0.xxx | XX.XXX | 0.xxx | XX.XXX |
| Placebo | 8 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | | | |
| HORIZANT | 12 | xx.xx | 0.xxx | 0.xxx | 0.xxx | X.XXX | X.XXX | 0.xxx | XX.XXX | 0.xxx | XX.XXX |
| Placebo | 12 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | | | |
| HORIZANT | 16 | xx.xx | 0.xxx | 0.xxx | 0.xxx | X.XXX | X.XXX | 0.xxx | XX.XXX | 0.xxx | XX.XXX |
| Placebo | 16 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | | | |
| HORIZANT | 20 | xx.xx | 0.xxx | 0.xxx | 0.xxx | X.XXX | X.XXX | 0.xxx | XX.XXX | 0.xxx | XX.XXX |
| Placebo | 20 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | | | |
| HORIZANT | 24 | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | X.XXX | 0.xxx | XX.XXX | 0.xxx | XX.XXX |
| Placebo | 24 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | | | |

| | | | | 95% | 95% CI | | 95% CI | | | Untransformed | | Transformed |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Arm | Week | Estimate | SE | Lower CI | Upper CI | Difference | SE | p-value | Cohen's d | p-value | Cohen's d | |
| HORIZANT | 27 | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | x.xxx | 0.xxx | XX.XXX | 0.xxx | XX.XXX | |
| Placebo | 27 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | | | | |
| HORIZANT | Overall | xx.xx | 0.xxx | 0.xxx | 0.xxx | X.XXX | x.xxx | 0.xxx | XX.XXX | 0.xxx | XX.XXX | |
| Placebo | Overall | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | | | | |

Table 129: POMS Total Mood Disturbance Score (mITT) -- Untransformed, Each Evaluation During Maintenance Period, No Imputation

| | | | H | ORIZANT | | | Placebo | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Week | N | Mean | SD | Median | Min | Max | N | Mean | SD | Median | Min | Max |
| 4 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 8 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 12 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 16 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 20 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 24 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 26 | XX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |

Table 130: POMS Tension-Anxiety Score (mITT) -- Full Model, Mixed Effects, Transformed, Entire Maintenance Period, No Imputation

Table 131: POMS Tension-Anxiety Score (mITT) -- Untransformed, Each Evaluation During Maintenance Period, No Imputation

Table 132: POMS Anger-Hostility Score (mITT) -- Full Model, Mixed Effects, Transformed, Entire Maintenance Period, No Imputation

**Table 133:** POMS Anger-Hostility Score (mITT) -- Untransformed, Each Evaluation During Maintenance Period, No **Imputation** POMS Vigor-Activity Score (mITT) -- Full Model, Mixed Effects, Transformed, Entire Maintenance Period, No **Table 134: Imputation** POMS Vigor-Activity Score (mITT) -- Untransformed, Each Evaluation During Maintenance Period, No **Table 135: Imputation** POMS Fatigue-Inertia Score (mITT) -- Full Model, Mixed Effects, Transformed, Entire Maintenance Period, **Table 136:** No Imputation **Table 137:** POMS Fatigue-Inertia Score (mITT) -- Untransformed, Each Evaluation During Maintenance Period, No **Imputation** POMS Confusion-Bewilderment Score (mITT) -- Full Model, Mixed Effects, Transformed, Entire Maintenance **Table 138:** Period, No Imputation **Table 139:** POMS Confusion-Bewilderment Score (mITT) -- Untransformed, Each Evaluation During Maintenance Period, No Imputation POMS Depression-Dejection Score (mITT) -- Full Model, Mixed Effects, Transformed, Entire Maintenance **Table 140:** Period, No Imputation

# Table 141: POMS Depression-Dejection Score (mITT) -- Untransformed, Each Evaluation During Maintenance Period, No Imputation

Table 142: Frequency of Subjects with Suicidal Ideation Any Time During the Study – mITT Subjects

| Number of Subjects R | Number of Subjects Reporting Suicidal Ideation by C-SSRS (%) | |
|---|---|---|
| Placebo | Placebo HORIZANT p-value | |
| (N=xx) | (N=xx) | - |
| xx (xx.x%) | xx (xx.x%) | 0.xxx |
| xx (xx.x%) | xx (xx.x%) | |

**Table 143:** Summary of Concomitant Medication Use – mITT Subjects

| | Number o | f Subjects (%) |
|------------------------|------------|----------------|
| | Placebo | HORIZANT |
| <b>Medication Name</b> | (N=xx) | (N=xx) |
| Medication Name #1 | xx (xx.x%) | xx (xx.x%) |
| Medication Name #2 | xx (xx.x%) | xx (xx.x%) |

# 12.1.6. Exploratory Analyses

## 12.1.6.1. No Heavy Drinking Days by Week, Month and Grace Periods

Table 144: Percentage of Subjects No Heavy Drinking Days (mITT) – Weeks 22-25, with Imputation<sup>a</sup>

| | Placebo<br>(N=xx) | HORIZANT (N=xx) | Total<br>(N=xxx) |
|-------------------|-------------------|-----------------|------------------|
| No Heavy Drinking | | | |
| Days | | | |
| Yes | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| No | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |

<sup>&</sup>lt;sup>a</sup>Missing day imputed as a heavy drinking day

Table 145: Percentage of Subjects No Heavy Drinking Days Weeks 22-25 – No Imputation (mITT)

| | Placebo<br>(N=xx) | HORIZANT (N=xx) | Total<br>(N=xxx) |
|-------------------|-------------------|-----------------|------------------|
| No Heavy Drinking | | | |
| Days | | | |
| Yes | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| No | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |

Table 146: Percentage of Subjects with No Heavy Drinking Days Weeks 22-25 – Full Model No Imputation Logistic Regression (mITT)

| | | | | | | | | | 95% | 6 CI |
|---|---|---|---|---|---|---|---|---|---|---|
| Parameter | | DF | Estimate | Standard<br>Error | Wald Chi-<br>Square | Pr > Chi-<br>Square | Cohen's<br>h | OR | Upper CI | Lower CI |
| Intercept | | 1 | XX.XXX | XX.XXX | XX.XXX | 0.xxx | | | | |
| Treatment | Horizant | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | 0.xxx | XX.XXX | XX.XXX | XX.XXX |

| | | | | | | | | | 95% | ∕₀ CI |
|---|---|---|---|---|---|---|---|---|---|---|
| Parameter | | DF | Estimate | Standard<br>Error | Wald Chi-<br>Square | Pr > Chi-<br>Square | Cohen's<br>h | OR | Upper CI | Lower CI |
| Site | Overall | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | | | | |
| Site | 1 | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | | XX.XXX | XX.XXX | XX.XXX |
| Site | 210 | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | | XX.XXX | XX.XXX | XX.XXX |
| Cov | | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | | xx.xxx | XX.XXX | XX.XXX |

Table 147: Percentage of Subjects No Heavy Drinking Days Weekly with Imputation<sup>a</sup> (mITT)

| | Placebo<br>(N=xx) | HORIZANT (N=xx) | Total<br>(N=xxx) |
|---|---|---|---|
| WK 2 Heavy Drinking Days | | | _ |
| Yes | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| No | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Repeat for all weeks | | | |

Repeated for weeks 3-25

<sup>&</sup>lt;sup>a</sup>Missing day imputed as a heavy drinking day

Table 148: Summary of Percentage of Subjects No Heavy Drinking Days (mITT) – Full Model, Weekly, with Imputation<sup>a</sup>

| | | | | | | | | | | 959 | % CI |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Model Week <sup>b</sup> | Parameter | | DF Estimate | | Standard<br>Error | Wald<br>Chi-<br>Square | Pr > Chi-<br>Square | Cohen's<br>h | OR | Upper<br>CI | Lower<br>CI |
| 2 | Treatment | Horizant | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | 0.xxx | XX.XXX | XX.XXX | XX.XXX |
| 3 | Treatment | Horizant | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | 0.xxx | XX.XXX | XX.XXX | XX.XXX |
| 4 25 | Treatment | Horizant | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | 0.xxx | xx.xxx | XX.XXX | XX.XXX |

<sup>&</sup>lt;sup>a</sup>Missing day is imputed as a heavy drinking day. <sup>b</sup> Separate models are created for each week only the treatment arm results are presented in the summary table. All models have the same factors, only the week is different

#### Adjusted Prevalence Estimates<sup>1</sup>

| | | | | 95% | 6 CI | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Arm | Week | Estimate | SE | Lower CI | Upper CI | Difference | SE | p-value | Cohen's h |
| HORIZANT | 2 | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | X,XXX | 0.xxx | XX.XXX |
| Placebo | 2 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 3 | xx.xx | 0.xxx | 0.xxx | 0.xxx | X.XXX | x.xxx | 0.xxx | XX.XXX |
| Placebo | 3 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 4 | xx.xx | 0.xxx | 0.xxx | 0.xxx | X.XXX | x.xxx | 0.xxx | XX.XXX |
| Placebo | 4 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 5 | xx.xx | 0.xxx | 0.xxx | 0.xxx | X.XXX | x.xxx | 0.xxx | XX.XXX |
| Placebo | 5 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 6 | xx.xx | 0.xxx | 0.xxx | 0.xxx | X.XXX | x.xxx | 0.xxx | XX.XXX |
| Placebo | 6 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 7 | xx.xx | 0.xxx | 0.xxx | 0.xxx | X.XXX | x.xxx | 0.xxx | XX.XXX |
| Placebo | 7 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 8 | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | X.XXX | 0.xxx | XX.XXX |
| Placebo | 8 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |

| | | | | 95% | 6 CI | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Arm | Week | Estimate | SE | Lower CI | Upper CI | -<br>Difference | SE | p-value | Cohen's h |
| HORIZANT | 9 | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | X.XXX | 0.xxx | XX.XXX |
| Placebo | 9 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 10 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | XX.XXX |
| Placebo | 10 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 11 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | XX.XXX |
| Placebo | 11 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 12 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | XX.XXX |
| Placebo | 12 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 13 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | XX.XXX |
| Placebo | 13 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 14 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | XX.XXX |
| Placebo | 14 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 15 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | XX.XXX |
| Placebo | 15 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 16 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | XX.XXX |
| Placebo | 16 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 17 | xx.xx | 0.xxx | 0.xxx | 0.xxx | X.XXX | x.xxx | 0.xxx | XX.XXX |
| Placebo | 17 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 18 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | XX.XXX |
| Placebo | 18 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 19 | xx.xx | 0.xxx | 0.xxx | 0.xxx | X.XXX | x.xxx | 0.xxx | XX.XXX |
| Placebo | 19 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 20 | XX.XX | 0.xxx | 0.xxx | 0.xxx | x.xxx | X.XXX | 0.xxx | XX.XXX |
| Placebo | 20 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 21 | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | X.XXX | 0.xxx | XX.XXX |
| Placebo | 21 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |

| | | | | 95% | 6 CI | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Arm | Week | Estimate | SE | Lower CI | Upper CI | Difference | SE | p-value | Cohen's h |
| HORIZANT | 22 | xx.xx | 0.xxx | 0.xxx | 0.xxx | X.XXX | x.xxx | 0.xxx | XX.XXX |
| Placebo | 22 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 23 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | XX.XXX |
| Placebo | 23 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 24 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | XX.XXX |
| Placebo | 24 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 25 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | XX.XXX |
| Placebo | 25 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |

<sup>&</sup>lt;sup>1</sup>The adjusted prevalence rates are obtained from the weekly logistic regression models.

Table 149: Percentage of Subjects No Heavy Drinking Days Weekly No Imputation (mITT)

| | Placebo<br>(N=xx) | HORIZANT (N=xx) | Total<br>(N=xxx) |
|---|---|---|---|
| WK 2 Heavy Drinking Days | | | |
| Yes | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| No | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Repeat for all weeks | | - | |

Repeated for weeks 3-25

Table 150: Summary of Percentage of Subjects No Heavy Drinking Days (mITT) – Full Model, Weekly, No Imputation Same as Table 137 without imputation

Table 151: Percentage of Subjects No Heavy Drinking Days Monthly with Imputation<sup>a</sup> (mITT)

| | Placebo<br>(N=xx) | HORIZANT (N=xx) | Total<br>(N=xxx) |
|---|---|---|---|
| Mo 1 Heavy Drinking Days | | | |
| Yes | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| No | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Mo 2 Heavy Drinking Days | | | |
| Yes | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| No | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Repeat for all months | | | |

Repeated for months 3-6

Table 152: Summary of Percentage of Subjects No Heavy Drinking Days (mITT) – Full Model, Monthly, with Imputation<sup>a</sup>

| | | | | | | | | | | 95% CI | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Model Month <sup>b</sup> | Parameter | | DF | Estimate | Standard<br>Error | Wald<br>Chi-<br>Square | Pr > Chi-<br>Square | Cohen's<br>h | OR | Upper<br>CI | Lower<br>CI |
| 1 | Treatment | Horizant | Х | XX.XXX | XX.XXX | XX.XXX | 0.xxx | 0.xxx | XX.XXX | XX.XXX | XX.XXX |
| 2 | Treatment | Horizant | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | 0.xxx | XX.XXX | XX.XXX | XX.XXX |
| 3 | Treatment | Horizant | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | 0.xxx | XX.XXX | XX.XXX | XX.XXX |
| 4 | Treatment | Horizant | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | 0.xxx | XX.XXX | XX.XXX | XX.XXX |
| 5 | Treatment | Horizant | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | 0.xxx | XX.XXX | XX.XXX | XX.XXX |
| 6 | Treatment | Horizant | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | 0.xxx | xx.xxx | XX.XXX | XX.XXX |

<sup>&</sup>lt;sup>a</sup>Missing day imputed as a heavy drinking day; <sup>b</sup> Separate models are created for each month; only the treatment arm results are presented in the summary table. All models have the same factors; only the month is different.

<sup>&</sup>lt;sup>a</sup>Missing day imputed as a heavy drinking day

# Adjusted Prevalence Estimates<sup>1</sup>

| | | | | 95% | 6 CI | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Arm | Month | Estimate | SE | Lower CI | Upper CI | Difference | SE | p-value | Cohen's h |
| HORIZANT | 1 | xx.xx | 0.xxx | 0.xxx | 0.xxx | X.XXX | x.xxx | 0.xxx | XX.XXX |
| Placebo | 1 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 2 | xx.xx | 0.xxx | 0.xxx | 0.xxx | X.XXX | x.xxx | 0.xxx | XX.XXX |
| Placebo | 2 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 3 | xx.xx | 0.xxx | 0.xxx | 0.xxx | X.XXX | x.xxx | 0.xxx | XX.XXX |
| Placebo | 3 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 4 | xx.xx | 0.xxx | 0.xxx | 0.xxx | X.XXX | x.xxx | 0.xxx | XX.XXX |
| Placebo | 4 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 5 | xx.xx | 0.xxx | 0.xxx | 0.xxx | X.XXX | x.xxx | 0.xxx | XX.XXX |
| Placebo | 5 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 6 | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | x.xxx | 0.xxx | XX.XXX |
| Placebo | 6 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | |

<sup>&</sup>lt;sup>1</sup>The adjusted prevalence rates are obtained from the monthly logistic regression models

**Table 153:** Percentage of Subjects No Heavy Drinking Days Monthly No Imputation (mITT)

| | Placebo<br>(N=xx) | HORIZANT (N=xx) | Total<br>(N=xxx) |
|---|---|---|---|
| Mo 1 Heavy Drinking Days | | | |
| Yes | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) |
| No | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Mo 2 Heavy Drinking Days | | | |
| Yes | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) |
| No | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Repeat for all months | | | |

Table 154: Summary of Percentage of Subjects No Heavy Drinking Days (mITT) – Full Model, Monthly, No Imputation Same as table 141 no imputation.

Table 155: Percentage of Subjects No Heavy Drinking Days - Weeks 18-25 with Imputation<sup>a</sup> (last 8 weeks) (mITT)

| | Placebo<br>(N=xx) | HORIZANT (N=xx) | Total<br>(N=xxx) |
|---------------------|-------------------|-----------------|------------------|
| Heavy Drinking Days | | | |
| Yes | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| No | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

<sup>&</sup>lt;sup>a</sup>Missing day imputed as a heavy drinking day

Table 156: Subjects with No Heavy Drinking Days (mITT) – Logistic Regression, Weeks 18-25 (last 8 weeks), with Imputation<sup>a</sup>

| | | | | | | | | | 95% CI | |
|---|---|---|---|---|---|---|---|---|---|---|
| Parameter | | DF | Estimate | Standard<br>Error | Wald Chi-<br>Square | Pr > Chi-<br>Square | Cohen's<br>h | OR | Upper CI | Lower CI |
| Intercept | | 1 | XX.XXX | XX.XXX | XX.XXX | 0.xxx | | | | |
| Treatment | Horizant | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | 0.xxx | XX.XXX | XX.XXX | XX.XXX |
| Site | Overall | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | | | | |
| Site | 1 | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | | XX.XXX | XX.XXX | XX.XXX |
| Site | 210 | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | | XX.XXX | XX.XXX | XX.XXX |
| Cov | | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | | xx.xxx | XX.XXX | XX.XXX |

<sup>&</sup>lt;sup>a</sup>Missing day imputed as a heavy drinking day

Table 157: Percentage of Subjects No Heavy Drinking Days - Weeks 18-25 No Imputation (last 8 weeks) (mITT) Same as Table 148 no imputation.

Table 158: Subjects with No Heavy Drinking Days (mITT) – Logistic Regression, Weeks 18-25 (last 8 weeks), No Imputation

Same as Table 149 no imputation.

Table 159: Percentage of Subjects No Heavy Drinking Days - Weeks 14-25 with Imputation<sup>a</sup> (last 12 weeks) (mITT)

Table 160: Subjects with No Heavy Drinking Days (mITT) – Logistic Regression, Weeks 14-25 (last 12 weeks), with Imputation<sup>a</sup>

Table 161: Percentage of Subjects No Heavy Drinking Days - Weeks 14-25 No Imputation (last 12 weeks) (mITT)

Table 162: Subjects with No Heavy Drinking Days (mITT) – Logistic Regression, Weeks 14-25 (last 12 weeks) , No Imputation

Table 163: Percentage of Subjects No Heavy Drinking Days - Weeks 10-25 (last 16 weeks) with Imputation<sup>a</sup> (mITT)

- Table 164: Subjects with No Heavy Drinking Days (mITT) Logistic Regression, Weeks 10-25 (last 16 weeks), with Imputation<sup>a</sup>
- Table 165: Percentage of Subjects No Heavy Drinking Days Weeks 10-25 (last 16 weeks) No Imputation (mITT)
- Table 166: Subjects with No Heavy Drinking Days (mITT) Logistic Regression, Weeks 10-25 (last 16 weeks) , No Imputation
- Table 167: Percentage of Subjects No Heavy Drinking Days Weeks 6-25 (last 20 weeks) with Imputation<sup>a</sup> (mITT)
- Table 168: Subjects with No Heavy Drinking Days (mITT) Logistic Regression, Weeks 6-25 (last 20 weeks), with Imputation<sup>a</sup>
- Table 169: Percentage of Subjects No Heavy Drinking Days Weeks 6-25 (last 20 weeks) No Imputation (mITT)
- Table 170: Subjects with No Heavy Drinking Days (mITT) Logistic Regression, Weeks 6-25 (last 20 weeks) , No Imputation
- Table 171: Percentage of Subjects No Heavy Drinking Days Weeks 2-25 (complete maintenance period) with Imputation<sup>a</sup> (mITT)
- Table 172: Subjects with No Heavy Drinking Days (mITT) Logistic Regression, Weeks 2-25 (complete maintenance period), with Imputation<sup>a</sup>
- Table 173: Percentage of Subjects No Heavy Drinking Days Weeks 2-25 (complete maintenance period) No Imputation (mITT)
- Table 174: Subjects with No Heavy Drinking Days (mITT) Logistic Regression, Weeks 2-25 (complete maintenance period), No Imputation

#### 12.1.6.2. Abstinent from Alcohol by Week, Month, and Grace Period

Table 175: Percentage of Subjects Abstinent from Alcohol Weeks 22-25 with Imputation<sup>a</sup> (mITT)

| | Placebo<br>(N=xx) | HORIZANT (N=xx) | Total<br>(N=xxx) |
|---|---|---|---|
| <b>Completely Abstinent</b> | | | |
| Yes | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| No | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |

<sup>&</sup>lt;sup>a</sup>Missing day imputed as a drinking day

Table 176: Subjects Abstinent from Alcohol (mITT) – Logistic Regression, Weeks 22-25, with Imputation<sup>a</sup>

| | | | | | | | | | 95% CI | |
|---|---|---|---|---|---|---|---|---|---|---|
| Parameter | | DF | Estimate | Standard<br>Error | Wald Chi-<br>Square | Pr > Chi-<br>Square | Cohen's<br>h | OR | Upper CI | Lower CI |
| Intercept | | 1 | XX.XXX | XX.XXX | XX.XXX | 0.xxx | | | | |
| Treatment | Horizant | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | 0.xxx | XX.XXX | XX.XXX | XX.XXX |
| Site | Overall | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | | | | |
| Site | 1 | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | | XX.XXX | XX.XXX | XX.XXX |
| Site | 210 | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | | XX.XXX | XX.XXX | XX.XXX |
| Cov | | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | | XX.XXX | XX.XXX | XX.XXX |

<sup>&</sup>lt;sup>a</sup>Missing day imputed as a drinking day

Table 177: Percentage of Subjects Abstinent from Alcohol Weekly with Imputation<sup>a</sup> (mITT)

| | Placebo | HORIZANT | Total |
|----------------------|------------|-----------|------------|
| | (N=xx) | (N=xx) | (N=xxx) |
| WK 2 Drinking Days | | | |
| Yes | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| No | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Repeat for all weeks | | | |

<sup>&</sup>lt;sup>a</sup>Missing day imputed as a drinking day

Repeated for weeks 3-25

Table 178: Summary of Subjects Abstinent from Alcohol (mITT) – Logistic Regression, Weekly, with Imputation<sup>a</sup>

| | | | | | | | | | | 959 | % CI |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Model Week <sup>b</sup> | Parameter | | DF | Estimate | Standard<br>Error | Wald<br>Chi-<br>Square | Pr > Chi-<br>Square | Cohen's<br>h | OR | Upper<br>CI | Lower<br>CI |
| 2 | Treatment | Horizant | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | 0.xxx | XX.XXX | XX.XXX | XX.XXX |
| 3 | Treatment | Horizant | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | 0.xxx | xx.xxx | XX.XXX | XX.XXX |
| 4 25 | Treatment | Horizant | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | 0.xxx | xx.xxx | XX.XXX | XX.XXX |

<sup>&</sup>lt;sup>a</sup>Missing day imputed as a drinking day, <sup>b</sup> Separate models are created for each week; only the treatment arm results are presented in the summary table. All models have the same factors; only the week is different.

#### **Adjusted Abstinence Estimates**<sup>1</sup>

| | | | | 95% | 6 CI | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Arm | Week | Estimate | SE | Lower CI | Upper CI | Difference | SE | p-value | Cohen's h |
| HORIZANT | 2 | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | X,XXX | 0.xxx | XX.XXX |
| Placebo | 2 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 3 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | XX.XXX |
| Placebo | 3 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 4 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | XX.XXX |
| Placebo | 4 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 5 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | XX.XXX |
| Placebo | 5 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 6 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | XX.XXX |
| Placebo | 6 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 7 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | XX.XXX |
| Placebo | 7 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 8 | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | X.XXX | 0.xxx | XX.XXX |
| Placebo | 8 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | |

| | | | | 95% | 6 CI | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Arm | Week | Estimate | SE | Lower CI | Upper CI | -<br>Difference | SE | p-value | Cohen's h |
| HORIZANT | 9 | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | X.XXX | 0.xxx | XX.XXX |
| Placebo | 9 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 10 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | XX.XXX |
| Placebo | 10 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 11 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | XX.XXX |
| Placebo | 11 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 12 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | XX.XXX |
| Placebo | 12 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 13 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | XX.XXX |
| Placebo | 13 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 14 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | XX.XXX |
| Placebo | 14 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 15 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | XX.XXX |
| Placebo | 15 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 16 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | XX.XXX |
| Placebo | 16 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 17 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | XX.XXX |
| Placebo | 17 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 18 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | XX.XXX |
| Placebo | 18 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 19 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | XX.XXX |
| Placebo | 19 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 20 | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | X.XXX | 0.xxx | XX.XXX |
| Placebo | 20 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 21 | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | X.XXX | 0.xxx | XX.XXX |
| Placebo | 21 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | |

| | | | | 95% | 6 CI | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Arm | Week | Estimate | SE | Lower CI | Upper CI | Difference | SE | p-value | Cohen's h |
| HORIZANT | 22 | xx.xx | 0.xxx | 0.xxx | 0.xxx | X.XXX | x.xxx | 0.xxx | XX.XXX |
| Placebo | 22 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 23 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | XX.XXX |
| Placebo | 23 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 24 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | XX.XXX |
| Placebo | 24 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 25 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | XX.XXX |
| Placebo | 25 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |

<sup>&</sup>lt;sup>1</sup>The adjusted prevalence rates are obtained from the weekly logistic regression models.

**Table 179:** Percentage of Subjects Abstinent from Alcohol Weekly No Imputation (mITT)

Table 180: Summary of Subjects Abstinent from Alcohol (mITT) – Logistic Regression, Weekly, No Imputation

**Table 181:** Percentage of Subjects Abstinent Monthly with Imputation<sup>a</sup> (mITT)

| | Placebo<br>(N=xx) | HORIZANT (N=xx) | Total<br>(N=xxx) |
|---|---|---|---|
| Mo 1 Drinking Days | | | |
| Yes | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| No | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Mo 2 Drinking Days | | | |
| Yes | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) |
| No | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Repeat for all months | | | |

Repeated for months 3-6

<sup>&</sup>lt;sup>a</sup>Missing day imputed as a drinking day.
Table 182: Summary of Subjects Abstinent from Alcohol (mITT) – Logistic Regression, Monthly, With Imputation<sup>a</sup>

**Table 183:** Percentage of Subjects Abstinent from Alcohol Monthly No Imputation (mITT)

Table 184: Summary of Subjects Abstinent from Alcohol (mITT) – Logistic Regression, Weekly, No Imputation

Table 185: Percentage of Subjects Abstinent from Alcohol - Weeks 18-25 with Imputation<sup>a</sup> (last 8 weeks) (mITT)

| | Placebo<br>(N=xx) | HORIZANT (N=xx) | Total<br>(N=xxx) |
|---------------|-------------------|-----------------|------------------|
| Drinking Days | | | |
| Yes | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| No | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

<sup>&</sup>lt;sup>a</sup>Missing day imputed as a drinking day.

Table 186: Subjects Abstinent from Alcohol (mITT) – Logistic Regression, Weeks 18-25 (last 8 weeks), with Imputation<sup>a</sup>

| | | | | | | | | 95% CI | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Parameter | | DF | Estimate | Standard<br>Error | Wald Chi-<br>Square | Pr > Chi-<br>Square | Cohen's<br>h | OR | Upper CI | Lower CI |
| Intercept | | 1 | XX.XXX | XX.XXX | XX.XXX | 0.xxx | | | | |
| Treatment | Horizant | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | 0.xxx | XX.XXX | XX.XXX | XX.XXX |
| Site | Overall | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | | | | |
| Site | 1 | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | | XX.XXX | XX.XXX | XX.XXX |
| Site | 210 | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | | XX.XXX | XX.XXX | XX.XXX |
| Cov | | X | XX.XXX | XX.XXX | xx.xxx | 0.xxx | | XX.XXX | XX.XXX | XX.XXX |

<sup>&</sup>lt;sup>a</sup>Missing imputed as a drinking day.

- Table 187: Percentage of Subjects Abstinent from Alcohol Weeks 18-25 No Imputation (last 8 weeks) (mITT)
- Table 188: Subjects Abstinent from Alcohol (mITT) Logistic Regression, Weeks 18-25 (last 8 weeks), No Imputation
- Table 189: Percentage of Subjects Abstinent from Alcohol Weeks 14-25 with Imputation<sup>a</sup> (last 12 weeks) (mITT)
- Table 190: Subjects Abstinent from Alcohol (mITT) Logistic Regression, Weeks 14-25 (last 12 weeks), with Imputation<sup>a</sup>
- Table 191: Percentage of Subjects Abstinent from Alcohol Weeks 14-25 No Imputation (last 12 weeks) (mITT)
- Table 192: Subjects Abstinent from Alcohol (mITT) Logistic Regression, Weeks 14-25 (last 12 weeks), No Imputation
- Table 193: Percentage of Subjects Abstinent from Alcohol Weeks 10-25 (last 16 weeks) with Imputation<sup>a</sup> (mITT)
- Table 194: Subjects Abstinent from Alcohol (mITT) Logistic Regression, Weeks 10-25 (last 16 weeks), with Imputation<sup>a</sup>
- Table 195: Percentage of Subjects Abstinent from Alcohol- Weeks 10-25 (last 16 weeks) No Imputation (mITT)
- Table 196: Subjects Abstinent from Alcohol (mITT) Logistic Regression, Weeks 10-25 (last 16 weeks), No Imputation<sup>a</sup>
- Table 197: Percentage of Subjects Abstinent from Alcohol Weeks 6-25 (last 20 weeks) with Imputation<sup>a</sup> (mITT)
- Table 198: Subjects Abstinent from Alcohol (mITT) Logistic Regression, Weeks 6-25 (last 20 weeks), with Imputation<sup>a</sup>
- Table 199: Percentage of Subjects Abstinent from Alcohol Weeks 6-25 (last 20 weeks) No Imputation (mITT)
- Table 200: Subjects Abstinent from Alcohol (mITT) Logistic Regression, Weeks 6-25 (last 20 weeks), No Imputation
- Table 201: Percentage of Subjects Abstinent from Alcohol Weeks 2-25 (complete maintenance period) with Imputation<sup>a</sup> (mITT)
- Table 202: Subjects Abstinent from Alcohol (mITT) Logistic Regression, Weeks 2-25 (complete maintenance period), with Imputation<sup>a</sup>
- Table 203: Percentage of Subjects Abstinent from Alcohol Weeks 2-25 (complete maintenance period) No Imputation (mITT)
- Table 204: Subjects Abstinent from Alcohol (mITT) Logistic Regression, Weeks 2-25 (complete maintenance period), No Imputation

### 12.1.6.3. WHO Drinking Grade Shifts by Week, Month, and Grace Period

**Table 205:** WHO Shift Baseline to Weeks 22-25, With Imputation<sup>a</sup> (mITT)

| | Week 22-25 Category <sup>b</sup> | | | | |
|---|---|---|---|---|---|
| Baseline | Abstinent | Low Risk | Medium Risk | High Risk | Very High Risk |
| Category | N (%) | n (%) | n (%) | n (%) | n (%) |
| High Risk | | | | | |
| Very High Risk | | | | | |

<sup>&</sup>lt;sup>a</sup> Multiple imputation for missing weeks

Same table for Horizant only subjects

Same table for Placebo only subjects

Table 206: WHO 1-Level Decrease in Alcohol Consumption Weeks 22-25 With Imputation<sup>a</sup> (mITT)

| | Placebo<br>(N=xx) | HORIZANT (N=xx) | Total<br>(N=xxx) |
|---|---|---|---|
| WHO 1-Level Decrease | | | |
| Yes | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| No | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) |

<sup>&</sup>lt;sup>a</sup> Multiple imputation for missing weeks

Table 207: WHO 1-Level Decrease in Alcohol Consumption (mITT) – Logistic Regression, Weeks 22-25, With Imputation<sup>a</sup>

| | | | | | | | | | 95% | 6 CI |
|---|---|---|---|---|---|---|---|---|---|---|
| Parameter | | DF | Estimate | Standard<br>Error | Wald Chi-<br>Square | Pr > Chi-<br>Square | Cohen's<br>h | OR | Upper CI | Lower CI |
| Intercept | | 1 | XX.XXX | XX.XXX | XX.XXX | 0.xxx | | | | _ |
| Treatment | Horizant | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | 0.xxx | XX.XXX | XX.XXX | XX.XXX |

<sup>&</sup>lt;sup>b</sup> Percent is based upon row denominator (eg # subjects with High Risk at baseline)

| | | | | | | | | | 95% | ∕₀ CI |
|---|---|---|---|---|---|---|---|---|---|---|
| Parameter | | DF | Estimate | Standard<br>Error | Wald Chi-<br>Square | Pr > Chi-<br>Square | Cohen's<br>h | OR | Upper CI | Lower CI |
| Site | Overall | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | | | | |
| Site | 1 | X | XX.XXX | xx.xxx | XX.XXX | 0.xxx | | XX.XXX | XX.XXX | XX.XXX |
| Site | 210 | X | XX.XXX | xx.xxx | XX.XXX | 0.xxx | | XX.XXX | XX.XXX | XX.XXX |
| Cov | | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | | xx.xxx | XX.XXX | XX.XXX |

<sup>&</sup>lt;sup>a</sup> Multiple imputation for missing weeks

Table 208: WHO 2-Level Decrease in Alcohol Consumption Weeks 22-25 With Imputation<sup>a</sup> (mITT)

| | Placebo<br>(N=xx) | HORIZANT (N=xx) | Total<br>(N=xxx) |
|---|---|---|---|
| WHO 2-Level Decrease | | | |
| Yes | xx (xx.x%) | xx(xx.x%) | xx (xx.x%) |
| No | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

<sup>&</sup>lt;sup>a</sup> Multiple imputation for missing weeks

Table 209: WHO 2-Level Decrease in Alcohol Consumption (mITT) – Logistic Regression, Weeks 22-25, With Imputation<sup>a</sup>

| | | | | | | | | | 95% | 6 CI |
|---|---|---|---|---|---|---|---|---|---|---|
| Parameter | | DF | Estimate | Standard<br>Error | Wald Chi-<br>Square | Pr > Chi-<br>Square | Cohen's<br>h | OR | Upper CI | Lower CI |
| Intercept | | 1 | XX.XXX | XX.XXX | XX.XXX | 0.xxx | | | | |
| Treatment | Horizant | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | 0.xxx | XX.XXX | XX.XXX | XX.XXX |
| Site | Overall | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | | | | |
| Site | 1 | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | | XX.XXX | XX.XXX | XX.XXX |
| Site | 210 | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | | XX.XXX | XX.XXX | XX.XXX |

| | | | | | | | | 95% CI | |
|---|---|---|---|---|---|---|---|---|---|
| Parameter | DF | Estimate | Standard<br>Error | Wald Chi-<br>Square | Pr > Chi-<br>Square | Cohen's<br>h | OR | Upper CI | Lower CI |
| Cov | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | | XX.XXX | XX.XXX | XX.XXX |

<sup>&</sup>lt;sup>a</sup> Multiple imputation for missing weeks

Table 210: WHO Shift Baseline to Weekly Time Period, with Imputation<sup>a</sup> (mITT)

| Baseline | Week 2 Category <sup>b</sup> | | | | |
|---|---|---|---|---|---|
| Category | Abstinent n (%) | Low Risk<br>n (%) | Medium Risk<br>n (%) | High Risk<br>n (%) | Very High Risk<br>n (%) |
| High Risk | | | | | |
| Very High Risk | | | | | |

Repeat for each week

Same table for Horizant only subjects

Same table for Placebo only subjects

Table 211: Percentage of Subjects WHO 1-Level Decrease in Alcohol Consumption Weekly with Imputation<sup>a</sup> (mITT)

| | Placebo<br>(N=xx) | HORIZANT (N=xx) | Total<br>(N=xxx) |
|---|---|---|---|
| WK 2 WHO 1-Level | | | |
| Decrease | | | |
| Yes | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) |
| No | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| Repeat for all weeks | · | · | |

<sup>&</sup>lt;sup>a</sup> Multiple imputation model used to impute missing weeks.

<sup>&</sup>lt;sup>b</sup> Percent is based upon row denominator (eg # subjects with High Risk at baseline)

<sup>a</sup>Multiple imputation model used to impute missing weeks.

Table 212: Summary of WHO 1-Level Decrease in Alcohol Consumption (mITT) – Logistic Regression, Weekly, with Imputation<sup>a</sup>

| | | | | | | | | | | 95% CI | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Model Week <sup>b</sup> | Parameter | | DF | Estimate | Standard<br>Error | Wald<br>Chi-<br>Square | Pr > Chi-<br>Square | Cohen's<br>h | OR | Upper<br>CI | Lower<br>CI |
| 2 | Treatment | Horizant | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | 0.xxx | XX.XXX | XX.XXX | XX.XXX |
| 3 | Treatment | Horizant | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | 0.xxx | XX.XXX | XX.XXX | XX.XXX |
| 4 25 | Treatment | Horizant | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | 0.xxx | XX.XXX | XX.XXX | XX.XXX |

<sup>&</sup>lt;sup>a</sup>Missing day imputed as a drinking day, <sup>b</sup> Separate models are created for each week; only the treatment arm results are presented in the summary table. All models have the same factors; only the week is different.

### **Adjusted Prevalence Estimates**<sup>1</sup>

| | | | | 95% CI | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Arm | Week | Estimate | SE | Lower CI | Upper CI | Difference | SE | p-value | Cohen's h |
| HORIZANT | 2 | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | X,XXX | 0.xxx | XX.XXX |
| Placebo | 2 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 3 | xx.xx | 0.xxx | 0.xxx | 0.xxx | X.XXX | x.xxx | 0.xxx | XX.XXX |
| Placebo | 3 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 4 | xx.xx | 0.xxx | 0.xxx | 0.xxx | X.XXX | X.XXX | 0.xxx | XX.XXX |
| Placebo | 4 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 5 | xx.xx | 0.xxx | 0.xxx | 0.xxx | X.XXX | X.XXX | 0.xxx | XX.XXX |
| Placebo | 5 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 6 | xx.xx | 0.xxx | 0.xxx | 0.xxx | X.XXX | X.XXX | 0.xxx | XX.XXX |
| Placebo | 6 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 7 | xx.xx | 0.xxx | 0.xxx | 0.xxx | X.XXX | x.xxx | 0.xxx | XX.XXX |

| | | | | 95% | 6 CI | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Arm | Week | Estimate | SE | Lower CI | Upper CI | -<br>Difference | SE | p-value | Cohen's h |
| Placebo | 7 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 8 | xx.xx | 0.xxx | 0.xxx | 0.xxx | X.XXX | X.XXX | 0.xxx | XX.XXX |
| Placebo | 8 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 9 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | X.XXX | 0.xxx | XX.XXX |
| Placebo | 9 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 10 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | X.XXX | 0.xxx | XX.XXX |
| Placebo | 10 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 11 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | X.XXX | 0.xxx | XX.XXX |
| Placebo | 11 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 12 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | XX.XXX |
| Placebo | 12 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 13 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | XX.XXX |
| Placebo | 13 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 14 | xx.xx | 0.xxx | 0.xxx | 0.xxx | X.XXX | X.XXX | 0.xxx | XX.XXX |
| Placebo | 14 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 15 | xx.xx | 0.xxx | 0.xxx | 0.xxx | X.XXX | X.XXX | 0.xxx | XX.XXX |
| Placebo | 15 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 16 | xx.xx | 0.xxx | 0.xxx | 0.xxx | X.XXX | x.xxx | 0.xxx | XX.XXX |
| Placebo | 16 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 17 | xx.xx | 0.xxx | 0.xxx | 0.xxx | X.XXX | x.xxx | 0.xxx | XX.XXX |
| Placebo | 17 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 18 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | XX.XXX |
| Placebo | 18 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 19 | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | X.XXX | 0.xxx | XX.XXX |
| Placebo | 19 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 20 | xx.xx | 0.xxx | 0.xxx | 0.xxx | X.XXX | X.XXX | 0.xxx | XX.XXX |

| | | | | 95% | 6 CI | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Arm | Week | Estimate | SE | Lower CI | Upper CI | Difference | SE | p-value | Cohen's h |
| Placebo | 20 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 21 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | XX.XXX |
| Placebo | 21 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 22 | xx.xx | 0.xxx | 0.xxx | 0.xxx | X.XXX | x.xxx | 0.xxx | XX.XXX |
| Placebo | 22 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 23 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | XX.XXX |
| Placebo | 23 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 24 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | XX.XXX |
| Placebo | 24 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 25 | XX.XX | 0.xxx | 0.xxx | 0.xxx | x.xxx | X.XXX | 0.xxx | XX.XXX |
| Placebo | 25 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | |

<sup>&</sup>lt;sup>1</sup>Prevalence estimates are obtained from the weekly logistic regression models.

Table 213: Percentage of Subjects WHO 2-Level Decrease in Alcohol Consumption Weekly with Imputation<sup>a</sup> (mITT)

| | Placebo<br>(N=xx) | HORIZANT (N=xx) | Total<br>(N=xxx) |
|---|---|---|---|
| WK 2 WHO 2-Level | | | |
| Decrease | | | |
| Yes | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| No | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| Repeat for all weeks | ` , | , , | , , |

<sup>&</sup>lt;sup>a</sup>Multiple imputation model used to impute missing weeks.

Table 214: Summary of WHO 2-Level Decrease in Alcohol Consumption (mITT) – Logistic Regression, Weekly, with Imputation<sup>a</sup>

| | | | | | | | | | | 959 | % CI |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Model Week <sup>b</sup> | Parameter | | DF | Estimate | Standard<br>Error | Wald<br>Chi-<br>Square | Pr > Chi-<br>Square | Cohen's<br>h | OR | Upper<br>CI | Lower<br>CI |
| 2 | Treatment | Horizant | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | 0.xxx | xx.xxx | XX.XXX | XX.XXX |
| 3 | Treatment | Horizant | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | 0.xxx | xx.xxx | XX.XXX | XX.XXX |
| 4 25 | Treatment | Horizant | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | 0.xxx | xx.xxx | XX.XXX | XX.XXX |

<sup>&</sup>lt;sup>a</sup>Missing day imputed as a drinking day, <sup>b</sup> Separate models are created for each week; only the treatment arm results are presented in the summary table. All models have the same factors; only the week is different.

#### **Adjusted Prevalence Estimates**<sup>1</sup>

| | 95% CI | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Arm | Week | Estimate | SE | Lower CI | Upper CI | Difference | SE | p-value | Cohen's h |
| HORIZANT | 2 | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | X.XXX | 0.xxx | XX.XXX |

| | | | | 95% | 6 CI | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Arm | Week | Estimate | SE | Lower CI | Upper CI | Difference | SE | p-value | Cohen's h |
| Placebo | 2 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 3 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | XX.XXX |
| Placebo | 3 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 4 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | XX.XXX |
| Placebo | 4 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 5 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | XX.XXX |
| Placebo | 5 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 6 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | XX.XXX |
| Placebo | 6 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 7 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | XX.XXX |
| Placebo | 7 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 8 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | XX.XXX |
| Placebo | 8 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 9 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | XX.XXX |
| Placebo | 9 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 10 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | XX.XXX |
| Placebo | 10 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 11 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | XX.XXX |
| Placebo | 11 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 12 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | XX.XXX |
| Placebo | 12 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 13 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | XX.XXX |
| Placebo | 13 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 14 | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | X.XXX | 0.xxx | XX.XXX |
| Placebo | 14 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 15 | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | x.xxx | 0.xxx | XX.XXX |

| | | | | 95% | 6 CI | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Arm | Week | Estimate | SE | Lower CI | Upper CI | Difference | SE | p-value | Cohen's h |
| Placebo | 15 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 16 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | XX.XXX |
| Placebo | 16 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 17 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | XX.XXX |
| Placebo | 17 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 18 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | X.XXX | 0.xxx | XX.XXX |
| Placebo | 18 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 19 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | X.XXX | 0.xxx | XX.XXX |
| Placebo | 19 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 20 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | X.XXX | 0.xxx | XX.XXX |
| Placebo | 20 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 21 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | XX.XXX |
| Placebo | 21 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 22 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | X.XXX | 0.xxx | XX.XXX |
| Placebo | 22 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 23 | xx.xx | 0.xxx | 0.xxx | 0.xxx | X.XXX | x.xxx | 0.xxx | XX.XXX |
| Placebo | 23 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 24 | XX.XX | 0.xxx | 0.xxx | 0.xxx | x.xxx | X.XXX | 0.xxx | XX.XXX |
| Placebo | 24 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | |
| HORIZANT | 25 | XX.XX | 0.xxx | 0.xxx | 0.xxx | x.xxx | X.XXX | 0.xxx | XX.XXX |
| Placebo | 25 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |

<sup>&</sup>lt;sup>1</sup>Prevalence estimates are obtained from the weekly logistic regression models.

- Table 215: WHO Shift Baseline to Weekly Time Period, No Imputation<sup>a</sup> (mITT)
- Table 216: Percentage of Subjects WHO 1-Level Decrease in Alcohol Consumption Weekly No Imputation (mITT)
- Table 217: Summary of WHO 1-Level Decrease in Alcohol Consumption (mITT) Logistic Regression, Weekly, No Imputation
- Table 218: Percentage of Subjects WHO 2-Level Decrease in Alcohol Consumption Weekly No Imputation (mITT)
- Table 219: Summary of WHO 2-Level Decrease in Alcohol Consumption (mITT) Logistic Regression, Weekly, No Imputation
- Table 220: WHO Shift Baseline to Monthly Time Period, with Imputation<sup>a</sup> (mITT)
- Table 221: Percentage of Subjects WHO 1-Level Decrease in Alcohol Consumption Monthly with Imputation (mITT)
- Table 222: Summary of WHO 1-Level Decrease in Alcohol Consumption (mITT) Logistic Regression, Monthly, with Imputation<sup>a</sup>
- Table 223: Percentage of Subjects WHO 2-Level Decrease in Alcohol Consumption Monthly with Imputation<sup>a</sup> (mITT)
- Table 224: Summary of WHO 2-Level Decrease in Alcohol Consumption (mITT) Logistic Regression, Monthly, with Imputation<sup>a</sup>
- Table 225: WHO Shift Baseline to Monthly Time Period, No Imputation<sup>a</sup> (mITT)
- Table 226: Percentage of Subjects WHO 1-Level Decrease in Alcohol Consumption Monthly No Imputation (mITT)
- Table 227: Summary of WHO 1-Level Decrease in Alcohol Consumption (mITT) Logistic Regression, Monthly, No Imputation
- Table 228: Percentage of Subjects WHO 2-Level Decrease in Alcohol Consumption Monthly No Imputation (mITT)
- Table 229: Summary of WHO 2-Level Decrease in Alcohol Consumption (mITT) Logistic Regression, Monthly, No Imputation
- Table 230: WHO Shift Baseline to Weeks 18-25 (last 8 weeks), with Imputation<sup>a</sup> (mITT)
- Table 231: Percentage of Subjects WHO 1-Level Decrease in Alcohol Consumption Weeks 18-25 with Imputation<sup>a</sup> (last 8 weeks) (mITT)
- Table 232: Subjects with WHO 1-Level Decrease in Alcohol Consumption (mITT) Logistic Regression, Weeks 18-25 (last 8 weeks), with Imputation<sup>a</sup>

- Table 233: Percentage of Subjects WHO 2-Level Decrease in Alcohol Consumption Weeks 18-25 with Imputation<sup>a</sup> (last 8 weeks) (mITT)
- Table 234: Subjects with WHO 2-Level Decrease in Alcohol Consumption (mITT) Logistic Regression, Weeks 18-25 (last 8 weeks), with Imputation<sup>a</sup>
- Table 235: WHO Shift Baseline to Weeks 18-25 (last 8 weeks), No Imputation<sup>a</sup> (mITT)
- Table 236: Percentage of Subjects WHO 1-Level Decrease in Alcohol Consumption Weeks 18-25 No Imputation (last 8 weeks) (mITT)
- Table 237: Subjects with WHO 1-Level Decrease in Alcohol Consumption (mITT) Logistic Regression, Weeks 18-25 (last 8 weeks), No Imputation
- Table 238: Percentage of Subjects WHO 2-Level Decrease in Alcohol Consumption Weeks 18-25 No Imputation (last 8 weeks) (mITT)
- Table 239: Subjects with WHO 2-Level Decrease in Alcohol Consumption (mITT) Logistic Regression, Weeks 18-25 (last 8 weeks), No Imputation
- Table 240: WHO Shift Baseline to Weeks 14-25 (last 12 weeks), with Imputation<sup>a</sup> (mITT)
- Table 241: Percentage of Subjects WHO 1-Level Decrease in Alcohol Consumption Weeks 14-25 with Imputation<sup>a</sup> (last 12 weeks) (mITT)
- Table 242: Subjects with WHO 1-Level Decrease in Alcohol Consumption (mITT) Logistic Regression, Weeks 14-25 (last 12 weeks), with Imputation<sup>a</sup>
- Table 243: Percentage of Subjects WHO 2-Level Decrease in Alcohol Consumption Weeks 14-25 with Imputation<sup>a</sup> (last 12 weeks) (mITT)
- Table 244: Subjects with WHO 2-Level Decrease in Alcohol Consumption (mITT) Logistic Regression, Weeks 14-25 (last 12 weeks), with Imputation<sup>a</sup>
- Table 245: WHO Shift Baseline to Weeks 14-25 (last 12 weeks), No Imputation<sup>a</sup> (mITT)
- Table 246: Percentage of Subjects WHO 1-Level Decrease in Alcohol Consumption Weeks 14-25 No Imputation (last 12 weeks) (mITT)
- Table 247: Subjects with WHO 1-Level Decrease in Alcohol Consumption (mITT) Logistic Regression, Weeks 14-25 (last 12 weeks), No Imputation

- Table 248: Percentage of Subjects WHO 2-Level Decrease in Alcohol Consumption Weeks 14-25 No Imputation (last 12 weeks) (mITT)
- Table 249: Subjects with WHO 2-Level Decrease in Alcohol Consumption (mITT) Logistic Regression, Weeks 14-25 (last 12 weeks), No Imputation
- Table 250: WHO Shift Baseline to Weeks 10-25 (last 16 weeks), with Imputation<sup>a</sup> (mITT)
- Table 251: Percentage of Subjects WHO 1-Level Decrease in Alcohol Consumption Weeks 10-25 (last 16 weeks) with Imputation<sup>a</sup> (mITT)
- Table 252: Subjects with WHO 1-Level Decrease in Alcohol Consumption (mITT) Logistic Regression, Weeks 10-25 (last 16 weeks), with Imputation<sup>a</sup>
- Table 253: Percentage of Subjects WHO 2-Level Decrease in Alcohol Consumption Weeks 10-25 (last 16 weeks) with Imputation<sup>a</sup> (mITT)
- Table 254: Subjects with WHO 2-Level Decrease in Alcohol Consumption (mITT) Logistic Regression, Weeks 10-25 (last 16 weeks), with Imputation<sup>a</sup>
- Table 255: WHO Shift Baseline to Weeks 10-25 (last 16 weeks), No Imputation<sup>a</sup> (mITT)
- Table 256: Percentage of Subjects WHO 1-Level Decrease in Alcohol Consumption Weeks 10-25 (last 16 weeks) No Imputation (mITT)
- Table 257: Subjects with WHO 1-Level Decrease in Alcohol Consumption (mITT) Logistic Regression, Weeks 10-25 (last 16 weeks), No Imputation
- Table 258: Percentage of Subjects WHO 2-Level Decrease in Alcohol Consumption Weeks 10-25 (last 16 weeks) No Imputation (mITT)
- Table 259: Subjects with WHO 2-Level Decrease in Alcohol Consumption (mITT) Logistic Regression, Weeks 10-25 (last 16 weeks), No Imputation
- Table 260: WHO Shift Baseline to Weeks 6-25 (last 20 weeks), with Imputation<sup>a</sup> (mITT)
- Table 261: Percentage of Subjects WHO 1-Level Decrease in Alcohol Consumption Weeks 6-25 (last 20 weeks) with Imputation<sup>a</sup> (mITT)
- Table 262: Subjects with WHO 1-Level Decrease in Alcohol Consumption (mITT) Logistic Regression, Weeks 6-25 (last 20 weeks), with Imputation<sup>a</sup>

- Table 263: Percentage of Subjects WHO 2-Level Decrease in Alcohol Consumption Weeks 6-25 (last 20 weeks) with Imputation<sup>a</sup> (mITT)
- Table 264: Subjects with WHO 2-Level Decrease in Alcohol Consumption (mITT) Logistic Regression, Weeks 6-25 (last 20 weeks), with Imputation<sup>a</sup>
- Table 265: WHO Shift Baseline to Weeks 6-25 (last 20 weeks), No Imputation<sup>a</sup> (mITT)
- Table 266: Percentage of Subjects WHO 1-Level Decrease in Alcohol Consumption Weeks 6-25 (last 20 weeks) No Imputation (mITT)
- Table 267: Subjects with WHO 1-Level Decrease in Alcohol Consumption (mITT) Logistic Regression, Weeks 6-25 (last 20 weeks), No Imputation
- Table 268: Percentage of Subjects WHO 2-Level Decrease in Alcohol Consumption Weeks 6-25 (last 20 weeks) No Imputation (mITT)
- Table 269: Subjects with WHO 2-Level Decrease in Alcohol Consumption (mITT) Logistic Regression, Weeks 6-25 (last 20 weeks), No Imputation
- Table 270: WHO Shift Baseline to Weeks 2-25 (complete maintenance period), with Imputation<sup>a</sup> (mITT)
- Table 271: Percentage of Subjects WHO 1-Level Decrease in Alcohol Consumption Weeks 2-25 (complete maintenance period) with Imputation<sup>a</sup> (mITT)
- Table 272: Subjects with WHO 1-Level Decrease in Alcohol Consumption (mITT) Logistic Regression, Weeks 2-25 (complete maintenance period), with Imputation<sup>a</sup>
- Table 273: Percentage of Subjects WHO 2-Level Decrease in Alcohol Consumption Weeks 2-25 (complete maintenance period) with Imputation<sup>a</sup> (mITT)
- Table 274: Subjects with WHO 2-Level Decrease in Alcohol Consumption (mITT) Logistic Regression, Weeks 2-25 (complete maintenance period), with Imputation<sup>a</sup>
- Table 275: WHO Shift Baseline to Weeks 2-25 (complete maintenance period), No Imputation<sup>a</sup> (mITT)
- Table 276: Percentage of Subjects WHO 1-Level Decrease in Alcohol Consumption Weeks 2-25 (complete maintenance period) No Imputation (mITT)
- Table 277: Subjects with WHO 1-Level Decrease in Alcohol Consumption (mITT) Logistic Regression, Weeks 2-25 (complete maintenance period), No Imputation

Table 278: Percentage of Subjects WHO 2-Level Decrease in Alcohol Consumption Weeks 2-25 (complete maintenance period) No Imputation (mITT)

Table 279: Subjects with WHO 2-Level Decrease in Alcohol Consumption (mITT) – Logistic Regression, Weeks 2-25 (complete maintenance period), No Imputation

#### 12.1.6.4. Abstinent from Cigarette Smoking

**Table 280:** Percentage of Subjects Abstinent from Cigarettes among Smokers Weeks 24 + 26 – No Imputation (mITT)

| | Placebo<br>(N=xx) | HORIZANT (N=xx) | Total<br>(N=xxx) |
|---|---|---|---|
| Completely Abstinent | | | |
| Yes | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| No | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |

Table 281: Subjects Abstinent from Cigarettes among Smokers (mITT) – Logistic Regression, Weeks 24 + 26, No Imputation

| | | | | | | | | 95% CI | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Parameter | | DF | Estimate | Standard<br>Error | Wald Chi-<br>Square | Pr > Chi-<br>Square | Cohen's<br>h | OR | Upper CI | Lower CI |
| Intercept | | 1 | XX.XXX | xx.xxx | XX.XXX | 0.xxx | | | | |
| Treatment | Horizant | X | XX.XXX | xx.xxx | XX.XXX | 0.xxx | 0.xxx | XX.XXX | XX.XXX | XX.XXX |
| Site | Overall | X | XX.XXX | xx.xxx | XX.XXX | 0.xxx | | XX.XXX | XX.XXX | XX.XXX |
| Site | 1 | X | XX.XXX | xx.xxx | XX.XXX | 0.xxx | | | | |
| Site | 210 | X | XX.XXX | xx.xxx | XX.XXX | 0.xxx | | | | |

| | | | | | | | | 95% | 6 CI |
|---|---|---|---|---|---|---|---|---|---|
| Parameter | DF | Estimate | Standard<br>Error | Wald Chi-<br>Square | Pr > Chi-<br>Square | Cohen's<br>h | OR | Upper CI | Lower CI |
| Cov | X | XX.XXX | xx.xxx | XX.XXX | 0.xxx | | XX.XXX | XX.XXX | XX.XXX |

Table 282: Percentage of Subjects Abstinent from Cigarettes among Smokers Weeks 24 + 26 – with Imputation<sup>a</sup> (mITT)

Table 283: Subjects Abstinent from Cigarettes among Smokers (mITT) – Logistic Regression, Weeks 24 + 26, No Imputation<sup>a</sup>

Table 284: Percentage of Subjects Abstinent from Cigarettes among Smokers Entire Maintenance Period – No Imputation (mITT)

Table 285: Subjects Abstinent from Cigarettes among Smokers (mITT) – Logistic Regression, Entire Maintenance Period, No Imputation

| | | | | | | | | | 95% | ∕₀ CI |
|---|---|---|---|---|---|---|---|---|---|---|
| Parameter | | DF | Estimate | Standard<br>Error | Wald Chi-<br>Square | Pr > Chi-<br>Square | Cohen's<br>h | OR | Upper CI | Lower CI |
| Intercept | | 1 | XX.XXX | XX.XXX | XX.XXX | 0.xxx | | | | |
| Treatment | Horizant | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | 0.xxx | XX.XXX | XX.XXX | XX.XXX |
| Site | Overall | X | XX.XXX | xx.xxx | xx.xxx | 0.xxx | | XX.XXX | XX.XXX | XX.XXX |
| Site | 1 | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | | | | |
| Site | 210 | X | XX.XXX | xx.xxx | xx.xxx | 0.xxx | | | | |
| Cov | | X | XX.XXX | xx.xxx | xx.xxx | 0.xxx | | XX.XXX | XX.XXX | XX.XXX |

Table 286: Percentage of Subjects Abstinent from Cigarettes among Smokers Entire Maintenance Period – with Imputation (mITT)

Table 287: Subjects Abstinent from Cigarettes among Smokers (mITT) – Logistic Regression, Entire Maintenance Period, with Imputation<sup>a</sup>

#### 12.1.6.5. Blood PEth Levels

Table 288: Blood PEth Levels (ng/mL) (mITT) – Analysis of Covariance, Transformed, Week 26, No Imputation

Type III Wald Tests

| Parameter | Num DF | Den DF | F Value | p-value |
|---------------|--------|--------|---------|---------|
| ARM | 1 | xxx | XXX.XX | 0.xxx |
| Site | 9 | xxx | XXX.XX | 0.xxx |
| Baseline PEth | 1 | xxx | XXX.XX | 0.xxx |

## **Least Squares Means**

| | | | 95% | 6 CI | | | Untran | sformed | Transformed | |
|---|---|---|---|---|---|---|---|---|---|---|
| Arm | Estimate | SE | Lower CI | Upper CI | Difference | SE | p-value | Cohen's d | p-value | Cohen's d |
| HORIZANT | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | X.XXX | 0.xxx | XX.XXX | 0.xxx | XX.XXX |
| Placebo | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | | | |

**Table 289:** Percentages of Negative Blood PEth Samples at Week 26 – No Imputation (mITT)

| | Placebo<br>(N=xx) | HORIZANT (N=xx) | Total<br>(N=xxx) |
|---|---|---|---|
| Blood PEth Test<br>Negative <sup>1</sup><br>Positive <sup>2</sup> | xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%) |

<sup>&</sup>lt;sup>1</sup>Not detectable with lower limit of quantitation (LLOQ) of 8 ng/mL.

<sup>&</sup>lt;sup>2</sup> PEth level > LLOQ.

Table 290: Samples with No Detectable Blood PEth Levels (mITT) – Logistic Regression, Week 26, No Imputation

| | | | | | | | | | 95% | 6 CI |
|---|---|---|---|---|---|---|---|---|---|---|
| Parameter | | DF | Estimate | Standard<br>Error | Wald Chi-<br>Square | Pr > Chi-<br>Square | Cohen's d | OR | Upper CI | Lower CI |
| Intercept | | 1 | XX.XXX | xx.xxx | XX.XXX | 0.xxx | | | | |
| Treatment | Horizant | X | XX.XXX | xx.xxx | XX.XXX | 0.xxx | 0.xxx | XX.XXX | XX.XXX | XX.XXX |
| Site | Overall | X | XX.XXX | xx.xxx | XX.XXX | 0.xxx | | xx.xxx | XX.XXX | XX.XXX |
| Site | 1 | X | XX.XXX | xx.xxx | XX.XXX | 0.xxx | | | | |
| Site | 210 | X | XX.XXX | xx.xxx | XX.XXX | 0.xxx | | | | |
| Cov | | X | XX.XXX | xx.xxx | XX.XXX | 0.xxx | | XX.XXX | XX.XXX | XX.XXX |

# 12.1.6.6. MINI AUD Symptoms

Table 291: MINI AUD Number of Symptoms (mITT) – Analysis of Covariance, Week 26, No Imputation

Type III Wald Tests

| Parameter | Num DF | Den DF | F Value | p-value |
|-----------|--------|--------|---------|---------|
| ARM | 1 | XXX | XXX.XX | 0.xxx |
| Site | 9 | xxx | XXX.XX | 0.xxx |
| MINI AUD | 1 | XXX | XXX.XX | 0.xxx |

### **Least Squares Means**

| | | | 95% | 6 CI | | | Untran | sformed | Transformed | |
|---|---|---|---|---|---|---|---|---|---|---|
| Arm | Estimate | SE | Lower CI | Upper CI | Difference | SE | p-value | Cohen's d | p-value | Cohen's d |
| HORIZANT | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | x.xxx | 0.xxx | XX.XXX | 0.xxx | XX.XXX |
| Placebo | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | | | |

#### 12.1.6.7 Continuous Secondary Endpoints With and Without Imputation for Last 4 Weeks and Entire Maintenance Period

Table 292: Percentage of Heavy Drinking Days per Week (mITT) – Mixed Effects, Transformed, Weeks 22-25, with Imputation<sup>a</sup>

**Type III Wald Tests** 

| Parameter | Num DF | Den DF | F Value | p-value |
|-----------|--------|--------|---------|---------|
| ARM | 1 | XXX | XXX.XX | 0.xxx |
| Week | 3 | XXX | XXX.XX | 0.xxx |
| Site | 9 | XXX | XXX.XX | 0.xxx |
| Cov | X | XXX | XXX.XX | 0.xxx |
| ARM*Week | 3 | XXX | XXX.XX | 0.xxx |

### **Least Squares Means**

| | | | | 95% | 6 CI | | | Untran | sformed | Trans | sformed |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Arm | Week | Estimate | SE | Lower CI | Upper CI | Difference | SE | p-value | Cohen's d | p-value | Cohen's d |
| HORIZANT | 22 | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | X,XXX | 0.xxx | XX.XXX | 0.xxx | XX.XXX |
| Placebo | 22 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | | | |
| HORIZANT | 23 | xx.xx | 0.xxx | 0.xxx | 0.xxx | X.XXX | x.xxx | 0.xxx | XX.XXX | 0.xxx | XX.XXX |
| Placebo | 23 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | | | |
| HORIZANT | 24 | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | x.xxx | 0.xxx | XX.XXX | 0.xxx | XX.XXX |
| Placebo | 24 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | | | |
| HORIZANT | 25 | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | x.xxx | 0.xxx | XX.XXX | 0.xxx | XX.XXX |
| Placebo | 25 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | | | |
| HORIZANT | Overall | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | X.XXX | 0.xxx | XX.XXX | 0.xxx | XX.XXX |
| Placebo | Overall | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | | | |

<sup>&</sup>lt;sup>a</sup>Missing weeks are imputed using a multiple imputation model.

Table 293: Percentage of Heavy Drinking Days per Week (mITT) -- Mixed Effects, Transformed, Weeks 2-25 No Imputation

**Type III Wald Tests** 

| Parameter | Num DF | Den DF | F Value | n voluo |
|-----------|--------|--------|---------|---------|
| rarameter | Num Dr | Den Dr | r value | p-value |
| ARM | 1 | XXX | XXX.XX | 0.xxx |
| Week | 23 | XXX | XXX.XX | 0.xxx |
| Site | 9 | XXX | XXX.XX | 0.xxx |
| Cov | X | XXX | XXX.XX | 0.xxx |
| ARM*Week | 23 | XXX | XXX.XX | 0.xxx |

### **Least Squares Means**

| | | | | 95% | 6 CI | | | Untran | sformed | Trans | sformed |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Arm | Week | Estimate | SE | Lower CI | Upper CI | Difference | SE | p-value | Cohen's d | p-value | Cohen's d |
| HORIZANT | 2 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | XX.XXX | 0.xxx | XX.XXX |
| Placebo | 2 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | | | |
| HORIZANT | 3 | xx.xx | 0.xxx | 0.xxx | 0.xxx | X.XXX | x.xxx | 0.xxx | XX.XXX | 0.xxx | XX.XXX |
| Placebo | 3 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | | | |
| HORIZANT | 4 | xx.xx | 0.xxx | 0.xxx | 0.xxx | X.XXX | x.xxx | 0.xxx | XX.XXX | 0.xxx | XX.XXX |
| Placebo | 4 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | | | |
| HORIZANT | 5 | xx.xx | 0.xxx | 0.xxx | 0.xxx | X.XXX | x.xxx | 0.xxx | XX.XXX | 0.xxx | XX.XXX |
| Placebo | 5 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | | | |
| HORIZANT | 6 | xx.xx | 0.xxx | 0.xxx | 0.xxx | X.XXX | x.xxx | 0.xxx | XX.XXX | 0.xxx | XX.XXX |
| Placebo | 6 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | | | |
| HORIZANT | 7 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | XX.XXX | 0.xxx | XX.XXX |

| | | | | 95% | % CI | | | Untrar | sformed | Trans | sformed |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Arm | Week | Estimate | SE | Lower CI | Upper CI | - Difference | SE | p-value | Cohen's d | p-value | Cohen's d |
| Placebo | 7 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | | | |
| HORIZANT | 8 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | XX.XXX | 0.xxx | xx.xxx |
| Placebo | 8 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | | | |
| HORIZANT | 9 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | XX.XXX | 0.xxx | xx.xxx |
| Placebo | 9 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | | | |
| HORIZANT | 10 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | X.XXX | 0.xxx | XX.XXX | 0.xxx | xx.xxx |
| Placebo | 10 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | | | |
| HORIZANT | 11 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | X.XXX | 0.xxx | XX.XXX | 0.xxx | xx.xxx |
| Placebo | 12 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | | | |
| HORIZANT | 13 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | X.XXX | 0.xxx | XX.XXX | 0.xxx | xx.xxx |
| Placebo | 13 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | | | |
| HORIZANT | 14 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | X.XXX | 0.xxx | XX.XXX | 0.xxx | xx.xxx |
| Placebo | 14 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | | | |
| HORIZANT | 15 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | X.XXX | 0.xxx | XX.XXX | 0.xxx | xx.xxx |
| Placebo | 15 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | | | |
| HORIZANT | 16 | xx.xx | 0.xxx | 0.xxx | 0.xxx | X.XXX | x.xxx | 0.xxx | XX.XXX | 0.xxx | xx.xxx |
| Placebo | 16 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | | | |
| HORIZANT | 17 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | X.XXX | 0.xxx | XX.XXX | 0.xxx | xx.xxx |
| Placebo | 17 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | | | |
| HORIZANT | 18 | xx.xx | 0.xxx | 0.xxx | 0.xxx | X.XXX | x.xxx | 0.xxx | XX.XXX | 0.xxx | xx.xxx |
| Placebo | 18 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | | | |
| HORIZANT | 19 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | X.XXX | 0.xxx | XX.XXX | 0.xxx | xx.xxx |
| Placebo | 19 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | | | |
| HORIZANT | 20 | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | X.XXX | 0.xxx | XX.XXX | 0.xxx | xx.xxx |
| Placebo | 20 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | | | |
| HORIZANT | 21 | XX.XX | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | XX.XXX | 0.xxx | XX.XXX |

| | | | | 95% | 6 CI | _ | | Untran | sformed | Tran | sformed |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Arm | Week | Estimate | SE | Lower CI | Upper CI | Difference | SE | p-value | Cohen's d | p-value | Cohen's d |
| Placebo | 21 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | | | |
| HORIZANT | 22 | xx.xx | 0.xxx | 0.xxx | 0.xxx | X.XXX | x.xxx | 0.xxx | XX.XXX | 0.xxx | XX.XXX |
| Placebo | 22 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | | | |
| HORIZANT | 23 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | XX.XXX | 0.xxx | XX.XXX |
| Placebo | 23 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | | | |
| HORIZANT | 24 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | XX.XXX | 0.xxx | XX.XXX |
| Placebo | 24 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | | | |
| HORIZANT | 25 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | XX.XXX | 0.xxx | XX.XXX |
| Placebo | 25 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | | | |
| HORIZANT | Overall | XX.XX | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | XX.XXX | 0.xxx | XX.XXX |
| Placebo | Overall | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | | | |

**Table 294:** Percentage of Heavy Drinking Days per Week (mITT) -- Mixed Effects, Transformed, Weeks 2-25, with

**Imputation** 

**Table 295:** Percentage of Days Abstinent per Week (mITT) – Mixed Effects, Transformed, Weeks 22-25, with Imputation

**Table 296:** Percentage of Days Abstinent per Week (mITT) – Mixed Effects, Transformed, Weeks 2-25, No Imputation

**Table 297:** Percentage of Days Abstinent per Week (mITT) – Mixed Effects, Transformed, Weeks 2-25, with Imputation

**Table 298:** Drinks per Week (mITT) – Mixed Effects, Transformed, Weeks 22-25, with Imputation

**Table 299:** Drinks per Week (mITT) – Mixed Effects, Transformed, Weeks 2-25, No Imputation

**Table 300:** Drinks per Week (mITT) – Mixed Effects, Transformed, Weeks 2-25, with Imputation

**Table 301:** Drinks per Drinking Day (mITT) – Mixed Effects, Transformed, Weeks 22-25, with Imputation

**Table 302:** Drinks per Drinking Day (mITT) – Mixed Effects, Transformed, Weeks 2-25, No Imputation

**Table 303:** Drinks per Drinking Day (mITT) – Mixed Effects, Transformed, Weeks 2-25, with Imputation

**Table 304:** ACQ-SR-R Score (mITT) – Mixed Effects, Transformed, Weeks 24 + 26, with Imputation

- Table 305: ACQ-SR-R Score (mITT) Mixed Effects, Transformed, Weeks 2-26, No Imputation
- Table 306: ACQ-SR-R Score (mITT) Mixed Effects, Transformed, Weeks 2-26, with Imputation
- Table 307: ImBIBe Score (mITT) Mixed Effects, Transformed, Weeks 24 + 26, with Imputation
- Table 308: ImBIBe Score (mITT) Mixed Effects, Transformed, Weeks 2-26, No Imputation
- Table 309: ImBIBe Score (mITT) Mixed Effects, Transformed, Weeks 2-26, with Imputation
- Table 310: Mean Cigarettes Smoked per Week among Smokers (mITT) Mixed Effects, Transformed, Weeks 24 + 26 with
  - **Imputation**
- Table 311: Mean Cigarettes Smoked per Week among Smokers (mITT) Mixed Effects, Transformed, Weeks 2-26, No
  - **Imputation**
- Table 312: Mean Cigarettes Smoked per Week among Smokers (mITT) Mixed Effects, Transformed, Weeks 2-26, with
  - **Imputation**
- Table 313: PSQI Score (mITT) Mixed Effects, Transformed, Weeks 24 + 26, with Imputation
- Table 314: PSQI Score (mITT) Mixed Effects, Transformed, Weeks 2-26, No Imputation

- Table 315: PSQI Score (mITT) Mixed Effects, Transformed, Weeks 2-26, with Imputation
- Table 316: PSQI Sleep Quality Score (mITT) Mixed Effects, Transformed, Weeks 24 + 26, with Imputation
- Table 317: PSQI Sleep Quality Score (mITT) Mixed Effects, Transformed, Weeks 2-26, No Imputation
- Table 318: PSQI Sleep Quality Score (mITT) Mixed Effects, Transformed, Weeks 2-26, with Imputation
- Table 319: PSQI Sleep Latency Score (mITT) Mixed Effects, Transformed, Weeks 24 + 26, with Imputation
- Table 320: PSQI Sleep Latency Score (mITT) Mixed Effects, Transformed, Weeks 2-26, No Imputation
- Table 321: PSQI Sleep Latency Score (mITT) Mixed Effects, Transformed, Weeks 2-26, with Imputation
- Table 322: PSQI Sleep Duration Score (mITT) Mixed Effects, Transformed, Weeks 24 + 26, with Imputation
- Table 323: PSQI Sleep Duration Score (mITT) Mixed Effects, Transformed, Weeks 2-26, No Imputation
- Table 324: PSQI Sleep Duration Score (mITT) Mixed Effects, Transformed, Weeks 2-26, with Imputation
- Table 325: PSQI Sleep Disturbance Score (mITT) Mixed Effects, Transformed, Weeks 24 + 26, with Imputation
- Table 326: PSQI Sleep Disturbance Score (mITT) Mixed Effects, Transformed, Weeks 2-26, No Imputation
- Table 327: PSQI Sleep Disturbance Score (mITT) Mixed Effects, Transformed, Weeks 2-26, with Imputation
- Table 328: PSQI Use of Sleep Medication Score (mITT) Mixed Effects, Transformed, Weeks 24 + 26, with Imputation
- Table 329: PSQI Use of Sleep Medication Score (mITT) Mixed Effects, Transformed, Weeks 2-26, No Imputation
- Table 330: PSQI Use of Sleep Medication Score (mITT) Mixed Effects, Transformed, Weeks 2-26, with Imputation
- Table 331: PSQI Daytime Dysfunction Score (mITT) Mixed Effects, Transformed, Weeks 24 + 26, with Imputation
- Table 332: PSQI Daytime Dysfunction Score (mITT) Mixed Effects, Transformed, Weeks 2-26, No Imputation
- Table 333: PSQI Daytime Dysfunction Score (mITT) Mixed Effects, Transformed, Weeks 2-26, with Imputation
- Table 334: BAI Score (mITT) Mixed Effects, Transformed, Weeks 24 + 26, with Imputation
- Table 335: BAI Score (mITT) Mixed Effects, Transformed, Weeks 2-26, No Imputation
- Table 336: BAI Score (mITT) Mixed Effects, Transformed, Weeks 2-26, with Imputation
- Table 337: BDI-II Score (mITT) Mixed Effects, Transformed, Weeks 24 + 26, with Imputation

Table 338: BDI-II Score (mITT) – Mixed Effects, Transformed, Weeks 2-26, No Imputation

Table 339: BDI-II Score (mITT) – Mixed Effects, Transformed, Weeks 2-26, with Imputation

#### 12.1.6.8 Subjects with No Heavy Drinking Days by Moderators

Table 340: Subjects with No Heavy Drinking Days by MINI Withdrawal (mITT) – Logistic Regression, Weeks 22-25, with Imputation<sup>a</sup>

| | | | | | | | | | 95% | 6 CI |
|---|---|---|---|---|---|---|---|---|---|---|
| Parameter | | DF | Estimate | Standard<br>Error | Wald Chi-<br>Square | Pr > Chi-<br>Square | Cohen's d | OR | Upper CI | Lower CI |
| Intercept | | 1 | XX.XXX | XX.XXX | XX.XXX | 0.xxx | | | | |
| Treatment | Horizant | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | 0.xxx | XX.XXX | XX.XXX | XX.XXX |
| Site | 1 | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | | | | |
| Site | 210 | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | | | | |
| Withdrawal | | 1 | XX.XXX | XX.XXX | XX.XXX | 0.xxx | 0.xxx | XX.XXX | XX.XXX | XX.XXX |
| Withdrawal x Tx | | X | XX.XXX | xx.xxx | XX.XXX | 0.xxx | | | | |

<sup>&</sup>lt;sup>a</sup>Missing day is imputed as a heavy drinking day

## **Adjusted Prevalence Estimates**

| | | | | | 95% | 6 CI | |
|---|---|---|---|---|---|---|---|
| Arm | Withdrawal | Estimate | SE | Cohen's h | Lower CI | Upper CI | p-value |
| HORIZANT | No | XX.XX | 0.xxx | 0.xxx | 0.xxx | 0.xxx | 0.xxx |
| Placebo | No | XX.XX | 0.xxx | | 0.xxx | 0.xxx | |
| HORIZANT | Yes | xx.xx | 0.xxx | 0.xxx | 0.xxx | 0.xxx | 0.xxx |
| Placebo | Yes | XX.XX | 0.xxx | | 0.xxx | 0.xxx | |

Additional models for moderators use the same shell with the moderator by treatment interaction and the adjusted prevalence table

- Table 341: Subjects with No Heavy Drinking Days by BAI (mITT) Logistic Regression, Weeks 22-25, with Imputation
- Table 342: Subjects with No Heavy Drinking Days by BAI (mITT) Logistic Regression, Weeks 22-25, with Imputation
- Table 343: Subjects with No Heavy Drinking Days by PSQI Total Score (mITT) Logistic Regression, Weeks 22-25, with Imputation
- Table 344: Subjects with No Heavy Drinking Days by Smoking Status (mITT) Logistic Regression, Weeks 22-25, with Imputation
- Table 345: Subjects with No Heavy Drinking Days by POMS Total Mood Disturbance (mITT) Logistic Regression, Weeks 22-25, with Imputation
- Table 346: Subjects with No Heavy Drinking Days by POMS Tension-Anxiety (mITT) Logistic Regression, Weeks 22-25, with Imputation
- Table 347: Subjects with No Heavy Drinking Days by POMS Depression-Dejection (mITT) Logistic Regression, Weeks 22-25, with Imputation
- Table 348: Subjects with No Heavy Drinking Days by POMS Confusion-Bewilderment (mITT) Logistic Regression, Weeks 22-25, with Imputation
- Table 349: Subjects with No Heavy Drinking Days by POMS Vigor-Anxiety (mITT) Logistic Regression, Weeks 22-25, with Imputation
- Table 350: Subjects with No Heavy Drinking Days by POMS Anger-Hostility (mITT) Logistic Regression, Weeks 22-25, with Imputation
- Table 351: Subjects with No Heavy Drinking Days by POMS Fatigue-Inertia (mITT) Logistic Regression, Weeks 22-25, with Imputation
- Table 352: Subjects with No Heavy Drinking Days by ACQ-SR-R (mITT) Logistic Regression, Weeks 22-25, with Imputation
- Table 353: Subjects with No Heavy Drinking Days by Number of Days Abstinent from Alcohol (7 Days Prior to Randomization) (mITT) Logistic Regression, Weeks 22-25, with Imputation
- Table 354: Subjects with No Heavy Drinking Days by Years Drinking Regularly (mITT) Logistic Regression, Weeks 22-25, with Imputation

Table 355: Subjects with No Heavy Drinking Days by Drinks per Week (28 Days Prior to Screening) (mITT) – Logistic Regression, Weeks 22-25, with Imputation
 Table 356: Subjects with No Heavy Drinking Days by Reducer Status (Change in Drinks per Day) (mITT) – Logistic Regression, Weeks 22-25, with Imputation
 Table 357: Subjects with No Heavy Drinking Days by Drinking Goal (mITT) – Logistic Regression, Weeks 22-25, with Imputation
 Table 358: Subjects with No Heavy Drinking Days by Total Dose (mITT) – Logistic Regression, Weeks 22-25, with Imputation
 Table 359: Subjects with No Heavy Drinking Days by BIS (mITT) – Logistic Regression, Weeks 22-25, with Imputation

# 12.2. Listings

**Listing 1. Subject Disposition - All Subjects** 

| Subject<br>ID | Date of<br>Consent | Treatment<br>Group | mITT | Eval-<br>uable | Study<br>Completion | (Day) Date of<br>Study Completion<br>or Early<br>Discontinuation | Reason for Early<br>Discontinuation | Subject<br>confined<br>or incar-<br>cerated | Start Date/ End<br>Date of incar-<br>ceration |
|---|---|---|---|---|---|---|---|---|---|
| XXX | mm/dd/yyyy | HORIZANT<br>Placebo<br>None | Yes<br>No | Yes<br>No | Yes<br>No | (xx) mm/dd/yyyy | xxxxxx | Yes<br>No | mm/dd/yyyy /<br>mm/dd/yyyy |

Note: Day is relative to Study Day 0.

Listing 2. Enrollment and Randomization – All Consented Subjects

| xxx HORIZANT mm/dd/yyyy Yes Yes mm/dd/yyyy xxx | Subject<br>ID | Treatment<br>Group | Date of<br>Consent | Did the subject meet all eligibility criteria? | Randomized? | Date of<br>Randomization | Kit<br>Number |
|---|---|---|---|---|---|---|---|
| Placebo No No | XXX | HORIZANT<br>Placebo | mm/dd/yyyy | Yes<br>No | Yes<br>No | mm/dd/yyyy | XXX |

**Listing 3. Reason not Eligible – Screen Failures** 

| Subject ID | Criterion Type | Criterion |
|------------|---------------------------------------|-----------|
| Xxx | Inclusion Criteria Exclusion Criteria | |

**Listing 4. Protocol Deviations – mITT Subjects** 

| Subject<br>ID | Treatment<br>Group | Deviation<br>Date | Protocol Deviation | Details |
|---|---|---|---|---|
| XXX | HORIZANT | mm/dd/yyyy | Subject Failed to Meet the Inclusion/Exclusion Criteria | |
| | Placebo | | Source Documentation was Not Available | |
| | | | Pregnancy Test Not Performed | |
| | | | Required study data was not obtained or obtained late | |
| | | | due to site error | |
| | | | Informed Consent Deviation | |
| | | | AE/SAE Reporting Deviation | |
| | | | Other Deviation: | XXXXXXXXXXXXX |

Note: Only subjects with protocol deviation are listed.

Listing 5. Subjects Excluded from the Efficacy Analysis or Evaluable Set

| Subject<br>ID | Treatment<br>Group | Reason for Exclusion from mITT | Reason for Exclusion from Evaluable Set |
|---|---|---|---|
| Xxx | HORIZANT<br>Placebo | XXXXXX | |

Note: Only subjects excluded from the efficacy analysis or evaluable set are listed.

**Listing 6. Demographics Data – mITT Subjects** 

| Subject<br>ID | Treatment<br>Group | Gender | Age<br>(yrs) | Ethnicity | Race | Marital Status |
|---|---|---|---|---|---|---|
| XXX | HORIZANT | Male | XX | Hispanic or Latino | American Indian or Alaska Native | Married |
| | Placebo | Female | | Not Hispanic or<br>Latino | Asian | Divorced |
| | | | | Unknown | Native Hawaiian or Other Pacific Islander | Living with Partner |
| | | | | | Black or African American | Widowed |
| | | | | | White | Separated |
| | | | | | Other | Never Married |
| | | | | | Unknown | Unknown |
| | | | | | | Missing |

**Listing 6. Demographics Data - mITT(continued)** 

| Subject<br>ID | Treatment<br>Group | Years of Education | Years of Formal Education (GED=12years) | Usual Employment Pattern in the last 30 days |
|---|---|---|---|---|
| XXX | HORIZANT<br>Placebo | XX | XXX | Full-time, 35+ hrs/week Part-time, regular hours Part-time, irregular hours/daywork Student Military service Unemployed Retired/Disabled Homemaker In controlled environment Unknown |

Listing 7. Baseline Drinking Characteristics – mITT Subjects

| Subject<br>ID | Treatment<br>Group | Drinks/Day<br>(Days -1 to -28) | Drinks/Day<br>(Days -1 to -14<br>Pre-<br>randomization) | Drinks/<br>Drinking Day<br>(Days -1 to -28) | Drinks/Drinking<br>Day (Days -1 to -<br>14 Pre-<br>randomization) | Weekly % Heavy Drinking Days (Days -1 to -28) | Weekly % Heavy Drinking Days (Days -1 to -14 Pre- randomization) |
|---|---|---|---|---|---|---|---|
| XXX | HORIZANT<br>Placebo | XXX.X | XXX.X | XXXX | XXX.X | | |

Note: Exclude the three abstinent days during pre-randomization period.

**Listing 7. Baseline Drinking Characteristics mITT (continued)** 

| Subject<br>ID | Treatment<br>Group | Weekly %Very<br>Heavy Drinking<br>Days<br>(Days -1 to -28) | Weekly % Very<br>Heavy Drinking<br>Days<br>(Days -1 to -14<br>Pre-<br>randomization) | Weekly % Days<br>Abstinent (Days<br>-1 to -28) | Weekly % Days<br>Abstinent (Days -<br>1 to -14 Pre-<br>randomization) |
|---|---|---|---|---|---|
| XXX | HORIZANT<br>Placebo | XXX.X | XXX.X | XXX.X | XXX.X |

Note: Exclude the three abstinent days during pre-randomization period.
**Listing 8. Baseline Smoking Characteristics – mITT Subjects** 

| Subject<br>ID | Treatment<br>Group | How often<br>do you<br>smoke? | How soon after<br>you wake up do<br>you smoke your<br>first cigarette? | Difficult to refrain from smoking? | Which cigarette do you hate to give up the most? | How many<br>cigarettes<br>per day? | Smoke more frequently during 1st hours of waking? | Do you smoke if you are ill and in bed? | Score |
|---|---|---|---|---|---|---|---|---|---|
| XXX | HORIZANT | Occasionally | Within 5 min | No | First morning | 10 or less | No | No | XX |
| | Placebo | Daily | Within 6-30 min | Yes | All others | 11-20 | Yes | Yes | |
| | | Not at all | Within 31-60 min | | | 21-30 | | | |
| | | | After 60 min | | | 31 or more | | | |

**Listing 9. Family Members with History of Alcohol Problems** 

| Subject ID | Treatment<br>Group | Relative 1 with<br>Problem | Relative 2 with Problem |
|---|---|---|---|
| XXX | HORIZANT | Father | Father |
| | Placebo | Mother | Mother |
| | | Brother | Brother |
| | | Sister | Sister |
| | | Child | Child |

Note: only list those family members with problems

**Listing 10. MINI DSM5 Disorders – mITT Subjects** 

| Subject<br>ID | Treatment<br>Group | Visit Date | Diagnosis | Timeframe |
|---|---|---|---|---|
| XXX | HORIZANT<br>Placebo | mm/dd/yyyy | xxxxxx | Current (2 weeks ) Past Recurrent |

Note: Only subjects with a diagnosis of a disorder will be listed.

Listing 11. MINI DSM5 AUD – mITT Subjects

| Subject<br>ID | Treatment<br>Group | Visit Date | # of Symptoms |
|---------------|---------------------|------------|---------------|
| XXX | HORIZANT<br>Placebo | mm/dd/yyyy | XX |

**Listing 12. Medical History – mITT Subjects** 

| 9 | Treatment<br>Group | SOC | Specify | Start Date | Ongoing |
|---|---|---|---|---|---|
| | HORIZANT<br>Placebo | Blood and Lymphatic System Cardiovascular Endocrinologic/Metabolic Gastrointestinal HEENT Hepatobiliary Hematologic/Oncologic Immune System Infectious Disease Musculoskeletal Nervous system Psychiatric Renal/Urinary Reproductive System Respiratory Skin Other:xxxxxxxxx | XXXXXXXXXX | mm/dd/yyyy | No<br>Yes |

Programming note: Only identify items that were scored "yes"

**Listing 13. Drinking Treatment History mITT** 

| Subject<br>ID No. | Treatment<br>Group | Age first<br>started<br>drinking<br>alcohol<br>regularly | Number of lifetime inpatient visits to get help with reducing or quitting drinking | Number of<br>lifetime inpatient<br>hospitalizations<br>for illnesses,<br>injuries, or<br>accidents due to<br>drinking | Number of times<br>in lifetime<br>underwent<br>alcohol<br>detoxification<br>using medication | Number of lifetime outpatient visits with a health professional to get help with reducing or quitting drinking | Number of group<br>meetings<br>attended for<br>alcohol problems<br>or drinking in<br>the past year |
|---|---|---|---|---|---|---|---|
| XXX | HORIZANT<br>Placebo | XXX | xxx | xxx | xxx | xxx | xxx |

## **Listing 14. Drinking Goal – mITT Subjects**

| Subject<br>ID | Treatment<br>Group | Visit Date | What GOAL have you chosen for yourself about drinking at this time? | How motivated are you to reach this goal | How confident you are that you will be able to reach this goal |
|---|---|---|---|---|---|
| XXX | HORIZANT | mm/dd/yyyy | Controlled use of alcohol | 1 = Not motivated | 1 = Not confident |
| | Placebo | | Temporary abstinence from drinking | 2, 3, 4, 5, 6, 7, 8, 9, | 2, 3, 4, 5, 6, 7, 8, 9, |
| | | | Occasional drinking when urges strongly felt | 10= Extremely motivated | 10= Extremely confident |
| | | | Total abstinence, but realize a slip is | 10- Extremely motivated | 10– Extremely confident |
| | | | possible | | |
| | | | Total abstinence-never drink again | | |
| | | | No goal | - | |

**Listing 15. Surgical History – mITT Subjects** 

| Subject<br>ID No. | Treatment<br>Group | Has the subject had any past surgeries? | Date of Surgery | Type of Surgery |
|---|---|---|---|---|
| XXX | HORIZANT<br>Placebo | Yes<br>No | mm/dd/yyyy | xxxxxxxxxxx |

**Listing 16. Physical Exam – mITT Subjects** 

| Subject ID No. | Treatment<br>Group | Exam Date | Body System | Specify | Any abnormal finding during the physical exam? | Describe clinically significant findings |
|---|---|---|---|---|---|---|
| XXX | HORIZANT<br>Placebo | mm/dd/yyyy | Oral Cavity HEENT Heart Lungs Abdomen Spleen Liver Extremities Skin Neurological Psychiatric General Appearance Other:xxxxxxxx | XXXXXXXXX | Yes<br>No | XXXXXXX |

Programming Note: Only report the items that are abnormal

Listing 17. Daily and Weekly Standard Drink Units (TLFB) During Treatment

| Subject<br>ID | Treatment<br>Group | Week | D1 | D2 | D3 | D4 | D5 | D6 | <b>D7</b> | Mean<br>drinks/day | Mean drinks/<br>drinking day | Heavy<br>drinking days | % days<br>abstinent |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| XXX | HORIZANT | 1 | XX | XX | XX | XX | XX | XX | XX | | | | |
| | Placebo | 2 | | | | | | | | | | | |
| | | 3, etc | | | | | | | | | | | |

## **Listing 18. Drinking Question – mITT Subjects**

| Subject<br>ID | Treatment<br>Group | Date of<br>Assessment | Did the subject have any drinking days since the last visit? | Did the subject have any heavy drinking days since the last visit? | Date of last visit |
|---|---|---|---|---|---|
| XXX | HORIZANT | mm/dd/yyyy | Yes | Yes | mm/dd/yyyy |
| | Placebo | | No | No | |

## Listing 19. Drinking Consequences, Craving, Impulsiveness, Anxiety and Depression Scores

| Subject<br>ID | Treatment<br>Group | Week | ImBIBe | ACQ-SR-R | BAI | BDI-II | BIS |
|---|---|---|---|---|---|---|---|
| XXX | HORIZANT<br>Placebo | | XXX | XXX | XXX | XXX | |

Listing 20. Pittsburg Sleep Quality Index Scores

| Subject<br>ID | Treatment<br>Group | Week | Subjective sleep quality | Sleep<br>latency | Sleep<br>duration | Habitual sleep<br>disturbances | Use of sleep<br>medication | Day time<br>dysfunction | Total<br>score |
|---|---|---|---|---|---|---|---|---|---|
| XXX | HORIZANT<br>Placebo | | XX | XX | XX | XX | XX | XX | XX |

## **Listing 21. Smoking Data-mITT Subjects**

| Subject<br>ID | Treatment<br>Group | Week | Visit Date | Over the past week, how many days did you smoke cigarettes? | On the days you smoked, how many cigarettes did you smoke on average? | Used any other tobacco or nicotine products during the past week? |
|---|---|---|---|---|---|---|
| XXX | HORIZANT<br>Placebo | 2, 3, 5, 7, 9, 13 | mm/dd/yyyy | X | XX | No<br>Yes |

## Listing 22. PEth Levels – mITT Subjects

| Subject<br>ID | Treatment<br>Group | Date collected | Week | PEth (ng/mL) | Last Date SDU <sup>a</sup> >0 reported prior to blood draw | Days since last<br>report of SDU<br>>0 prior to<br>blood draw |
|---|---|---|---|---|---|---|
| XXXX | HORIZANT | mm/dd/yyyy | | | | |
| | Placebo | | | | | |

<sup>&</sup>lt;sup>a</sup>SDU is the standard drink unit obtained from the Timeline Follow Back

Listing 23. MINI AUD End of Study – mITT Subjects

| Subject<br>ID | Treatment<br>Group | | | | | | Item | | | | | | # of Symptoms |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | - | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | |
| XXX | HORIZANT | Y | Y | Y | Y | Y | Y | Y | Y | Y | Y | Y | |
| | Placebo | N | N | N | N | N | N | N | N | N | N | N | |
| | | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | |
| tem# | List of Items | | | | | | | | | | | | |
| 1 | a. During the | times whe | n you dra | nk alcol | nol, did | you end | l up drir | king m | ore than | you plan | ned when | you star | ted? |
| 2 | | b. Did you repeatedly want to reduce or control your alcohol use? Did you try to cut down or control your alcohol use, but failed? IF YES TO EITHER, MARK YES. | | | | | | | | | | | |
| 3 | c. On the days alcohol? | c. On the days that you drank, did you spend substantial time obtaining alcohol, drinking, or recovering from the effects of alcohol? | | | | | | | m the effects of | | | | |
| 4 | d. Did you cra | ive or have | e a strong | desire o | r urge t | to use al | lcohol? | | | | | | |
| 5 | e. Did you spe | end less tir | ne meetin | g your i | espons | ibilities | at work | at scho | ool, or at | home, be | ecause of | your rep | eated drinking? |
| 6 | f. If your drin | | | | - | | | | | | | | Č |
| 7 | g. Were you i | ntoxicated | more tha | n once i | n any s | ituation | | | | | | | ample, driving a ca |
| 8 | h. Did you co:<br>problems? | riding a motorbike, using machinery, boating, etc.? h. Did you continue to use alcohol, even though it was clear that the alcohol had caused or worsened psychological or physical problems? i. Did you reduce or give up important work, social or recreational activities because of your drinking? j. Did you need to drink a lot more in order to get the same effect that you got when you first started drinking or did you get much less effect with continued use of the same amount? | | | | | | | | | | | |
| ) | i. Did you red | | | | | | | | | | | | |
| 10 | j. Did you nee | | | | | | | | | | | | |
| 11 | hand tremor o | r "the shal | kes"; trou | ble slee | oing; na | usea or | vomitin | g; heari | ng or se | eing thin | gs other p | eople coi | ating or heart rate;<br>uld not see or hear<br>ese, check yes for |

K2. Did you drink alcohol to reduce or avoid withdrawal symptoms or to avoid being hung over? If K1 or K2 = yes, then score

this question), OR

as yes.

**Listing 24. Exit Interview – mITT Subjects** 

| Subject<br>ID | Treatment<br>Group | Visit Date | What study drug do you believe you were taking? | Why do you think you received that drug? | Do you feel the study drug helped you to reduced drinking? | How would you describe your experience taking the study drug? |
|---|---|---|---|---|---|---|
| | | | | | | Experienced no unwanted side effects and benefited from |
| XXX | HORIZANT | mm/dd/yyyy | Placebo | Had side effects | Very Much | taking the medication |
| | | | | | | Experienced some unwanted side effects but benefited from |
| | Placebo | | Active medication | Had no side effects | Much | taking the medication |
| | | | | | | Experienced a lot unwanted |
| | | | Both placebo and | | | side effects but benefited from |
| | | | active | Staff told me | Moderately | taking the medication |
| | | | | Staff treatment me | | Experienced no unwanted side effects but did not benefit |
| | | | Don't know | different | A Little | from taking the medication |
| | | | 2011 ( 11110 11 | different | 11 21000 | Experienced some unwanted |
| | | | | No improvement in | | side effects and did not benefit |
| | | | Other substance | drinking | Not Little | from taking the medication |
| | | | | TT- 4 in a manage in | | Experienced a lot of unwanted |
| | | | | Had improvement in drinking | Not at all | side effects and did not benefit from taking the medication |
| | | | | Had a hunch | Not at all | from taking the medication |
| | | | | I just felt different | | |
| | | | | Other: xxxxx | - | |

**Listing 24. Exit Interview – mITT Subjects (Continued)** 

| Treatment<br>Group | Visit Date | If a friend were in need of help<br>for a drinking problem, would<br>you recommend taking the study<br>drug to him/her? | If you were to need treatment in the future, would you choose to take the study drug again? | How much do you think of yourself as wanting to please other people (people pleaser)? |
|---|---|---|---|---|
| HORIZANT<br>Placebo | mm/dd/yyyy | Yes, definitely Yes, generally | Definitely yes Probably yes | More than average Average |
| | | Neither yes nor no | Maybe | Less than average |
| | | No, not really | Probably not | |
| | | No, definitely not | Definitely not | |
| | Group | Group Visit Date HORIZANT mm/dd/yyyy | Treatment Group Visit Date for a drinking problem, would you recommend taking the study drug to him/her? HORIZANT Placebo mm/dd/yyyy Yes, definitely Yes, generally Neither yes nor no No, not really | Treatment Group Visit Date for a drinking problem, would you recommend taking the study drug to him/her? Yes, definitely Placebo Yes, generally Neither yes nor no No, not really for a drinking problem, would treatment in the future, would you choose to take the study drug again? Definitely yes Probably yes Maybe Probably not |

**Listing 25. Other Services Use – mITT Subjects** 

| Subject<br>ID | Group | Date | Week | Since your last visit<br>did you attend any<br>AA, 12-step, SOS, or<br>similar group<br>meeting? | How<br>many? | Have you visited another health professional to get help reducing drinking? | What type of professional? |
|---|---|---|---|---|---|---|---|
| XXX | HORIZANT | mm/dd/yyyy | XX | Yes | XXXX | Yes | xxxxx |
| | Placebo | | | No | | No | |

Listing 26. Blood for DNA and RNA Testing – mITT Subjects

| Subject<br>ID | Treatment<br>Group | Was blood drawn for DNA testing? | Date of blood<br>draw for DNA<br>testing? | Was blood drawn for RNA testing? | Date of blood<br>draw for RNA<br>testing: | Did the subject agree to optional genetics testing for a broader range of research? |
|---|---|---|---|---|---|---|
| XXXX | HORIZANT | Yes | mm/dd/yyyy | Yes | mm/dd/yyyy | Yes |
| | Placebo | No | | No | | No |

**Listing 27. Drug Exposure – mITT Subjects** 

| Subject | Treatment | Study | Date Start of | Date End of | # Capsules | # Capsules | Reason for Discontinuation |
|---|---|---|---|---|---|---|---|
| ID No. | Group | Week | Week | Week | Prescribed | Taken | |
| XXX | HORIZANT<br>Placebo | 1, 2, 3, 4,<br>5, 6, 7, 8,<br>9, 10, 11,<br>12, 13, 14,<br>15, 16, 17,<br>18, 19, 20,<br>21, 22, 23<br>24, 25, 26 | mm/dd/yyyy | mm/dd/yyyy | xx | XX | |

Listing 28. Adverse Events - mITT Subjects

| Subject<br>ID | Treatment<br>Group | Adverse Event (Verbatim) S: SOC P: PT Term | Start Date/<br>Day | Stop Date/<br>Day | Duration<br>in Days | Severity | Relation-<br>ship | Actions<br>Taken | Outcome | Serious |
|---|---|---|---|---|---|---|---|---|---|---|
| | HORIZAN | | mm/dd/yyy | | | | | | | |
| XXX | T | Verbatim | y | mm/dd/yyyy | | 1 | 1 | 1 | 1 | Yes |
| | Placebo | S: xxxx | XX | XX | | 2 | 2 | 2 | 2 | No |
| | | P: xxxx | | | | 3 | 3 | 3 | 3 | |
| | | | | | | 4 | 4 | 4 | 4 | |
| | | | | | | | 5 | 5 | 5 | |
| | | | | | | | | 6 | | |

Notes: Day is relative to Study Day 0.

Severity: 1=Mild; 2=Moderate; 3=Severe; 4=Potentially Life-threatening.

Relationship: 1= Unrelated; 2=Unlikely; 3=Possibly; 4=Probably; 5=Definitely

Action Taken Due to AE: 1=None; 2=Treated with Drugs; 3=Non-drug treatment; 4=ER/Outpatient visit; 5=Hospitalization; 6=Referral for treatment

Outcome: 1=Resolved; 2=Recovered with sequelae; 3=Ongoing; 4=Required treatment; 5=Unknown

Programmer's Note: If "Were any AEs reported?" checkbox=No, then display "None Reported" in the Adverse Event column and SOC/PT column. If an AE started and stopped the same day, the duration is 1 day.

**Listing 29. Serious Adverse Events - mITT Subjects** 

CAF

| Subject<br>ID | Treatment<br>Group | Verbatim S: SOC P: PT | Start Date/<br>Day | Stop Date/<br>Day | SAE Category | Severity | Relationship |
|---|---|---|---|---|---|---|---|
| XXX | HORIZANT | Verbatim | mm/dd/yyyy | mm/dd/yyyy | Death | 1 | 1 |
| | Placebo | S: XXX | Xx | Xx | Life-threatening | 2 | 2 |
| | | P: XX | | | Hospitalization | 3 | 3 |
| | | | | | Disability | 4 | 4 |
| | | | | | Congenital Anomaly/Birth | | |
| | | | | | Defect | 5 | 5 |
| | | | | | Required Intervention to Prevent | | |
| | | | | | Permanent Impairment / Damage | | |
| | | | | | Other | | |

**Listing 29. Serious Adverse Events - mITT Subjects (continued)** 

| Subject<br>ID No. | SAE | Continued<br>Study<br>Participation | Study Drug<br>Start Date | Date of last<br>administration<br>of study drug<br>prior to SAE | SAE Abated after study drug stopped? | Continued<br>study drug<br>Administration | SAE<br>reappeared<br>after<br>rechallenge? | Outcome |
|---|---|---|---|---|---|---|---|---|
| XXX | Verbatim | Yes | mm/dd/yyyy | mm/dd/yyyy | Yes | Yes | Yes | 1 |
| | | No | | | No | No | No | 2 |
| | | | | | n/a | | n/a | 3 |

Notes: Day is relative to Study Day 0.

Severity: 1=Mild; 2=Moderate; 3=Severe; 4=Potentially Life-threatening.

Relationship: 1= Unrelated; 2=Unlikely; 3=Possibly; 4=Probably; 5=Definitely

Outcome: 1=Recovered/Resolved; 2=Recovering/Resolving; 3=Not Recovered/Not Resolved; 4=Recovered/Resolved With Sequelae; 5=Fatal (Date of Death)

**Listing 30. POMS Scores** 

| | | | Scores | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Subject<br>ID | Treatment<br>Group | Week | Total Mood<br>Disturbance | Tension | Depression | Anger | Fatigue | Confusion | Vigor |
| XXX | HORIZANT<br>Placebo | | XXX | xxx | XXX | XXX | XXX | XXX | XXX |

Listing 31. Columbia-Suicide Severity Scale – mITT Subjects

| | | | | Response<br>to<br>Question: | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subjec<br>t ID | Treatment<br>Group | Visit Date | Study<br>Week | Q1 | Q2 | Q3 | Q4 | Q5 | Q6 | <b>Q</b> 7 | Q8 | Q9 | Q10 | Q11 | Q12 | Q13 |
| XXX | HORIZANT | mm/dd/yyyy | -1, 2, 4 | Yes | Yes | Yes | Yes | Yes | Yes | Type 1 | 1 | 1 | 0 | 0 | 0 | Yes |
| | Placebo | | 6, 8, 10, | No | No | No | No | No | No | Type 2 | 2 | 2 | 1 | 1 | 1 | No |
| | | | 12, 14, 16 | | | | | | | Type 3 | 3 | 3 | 2 | 2 | 2 | |
| | | | 18, 20, 22 | | | | | | | Type 4 | 4 | 4 | 3 | 3 | 3 | |
| | | | 24, 26 | | | | | | | Type 5 | 5 | 5 | 4 | 4 | 4 | |
| | | | | | | | | | | • • | | | 5 | 5 | 5 | |

#### **Suicide Ideation**

- 1. Have you wished you were dead or wished you could go to sleep and not wake up?
- 2. Have you actually had any thoughts of killing yourself?
- 3. Have you been thinking about how you might do this?
- 4. Have you had these thoughts and had some intention of acting on them?
- 5. Have you started to work out or worked out the details of how to kill yourself?
- 6. Do you intend to carry out this plan?

### **Intensity of Ideation**

- 7. The following features should be rated with respect to the most severe type of ideation (i.e. 1-5 with 1 being the least severe and 5 being the most severe)
- 8. How many times have you had these thoughts?1=Less than once a week; 2=Once a week; 3=2-5 times a week; 4=Daily or almost; 5=Many times each day
- 9. When you have the thoughts, how long do they last? 1=Fleeting-few seconds or minutes; 2=Less than 1 hr-some of the time; 3=1-4 hrs/a lot of time; 4=4-8 hrs/most of day; 5=More than 8 hours/persistent or continuous
- 10. Could/can you stop thining about killing yourself or wanting to die if you want to? 1=Easily; 2=Little Difficulty; 3=Some Difficulty; 4=Lot of Difficulty; 5=Unable to control; 0=Does not attempt to control
- 11. Are there things that stop you from wanting to die or acting on thoughts of committing suicide? 1=Definite deterrents; 2=Probably Deterrents; 3=Uncertain Deterrents; 4=Unlikely Deterrents; 5=No Deterrents; 0=Does not apply
- 12. What sort of reasons did you have for thinking about wanting to die or killing yourself? Was it to end pain or stop the way you were feeling or to get attention, revenge or reaction from others 1=Completely to get attention or revenge or reaction; 3=Equally to get attention or revenge or reaction and stop pain; 4=Mostly to stop pain; 5=Completely to stop pain; 0=Does not apply

#### **Suicidal Behavior**

13. Have you made a suicide attempt?

**Listing 31. Columbia-Suicide Severity Scale mITT (continued)** 

| | | | Response to Question: | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject ID No. | Treatment<br>Group | Study<br>Week | Q14 | Q15 | Q16 | Q17 | Q18 | Q19 | Q20 | Q21 | Q22 | Q23 | Q24 |
| XXX | HORIZANT | -1, 2, 4 | XX | Yes | Yes | XX | Yes | XX | Yes | Yes | Yes | 0 | 0 |
| | Placebo | 6, 8, 10 | | No | No | | No | | No | No | No | 1 | 1 |
| | | 12, 14, 16 | | | | | | | | | | 2 | 2 |
| | | 18, 20, 22 | | | | | | | | | | 3 | |
| | | 24, 26 | | | | | | | | | | 4 | |
| | | | | | | | | | | | | 5 (date mm/dd/yyyy) | |

- 14. Number of attempts
- 15. Has the subject engaged in non-suicidal self-injurious behavior?
- 16. Has there been a time when you started to do something to end your life but someone or something stopped you before actually did anything?
- 17. Number interrupted
- 18. Has there been a time when you stared to do something to try to end your life but you stopped yourself before you actually did anything?
- 19. Number aborted
- 20. Have you taken any step towards making a suicide attempt or preparing to kill yourself?
- 21. Suicidal behavior was present during the assessment period
- 22. Completed suicide?
- 23. Actual Lethality/Medical Damage; 0=No physical damage; 1=Minor physical damage; 2=Moderate physical Damage; 3=Moderately severe physical damage; 4=Severe physical damage; 5=Death
- 24. Potential Lethality; 0=Behavior not likely to result in injury; 1=Behavior likely to result in injury, but not death; 2=Behavior likely to result in death

**Listing 32. Blood Chemistries – mITT Subjects** 

| Subject<br>ID | Treatment<br>Group | Visit Date | Test Name | Result | Units | Flag | Evaluation |
|---|---|---|---|---|---|---|---|
| XXXX | HORIZANT | mm/dd/yyyy | Creatinine | X.XX | mg/dL | H (high) | WNL |
| | Placebo | | Total Bilirubin | XXX | mg/dL | L (low) | Abnormal, NCS |
| | | | ALT | XX.X | U/L | | Abnormal, CS |
| | | | AST | X.XX | U/L | | |
| | | | GGT | XX.X | U/L | | |

Listing 33. Pregnancy Test/Birth Control Data – mITT Subjects

| Subject ID | Treatment Group | Pregnancy Test<br>Performed? | Pregnancy Test<br>Date | Pregnancy<br>Result | Methods of birth control |
|---|---|---|---|---|---|
| XXX | HORIZANT | Not Done | mm/dd/yyyy | Negative | Oral Contraceptive |
| | Placebo | | | Positive | Contraceptive Sponge |
| | | | | | Contraceptive Skin Patch |
| | | | | | Double Barrier |
| | | | | | Intrauterine |
| | | | | | Etonogestrel implant |
| | | | | | Medroxyprogesterone |
| | | | | | Complete Abstinence |
| | | | | | Hormonal Viginal contraceptive Ring |
| | | | | | Surgically Sterile |
| | | | | | Postemopausal |
| | | | | | Partner surgically Sterile |
| | | | | | Other: xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |

Programming note: Only indicate birth control methods that were indicated as Yes

**Listing 34. Blood Alcohol Concentration – mITT Subjects** 

| Subject<br>ID | Treatment<br>Group | Visit Date | Study<br>Week | BAC<br>Performed | Time of BAC | BAC % |
|---|---|---|---|---|---|---|
| XXX | HORIZANT | mm/dd/yyyy | Screen | Done | hh:mm | x.xxx |
| | Placebo | | 2 | Not Done | | |
| | | | 4 | | | |
| | | | 6 | | | |
| | | | 8 | | | |
| | | | 10, 12 | | | |
| | | | 16, 20 | | | |
| | | | 24, 26 | | | |
| | | | 27 | | | |

**Listing 35. Urine Drug Screen** 

| Subject<br>ID | Treatment<br>Group | Visit Date | Study<br>Week | AMP | Benzos | Coc | Bup | Meth | Methadone | Opioids | THC |
|---|---|---|---|---|---|---|---|---|---|---|---|
| XXX | HORIZANT | mm/dd/yyyy | Screen | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes |
| | Placebo | | 2, 4 | No | No | No | No | No | No | No | No |
| | | | 6, 8 | | | | | | | | |
| | | | 10, 12 | | | | | | | | |
| | | | 16, 20 | | | | | | | | |
| | | | 24, 26 | | | | | | | | |
| | | | 27 | | | | | | | | |

Listing 36. Vital Signs and Body Weights- mITT Subjects

| Subject ID | Treatment<br>Group | Visit Date | Study<br>Week | Weight (Kg) | Heart Rate (beats/min) | Systolic Pressure (mmHg) | Diastolic Pressure<br>(mmHg) |
|---|---|---|---|---|---|---|---|
| XXX | HORIZANT | mm/dd/yyyy | Screening | XXX | XXX | xxx | xxx |
| | Placebo | | 4 | | | | |
| | | | 8 | | | | |
| | | | 12, 16, 20 | | | | |
| | | | 24, 26, 27 | | | | |

**Listing 37. ECG – mITT Subjects** 

| Subject ID | Treatment Group | Visit Date | Study<br>Week | Result | If abnormal, specify finding |
|---|---|---|---|---|---|
| xxx | HORIZANT<br>Placebo | mm/dd/yyyy | Screen 1<br>27 | Normal<br>Abnormal, NCS<br>Abnormal, CS | xxxxxxxxxx |

**Listing 38. Prior and Concomitant Medications – mITT Subjects** 

| Subject<br>ID | Treatment<br>Group | Prior<br>Med? | Verbatin Med/<br>Coded Med | Indication | Route | Frequency | Dose | Start Date | Stop Date | Continuing? |
|---|---|---|---|---|---|---|---|---|---|---|
| XXX | HORIZANT | Yes | xxx/ xxxx/ xxxxxx | XXXXXX | XXXXXX | XXXXXX | XXXXXX | dd/mmm/yyyy | dd/mmm/yyyy | Yes |
| XXX | Placebo | No | xxx/ xxxx/ xxxxxx | | | | | | | No |

Concomitant medications will be coded to a drug term using the WHO Drug Dictionary (recent version).

Listing 39. Comments – mITT Subjects

| Subject ID | Treatment<br>Group | | Comments |
|------------|---------------------|--------------|----------|
| Xxx | HORIZANT<br>Placebo | xxxxxxxxxxxx | |

## 12.3. Figures

Figure 1: Percentage of Subjects No Heavy Drinking Days Weeks 22-25 with Imputation



Programmer note: Use percent on y-axis, bar graph of PSNHDD add Cohen's h, \* a significant p-value, put values on graph

Figure 2: Percentage of Subjects Abstinent Weeks 22-25 No Imputation



Programmer note: bar graph of PSA add Cohen's h, \* a significant p-value, put values on graph

Figure 3: Percentage of Subjects with WHO 1-Level Decrease in Alcohol Consumption Weeks 22-25 No Imputation



Programmer note: bar graph of WHO 1-level add Cohen's h, \* a significant p-value, put values on graph

Figure 4: Percentage of Subjects with WHO 2-Level Decrease in Alcohol Consumption Weeks 22-25 No Imputation



Programmer note: bar graph of WHO 2-level add Cohen's h, \* a significant p-value, put values on graph

Figure 5: Weekly Percentage of Subjects No Heavy Drinking Days with Imputation (mITT)

Programmer note: graph of estimates out to 25 weeks. Include 95% confidence intervals for each estimate and \* on statistically significant differences between treatment groups.

Figure 6: Monthly Percentage of Subjects No Heavy Drinking Days with Imputation (mITT)

Note: 4 week month periods start on Week 2 of maintenance period

Figure 7: Weekly Percentage of Subjects Abstinent with Imputation (mITT)

Figure 8: Monthly Percentage of Subjects Abstinent with Imputation (mITT)

Note: 4 week month periods start on Week 2 of maintenance period

- Figure 9: Weekly Percentage WHO 1-Level Decrease in Alcohol Consumption No Imputation (mITT)
- Figure 10: Monthly Percentage WHO 1-Level Decrease in Alcohol Consumption No Imputation (mITT)

Note: 4 week month periods start on Week 2 of maintenance period

- Figure 11: Weekly Percentage WHO 2-Level Decrease in Alcohol Consumption No Imputation (mITT)
- Figure 12: Monthly Percentage WHO 2-Level Decrease in Alcohol Consumption No Imputation (mITT)

Note: 4 week month periods start on Week 2 of maintenance period

## Figure 13: Cumulative Grace Periods for Percentage of Subjects No Heavy Drinking Days with Imputation (mITT)

Programmer note put all of the grace periods (full maintenance period, last 20 weeks, 16 weeks, 12 weeks, 8 weeks, and 4 weeks) on the same graph

## Figure 14: Cumulative Grace Periods for Percentage of Subjects Abstinent No Imputation (mITT)

Programmer note put all of the grace periods (full maintenance period, last 20 weeks, 16 weeks, 12 weeks, 8 weeks, and 4 weeks) on the same graph

# Figure 15: Cumulative Grace Periods for Percentage WHO 1-Level Decrease in Alcohol Consumption no Imputation (mITT)

Programmer note put all of the grace periods (full maintenance period, last 20 weeks, 16 weeks, 12 weeks, 8 weeks, and 4 weeks) on the same graph

## Figure 16: Cumulative Grace Periods for Percentage WHO 2-Level Decrease in Alcohol Consumption no Imputation (mITT)

Programmer note put all of the grace periods (full maintenance period, last 20 weeks, 16 weeks, 12 weeks, 8 weeks, and 4 weeks) on the same graph

- Figure 17: Percentage Days Abstinent per Week Least Squares Means (Untransformed) no Imputation (mITT)
- Figure 18: Percent Heavy Drinking Days per Week Lease Squares Means (Untransformed) no Imputation (mITT)
- Figure 19: Mean Drinks per Week Lease Squares Means (Untransformed) no Imputation (mITT)
- Figure 20: Mean Drinks per Drinking Day by Week Least Squares Means (Untransformed) no Imputation (mITT)
- Figure 21: Weekly Number of Cigarettes Smoked in Smokers Over Entire Maintenance Period – Least Squares Means no Imputation (mITT)

Programmer note: graph of estimates out to 25 weeks. Include 95% confidence intervals for each estimate and \* on statistically significant differences between treatment groups.

- Figure 22: ACQ-SR-R Score by Visit Least Squares Means (Untransformed) no Imputation (mITT)
- Figure 23: ImBIBe Score by Visit Least Squares Means (Untransformed) no Imputation (mITT)
- Figure 24: PSQI Score by Visit Least Squares Means (Untransformed) no Imputation (mITT)
- Figure 25: PSQI Sleep Quality Score by Visit Least Squares Means (Untransformed) no Imputation (mITT)
- Figure 26: PSQI Sleep Latency Score by Visit Least Squares Means (Untransformed) no Imputation (mITT)
- Figure 27: PSQI Sleep Duration Score by Visit Least Squares Means (Untransformed) no Imputation (mITT)
- Figure 28: PSQI Sleep Disturbanced Score by Visit Least Squares Means (Untransformed) no Imputation (mITT)
- Figure 29: PSQI Use of Sleep Medication Score by Visit Least Squares Means (Untransformed) no Imputation (mITT)
- Figure 30: PSQI Daytime Dysfuction Score by Visit Least Squares Means (Untransformed) no Imputation (mITT)
- Figure 31: BAI by Visit Least Squares Means (Untransformed) no Imputation (mITT)
- Figure 32: BDI-II by Visit Least Squares Means (Untransformed) no Imputation (mITT)
- Figure 33: ROC BAI by PSNHDD Weeks 22-25 (mITT)
- Figure 34: ROC BDI-II by PSNHDD Weeks 22-25 (mITT)
- Figure 35: ROC PSQI Total Score by PSNHDD Weeks 22-25 (mITT)

- Figure 36: ROC POMS Total Score by PSNHDD Weeks 22-25 (mITT)
- Figure 37: ROC POMS Tension-Anxiety by PSNHDD Weeks 22-25 (mITT)
- Figure 38: ROC POMS Depression-Dejection by PSNHDD Weeks 22-25 (mITT)
- Figure 39: ROC POMS Vigor-Activity by PSNHDD Weeks 22-25 (mITT)
- Figure 40: ROC POMS Fatigue-Inertia by PSNHDD Weeks 22-25 (mITT)
- Figure 41: ROC POMS Anger-Hostility by PSNHDD Weeks 22-25 (mITT)
- Figure 42: ROC POMS Confusion-Bewilderment by PSNHDD Weeks 22-25 (mITT)
- Figure 43: ROC ACQ-SR-R by PSNHDD Weeks 22-25 (mITT)
- Figure 44: ROC Days Abstinent (7 Days Prior to Randomization) by PSNHDD Weeks
  - 22-25 (mITT)
- Figure 45: ROC Years Drinking Regularly by PSNHDD Weeks 22-25 (mITT)
- Figure 46: ROC Drinks per Week by PSNHDD Weeks 22-25 (mITT)
- Figure 47: ROC Reducer by PSNHDD Weeks 22-25 (mITT)
- Figure 48: ROC BIS by PSNHDD Weeks 22-25 (mITT)
- Figure 49: ROC Total Dose by PSNHDD Weeks 22-25 (mITT)
- Figure 50: Clinical Chemistry Values Over Time

## Appendix A. Scale and Scoring Instructions for Pittsburg Sleep Quality Index

### Instructions:

The following questions relate to your usual sleep habits during the past month *only*. Your answers should indicate the most accurate reply for the *majority* of days and nights in the past month. Please answer all questions.

| 1. Du | ring the past month, wh | nen have you usually go<br>USUAL BED TIME . | | |
|---|---|---|---|---|
| 2. Du | ring the past month, ho | w long (in minutes) has NUMBER OF MINUTE | s it usually take you to fa | all asleep each night? |
| 3. Dur | ring the past month, wh | en have you usually go<br>USUAL GETTING UP TII | otten up in the morning' | ? |
| 4. Dur<br>tha | n the number of hours | w many hours of <i>actua</i><br>you spend in bed.)<br>OURS OF SLEEP PER N | | ight? (This may be different |
| 5. Dur | | w often have you had to | best response. Please a<br>rouble sleeping becaus | |
| | Not during the | | Once or | Three or more |
| | past month | once a week | twice a week | times a week |
| (b) | Wake up in the middle | e of the night or early m | noming | |
| | Not during the | Less than | Once or | Three or more |
| | past month | once a week | twice a week | times a week |
| (c) | Have to get up to use | the bathroom | | |
| | Not during the | Less than | Once or | Three or more |
| | past month | once a week | twice a week | times a week |
| (d) | Cannot breathe comfo | ortably | | |
| | Not during the | Less than | Once or | Three or more |
| | past month | Less than once a week | twice a week | times a week |
| (e) | Cough or snore loudly | | | |
| | Not during the | Less than | Once or | Three or more |
| | past month | once a week | twice a week | times a week |
| (f) i | Feel too cold | | | |
| | Not during the | Less than | Once or | Three or more |
| | past month | once a week | twice a week | times a week |
| (g) | Feel too hot | | | |
| | Not during the | Less than | Once or | Three or more |
| | past month | once a week | twice a week | times a week |
| (h) | Had bad dreams | | | |
| | Not during the | Less than | Once or | Three or more |
| | past month | once a week | twice a week | times a week |
| | Have pain | | | |
| | Not during the | Less than | Once or | Three or more |
| | past month | | twice a week | times a week |

| | (j) Other reason(s), plea | ase describe | | |
|---|---|---|---|---|
| | How often during the past month have you had trouble sleeping because of this? | | | |
| | Not during the | Less than | Once or | Three or more |
| | past month | once a week | twice a week | times a week |
| 6. | During the past month, | how would you rate yo | our sleep quality overal | 1? |
| | Very good | | | |
| | Fairly good | | | |
| | Fairly bad | | | |
| | Very bad | <del></del> | | |
| 7. | During the past month, you sleep? | how often have you ta | ken medicine (prescribe | ed or "over the counter") to hel |
| | | Less than | Once or | Three or more |
| | nast month | once a week | twice a week | times a week |
| 8. | During the past month, | how often have you ha | | e while driving, eating meals, o |
| | engaging in social active Not during the | | Once or | Three or more |
| | not during the | Cess triair | twice a week | times a week |
| 9. | During the past month, | how much of a probler | m has it been for you to | keep up enough enthusiasm t |
| | get things done? | | | |
| | No problem | | - | |
| | | slight problem | | |
| | | of a problem | | |
| | A very big p | | | |
| 10. | Do you have a bed part | | | |
| | • | ner or roommate | | |
| | | mmate in other room | | |
| | | ame room, but not san | ne bed | • |
| | Partner in sa | | | |
| | - | or bed partner, ask h | im/her how often in the | past month you have had |
| | (a) Loud snoring | | | _ |
| | Not during the | Less than | Once or | Three or more |
| | | | | times a week |
| | (b) Long pauses between | | ρ | |
| | Not during the | Less than | Once or | Three or more |
| | | | twice a week | times a week |
| | (c) Legs twitching or jerl | king while you sleep | | |
| | Not during the | Less than | Once or | Three or more |
| | past month | once a week | twice a week | times a week |
| | (d) Episodes of disorient | tation or confusion dur | ring s <del>lee</del> p | |
| | Not during the | Less than | Once or | Three or more |
| | past month | once a week | twice a week | times a week |
| | (e) Other restlessness w | rhile you sleep; please | describe | |
| | Not during the | Less than | Once or | Three or more |
| | past month | once a week | twice a week | times a week |

## Scoring Instructions for the Pittsburgh Sleep Quality Index

The Pittsburgh Sleep Quality Index (PSQI) contains 19 self-rated questions and 5 questions rated by the bed partner or roommate (if one is available). Only self-rated questions are included in the scoring. The 19 self-rated items are combined to form seven "component" scores, each of which has a range of 0-3 points. In all cases, a score of "0" indicates no difficulty, while a score of "3" indicates severe difficulty. The seven component scores are then added to yield one "global" score, with a range of 0-21 points, "0" indicating no difficulty and "21" indicating severe difficulties in all areas.

Scoring proceeds as follows:

Examine question #6, and assign scores as follows:

| Response | Component 1 score |
|---------------|-------------------|
| "Very good" | 0 |
| "Fairly good" | 1 |
| "Fairly bad" | 2 |
| "Very bad" | 3 |

Component 1 score: \_\_\_\_\_

#### Component 2: Sleep latency

1. Examine question #2, and assign scores as follows:

| Response | Score |
|---------------|-------|
| ≤ 15 minutes | 0 |
| 16-30 minutes | 1 |
| 31-60 minutes | 2 |
| > 60 minutes | 3 |

Question #2 score: \_\_\_\_\_

2. Examine question #5a, and assign scores as follows:

| Response | Score |
|----------------------------|-------|
| Not during the past month | 0 |
| Less than once a week | 1 |
| Once or twice a week | 2 |
| Three or more times a week | 3 |

Question #5a score: \_\_\_\_\_

3. Add #2 score and #5a score

Sum of #2 and #5a: \_\_\_\_\_

4. Assign component 2 score as follows:

| Sum of #2 and #5a | Component 2 score |
|-------------------|-------------------|
| 0 | 0 |
| 1-2 | 1 |
| 3-4 | 2 |
| 5-6 | 3 |

Component 2 score: \_\_\_\_\_

#### Component 3: Sleep duration

Examine question #4, and assign scores as follows:

| Response | Component 3 score |
|-----------|-------------------|
| > 7 hours | 0 |
| 6-7 hours | 1 |
| 5-6 hours | 2 |
| < 5 hours | 3 |

Component 3 score: \_\_\_\_\_

| Component 4: Habitual sleep efficiency | | |
|---|---|---|
| (1) Write the number of hours slept (questi | | - |
| (2) Calculate the number of hours spent in | bed: | |
| Getting up time (question | # 3): | |
| — Bedtime (question # 1): | | |
| Number of hours spent in | bed: | |
| (3) Calculate habitual sleep efficiency as f | | |
| (Number of hours slept/Number of hou | | 0 = Habitual sleep efficiency (%) |
| () × 100 = | | |
| (4) Assign component 4 score as follows: | | |
| Habitual sleep efficiency % | Component 4 score | |
| > 85% | 0 | |
| 75-84% | 1 | |
| 65-74% | 2 | |
| < 65% | 3 | |
| \ 65 /e | • | Component 4 score: |
| Component 5: Sleep disturbances | | Component vocare. |
| (1) Examine questions # 5b-5j, and assign | scores for each que | stion as follows: |
| Response | Score | |
| Not during the past month | 0 | |
| Less than once a week | 1 | |
| Once or twice a week | 2 | |
| Three or more times a week | | |
| | #5b score | |
| | c score | |
| | d score | |
| | e score | |
| | f score | |
| | g score<br>h score | |
| | i score | |
| | j score | |
| (2) Add the scores for questions # 5b-5j: | , 300/0 | |
| | b-5j: | |
| (3) Assign component 5 score as follows: | o o, | |
| | mponent 5 score | |
| 0 | 0 | |
| 1-9 | 1 | |
| 10.10 | 2 | |
| 19-18<br>19-27 | 3 | |
| 13-21 | · · | Component 5 score: |
| Component 6: Use of sleeping medical | tion | |
| Examine question # 7 and assign scores as follows: | | |
| Response Component 6 score | | |
| Not during the past month 0 | | |
| Less than once a week | 1 | |
| Once or twice a week | 2 | |

3

Component 6 score: \_\_\_\_\_

Three or more times a week

| Component 7: Daytime dysfunction | on · | |
|---|---|---|
| (1) Examine question # 8, and assign | | |
| Response | Score | |
| Never | 0 | |
| Once or twice | 1 | |
| Once or twice each we | ek 2 | |
| Three or more times ea | ach week 3 | |
| | Question # 8 score: | |
| (2) Examine question # 9, and assign | n scores as follows: | |
| Response | Score | |
| No problem at all | О О | |
| Only a very slight prob | lem 1 | |
| Somewhat of a probler | n 2 | |
| A very big problem | 3 | |
| | Question # 9 score: | |
| (3) Add the scores for question # 8 a | .nd # 9: | |
| • | Sum of #8 and #9: | |
| (4) Assign component 7 score as follows: | | |
| Sum of # 8 and #9 | Component 7 score | |
| 0 | 0 | |
| 1-2 | 1 | |
| 3-4 | 2 | |
| 5-6 | 3 | |
| | | Component 7 score: |
| Global PSQI Score | | |
| Add the seven component score | s together: | |

Global PSQI Score: \_\_\_\_\_